### STATISTICAL ANALYSIS PLAN

A Phase 3, Multicenter, Randomized, Double-Blind, Placebo- and Active Comparatortrolled, Parallel-Group Study to Evaluate the Efficacy and Safety of Bimekizumab in AdultSubjects with Moderate to Severe Chronic Plaque Psoriasis

mendment Number Date
AP
nent 1 Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Binekizumab in Adult

**SAP/Amendment Number** 

Final SAP Amendment 1

Amendment 2


This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


## **TABLE OF CONTENTS**

| LIST O | F ABBRE | EVIATIONS | 7 |
|---|---|---|---|
| 1 IN | ΓRODUC | TION | 10 |
| 2 PR | OTOCOL | SUMMARY | 10 |
| 2.1 Stu | dy object | ives | 10 |
| 2.1.1 | Prim | ary objective | 10 |
| 2.1.2 | | ndary objectives | |
| 2.1.3 | Othe | r objectives | |
| 2.2 Stu | dy variab | les | 5511 |
| 2.2.1 | Effic | r objectives les acy variables Primary efficacy variables Secondary efficacy variables Other efficacy variables macokinetic variable y variables Secondary safety variables Other safety variables macogenomic variables unological variable and conduct y description y periods Screening Period Initial Treatment Period | |
| 2. | 2.1.1 | Primary efficacy variables | 11 |
| 2. | 2.1.2 | Secondary efficacy variables | 11 |
| 2. | 2.1.3 | Other efficacy variables | 12 |
| 2.2.2 | Phari | macokinetic variable | 13 |
| 2.2.3 | Safet | y variables | 13 |
| 2. | 2.3.1 | Secondary safety variables | 13 |
| 2. | 2.3.2 | Other safety variables | 13 |
| 2.2.4 | Phari | macogenomic variables | 14 |
| 2.2.5 | Imm | unological variable | 14 |
| 2.3 Stu | dy design | and conduct | 14 |
| 2.3.1 | Study | y description | 14 |
| 2.3.2 | Study | y periods | 14 |
| 2. | 3.2.1 | Screening Period | 14 |
| 2. | 3.2.2 | Initial Treatment Period | 15 |
| 2. | 3.2.3 | Maintenance Treatment Period | 15 |
| 2. | 3.2.4 | Safety Follow-Up Period | 16 |
| | 3.2.5 | Premature End of Treatment | |
| 2.3.3 | Study | duration per subject | 16 |
| 2.3.4 | Plam | ned number of subjects and sites | 16 |
| 2.3.5 | V V | cipated regions and countries | |
| 2.4 Det | erminatio | on of sample size | 17 |
| 3 DA | TA ANA | LYSIS CONSIDERATIONS | 17 |
| 3.1 Gei | neral pres | entation of summaries and analyses | 17 |
| 3.2 Det | finition of | Baseline values | 19 |
| 3.3 Ma | pping of | data from early withdrawal visits | 19 |
| 3.4 Pro | tocol dev | iations | 20 |
| 3.5 An | alysis sets | S | 20 |
| 3 5 1 | Enro | lled Set | 20 |

| 3 | .5.2 | Randomized Set | |
|---|---|---|---|
| 3 | .5.3 | Safety Set | 20 |
| 3 | .5.4 | Full Analysis Set. | 20 |
| 3 | .5.5 | Active Medication Set | 20 |
| 3 | .5.6 | Maintenance Set | 20 |
| 3 | .5.7 | Per Protocol Set | 20 |
| 3 | .5.8 | Pharmacokinetics Per-Protocol Set | 21 |
| 3.6 | Treatn | Pharmacokinetics Per-Protocol Set | |
| 3.7 | Center | r pooling strategy | 21 |
| 3.8 | Codin | g dictionaries | 22 |
| 3.9 | Relati | ve day | 22 |
| 3.10 | ) Chang | ges to protocol-defined analyses | 22 |
| 4 | STAT | ISTICAL/ANALYTICAL ISSUES | 23 |
| 4.1 | Adjus | tments for covariates. | 23 |
| 4.2 | Handl | ing of dropouts or missing data | 23 |
| 4 | .2.1 | Handling missing data for efficacy variables | 23 |
| | 4.2.1 | .1 Handling missing data for the primary efficacy variable | 24 |
| | 4.2.1 | | |
| | 4.2.1 | | 24 |
| | 4.2.1 | | 24 |
| | 4.2.1 | | 24 |
| | 4.2.1 | | |
| 4 | .2.2 | Handling missing data for safety variables | 30 |
| 4.3 | Interir | n analyses and data monitoring | 30 |
| 4.4 | Multio | center studies | 31 |
| 4.5 | Multip | ple comparisons/multiplicity | 31 |
| 4.6 | Use of | f an efficacy subset of subjects | 33 |
| 4.7 | | e-control studies intended to show equivalence | |
| 4.8 | | ination of subgroups | |
| 5 | | Y POPULATION CHARACTERISTICS | |
| 5.1 | .~~ | et disposition | |
| 5.2 | Protoc | col deviations | 34 |
| | DEMO | OGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 34 |
| <b>6</b> .1 | Demo | graphics | 34 |
| 6.2 | | Baseline characteristics | |
| 6.3 | Medic | al history and concomitant diseases | 36 |
| 6.4 | | and concomitant medications | |
| 7 | MEAS. | SUREMENTS OF TREATMENT COMPLIANCE | 37 |

| 8 EFFICA | CY ANALYSES | 39 |
|---|---|---|
| 8.1 Statistics | al analysis of the co-primary efficacy variables | 39 |
| 8.1.1 I | Derivations of co-primary efficacy variables | 39 |
| 8.1.1.1 | Psoriasis Area and Severity Index (PASI) | 39 |
| 8.1.1.2 | PASI90 response at Week 16 | 40 |
| 8.1.1.3 | Investigator's Global Assessment (IGA) Response at Week 16 | 40 |
| 8.1.2 I | Primary analysis of the co-primary efficacy variables | 40 |
| 8.1.3 | Sensitivity Analysis #1 | 42 |
| 8.1.3.1 | Sensitivity Analysis #1 | 42 |
| 8.1.3.2 | Sensitivity Analysis #2 | 42 |
| 8.1.3.3 | Sensitivity Analysis #3 | 43 |
| 8.1.3.4 | Sensitivity Analysis #4 | 43 |
| 8.1.3.5 | Sensitivity Analysis #5 | 43 |
| 8.1.3.6 | Sensitivity Analysis #1 Sensitivity Analysis #2 Sensitivity Analysis #3 Sensitivity Analysis #4 Sensitivity Analysis #5 Sensitivity Analysis #6 Sensitivity Analysis #7 al analysis of the secondary officers variables | 43 |
| 8.1.3.7 | Sensitivity Analysis #7 | 43 |
| 8.2 Statistics | al analysis of the secondary efficacy variables | 44 |
| 8.2.1 I | Derivations of secondary efficacy variables PASI100 response at Week 16 IGA Response at Week 16 PASI75 response at Week 4 | 44 |
| 8.2.1.1 | PASI100 response at Week 16 | 44 |
| 8.2.1.2 | IGA Response at Week 16 | 44 |
| 8.2.1.3 | PASI75 response at Week 4 | 44 |
| 8.2.1.4 | Patient Symptom Diary (PSD) | 44 |
| 8.2.1.5 | | 45 |
| 8.2.1.6 | | |
| 8.2.1.7 | 1 | |
| | Primary analysis of the secondary efficacy variables | |
| 8.2.2.1 | | |
| 8.2.2.2 | 3 | |
| 8.2.2.3 | | |
| | Sensitivity analyses of the secondary efficacy variables | |
| V ) | al analysis of the other efficacy variables | |
| | PASI | |
| 8.3.1.1 | | |
| 8.3.1.2 | | |
| 0212 | Initial Treatment Period | |
| 8.3.1.3 | | |
| | Modified Nail Psoriasis Severity Index (mNAPSI) score | |
| | IGA response | 30<br>51 |

| UCB<br>Statistical An | alysis Plan Bimekizumab | 13 Sep 2019<br>PS0009 |
|---|---|---|
| 8.3.5 | Product of IGA and BSA (IGAxBSA) | 52 |
| 8.3.6 | Dermatology Life Quality Index (DLQI) | 52 |
| 8.3.7 | Patient's Global Assessment of Disease Activity (PGADA) for arthritis v analog scale (VAS) | isual |
| 8.3.8 | Patient Global Assessment of PSO score | 54 |
| 8.3.9 | Patient Symptom Diary (PSD) | 54 |
| 8.3.10 | Health Assessment Questionnaire-Disability Index (HAQ-DI) score | 54 011 |
| 8.3.11 | Psoriatic Arthritis Screening and Evaluation (PASE) | |
| 8.3.12 | Short Form – 36 Items Health Survey (SF-36) | |
| 8.3.13 | Psoriatic Arthritis Screening and Evaluation (PASE) Short Form – 36 Items Health Survey (SF-36) Euro-Quality of Life 5-Dimensions, 3 levels (EQ-5D-3L) | 56 |
| 8.3.14 | Work Productivity and Activity Impairment Questionnaire – Specific He | alth |
| 8.4 Statist | Problem (WPAI-SHP) ical analysis of PsA related efficacy variables ACR20, ACR50, and ACR70 responses Swollen and tender joint counts (66/68 joints evaluations) | 57 |
| 8.4.1 | ACR20, ACR50, and ACR70 responses | 57 |
| 8.4.2 | Swollen and tender joint counts (66/68 joints evaluations) | 58 |
| 8.4.3 | PGADA | 58 |
| 8.4.4 | Physician's Global Assessment of Disease Activity (PhGADA) | 58 |
| 8.4.5 | Patient's Assessment of Arthritis Pain VAS | 58 |
| 8.4.6 | Patient's Assessment of Arthritis Pain VAS. HAQ-DI onal statistical analysis of other efficacy variables. | 58 |
| 8.5 Additi | onal statistical analysis of other efficacy variables | 59 |
| 9.1 Pharm | acokinetics AND PHARMACODYNAMICS | 61 |
| 9.2 Pharm | nacodynamics | 61 |
| 9.3 Immu | nogenicity | 62 |

Auto-antibodies 62

10 SAFETY ANALYSES 64 10.1 Extent of exposure 65

10.2.1 10.2.2 10?

10.2.3.1

10.2.3.2

10.2.3.3 10.2.3.4

9.3.1

9.3.2

10.1.1

10.1.2

| 04 41 41 1 | A 1 | | D1 |
|-------------|-----|-------|------|
| Statistical | Ana | lysis | Plan |

| 10.2.3.5 | Suicidal Ideation and Behavior (SIB) | 75 |
|---|---|---|
| 10.2.3.6 | Inflammatory bowel disease | 75 |
| 10.2.3.7 | Anaphylactic reaction | 76 |
| 10.2.3.8 | Hepatic events and drug-induced liver injuries | 76 |
| 10.3 Clinical laboration | oratory evaluations | 76 |
| | physical findings, and other observations related to safety | |
| 10.4.1 Vita | l signs | 79 |
| 10.4.2 Phys | rical examinationtrocardiograms | 80 |
| 10.4.3 Elec | trocardiograms er safety variables Assessment and management of TB and TB risk factors | S 80 |
| 10.4.4 Othe | er safety variables | 80 |
| 10.4.4.1 | Assessment and management of TB and TB risk factors | 80 |
| 10.4.4.2 | Electronic Columbia Suicide Severity Rating Scale (eC-SSRS) | 80 |
| 10.4.4.3 | Pregnancy testing | 81 |
| 10.4.4.4 | Pregnancy testing | 81 |
| 10.4.4.5 | Patient Health Questionnaire 9 (PHQ-9) scores | 81 |
| 11 REFERENCE | TEC . C.V | 0.3 |
| 12 APPENDIX | CES | 84 |
| 12.1 Appendix A | : MedDRA algorithmic approach to anaphyalaxis | 84 |
| 12.2 Appendix B | : Definition of CTCAE grades | 86 |
| 13 AMENDMI | ENT(S) TO THE STATISTICAL ANALYSIS PLAN | 87 |
| 13.1 Amendment | 1 | 87 |
| 13.2 Amendment | 2 | 107 |
| STATISTICAL A | ANALYSIS PLAN SIGNATURE PAGE | 121 |
| ment cannot be us | : MedDRA algorithmic approach to anaphyalaxis : Definition of CTCAE grades | |


13 Sep 2019

**AST** 

PS0009

Aspartate aminotransferase

### LIST OF ABBREVIATIONS

**ADAb** anti-bimekizumab antibodies

ΑE adverse event AH Abnormal high ΑL Abnormal low

ALT Alanine aminotransferase **AMS** Active Medication Set ANA Anti-nuclear antibodies **ANCOVA** Analysis of covariance

al and any extensions of waitations thereof.

on and any extensions of waitations thereof. ATC Anatomical Therapeutic Chemical

**BKZ** bimekizumab

**BLQ** below level of quantification

BMI body mass index

**BSA** body surface area

cumulative distribution function **CDF** 

CI confidence interval

**CMH** Cochran-Mantel-Haenszel

clinical study report **CSR** 

**CTCAE** Common Terminology Criteria for Adverse Events

CVcoefficient of variation

**DLQI** Dermatology Life Quality Index **DMC Data Monitoring Committee EAER** exposure adjusted event rate **EAIR** exposure adjusted incidence rate

**ECG** electrocardiogram

Electronic Case Report Form **eCRF** 

Euro-Quality of Life 5-Dimensions, 3 levels

Enrolled Set

eC-SSRS electronic Columbia Suicide Severity Rating Scale

**FAS** Full Analysis Set

**GGT** Gamma-glutamyltransferase

**HAQ-DI** Health Assessment Questionnaire-Disability Index

HLT High Level Term


**ICF** Informed consent form Janyextensions or variations thereof. **IGA** Investigator's Global Assessment **IGRA** Interferon-gamma release assay **IMP** investigational medicinal product LFT liver function test lower level of quantification LLOQ last observation carried forward **LOCF MACE** Major adverse cardiovascular events MAR missing at random **MCID** minimal clinically important difference **MCMC** Markov Chain Monte Carlo **MCS** Mental Component Summary Medical Dictionary for Regulatory Activities MedDRA multiple imputation MI modified Nail Psoriasis Severity Index **mNAPSI** missing not at random **MNAR** Maintenance Set MS neutralizing anti-bimekizumab antibodies nADAb NRI non-responder imputation OC Observed case **PASE** Psoriatic Arthritis Screening and Evaluation **PASI** Psoriasis Area and Severity Index **PCS** Physical Component Summary PD pharmacodynamics **PEOT** Premature end of treatment PF Physical function **PGA** Patient's Global Assessment **PGADA** Patient's Global Assessment of Disease Activity PHQ-9 Patient Health Questionnaire pharmacokinetics PK-PPS Pharmacokinetics Per-Protocol Set pp-IGA palmoplantar Investigator's Global Assessment Per Protocol Set **PRO** patient-reported outcome

| <del>-</del> | | |
|---|---|---|
| | PsA | psoriatic arthritis |
| | PSD | Patient symptom diary |
| | PSO | Psoriasis |
| | PT | preferred term |
| | Q4W | every four weeks |
| | QOL | quality of life |
| | RS | Randomized Set |
| | SAE | serious adverse event |
| | SIB | suicidal ideation and behavior |
| | sc | subcutaneously |
| | scalp IGA | every four weeks quality of life Randomized Set serious adverse event suicidal ideation and behavior subcutaneously scalp-specific IGA standard deviation statistical analysis plan Short Form 36 item Health Survey Safety Follow-Up Standard MedDRA query system organ class Safety Set |
| | SD | standard deviation |
| | SAP | statistical analysis plan |
| | SF-36 | Short Form 36 item Health Survey |
| | SFU | Safety Follow-Up |
| | SMQ | Standard MedDRA query |
| | SOC | system organ class |
| | SS | Safety Set |
| | TB | tuberculosis |
| | TEAE | treatment-emergent adverse event |
| | TNF | Tumor necrosis factor |
| | ULN | Upper limit of normal |
| | VAS | visual analog scale |
| | WBC | white blood cell |
| | WHO | World Health Organization |
| | WHO-DD | World Health Organization Drug Dictionary |
| | WPAI-SHP | Work productivity and activity impairment questionnaire |
| | TEAE TNF ULN VAS WBC WHO WHO-DD WPAI-SHP | |
| E GOCTILLE | | |
| (Kis | | |


### INTRODUCTION

ns or variations thereof. This statistical analysis plan (SAP) defines the scope of statistical analyses and provides a detailed description of statistical methodology for the statistical analyses to support the final clinical study report (CSR). The SAP is based on the following study document: Protocol Amendment 4, 21 May 2019.

#### 2 PROTOCOL SUMMARY

#### 2.1 Study objectives

#### 2.1.1 **Primary objective**

The primary objective of the study is to compare the efficacy of bimekizumab (BKZ) administered subcutaneously (sc) for 16 weeks versus placebo in the treatment of the subjects with moderate to severe chronic plaque psoriasis (PSO). and any

#### 2.1.2 Secondary objectives

The secondary objectives of the study are to:

- Evaluate the efficacy of bimekizumab compared to placebo at achieving complete clearance Psoriasis Area and Severity Index 100 [PASI100] after 16 weeks of treatment
- Evaluate the efficacy of bimekizumab compared to placebo after 4 weeks of treatment
- Evaluate the efficacy of bimekizumab compared to ustekinumab after 4 weeks, 12 weeks, 16 weeks, and 52 weeks of treatment
- Evaluate the change in itch, pain, and scaling of bimekizumab compared to placebo after 16 weeks of treatment as reported by subjects using the Patient Symptom Diary
- Evaluate the change in psoriatic scalp disease of bimekizumab compared to placebo after 16 weeks of treatment in subjects with scalp PSO at Baseline
- Assess TEAEs, SAEs, and TEAEs leading to withdrawal adjusted by duration of subject exposure to study treatment

#### Other objectives 2.1.3

The other objectives of the study are to demonstrate the effects of bimekizumab on aspects of the disease:

- Assess the efficacy of bimekizumab over time
- Assess the change of skin-related quality of life (QOL)
- Assess the change of general health-related QOL
- Assess the change in nail PSO over time in subjects with nail PSO at Baseline
- Assess the change in scalp PSO over time in subjects with scalp PSO at Baseline
- Assess the change in palmoplantar PSO over time in subjects with palmoplantar PSO at Baseline

- Assess the change in physical function (as measured by the Health Assessment Questionnaire-Disability Index [HAQ-DI] over time in subjects with psoriatic arthritis (PsA) at Baseline

- Assess the change in symptoms of PSO as reported by subjects using the Patient Symptom Diary (all items) through Week 16

  Assess the PK of bimekizumal

- Assess the immunogenicity of bimekizumab
- Assess work productivity
- Assess the effect of bimekizumab on gene and protein expression, and explore the relationship between genomic, genetic, and proteomic biomarkers and disease biology, drug treatment and inflammatory and immune responses (from consenting subjects who agree to participate in the biomarker substudy)
- Assess the safety and tolerability of bimekizumab

#### 2.2 Study variables

#### 2.2.1 Efficacy variables

## Primary efficacy variables 2.2.1.1

The co-primary efficacy variables are the PASI90 response (defined as a subject that achieves 90% reduction from Baseline in the PASI score) at Week 16 and the Investigator's Global Assessment (IGA) response (defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline) at Week 16.

### Secondary efficacy variables 2.2.1.2

The secondary efficacy variables are:

- PASI100 response at Week 16
- IGA response (defined as Clear with at least a 2-category improvement relative to Baseline) at Week 16
- PASI75 response at Week 4
- Patient Symptom Diary responses for itch, pain, and scaling at Week 16
- Scalp IGA response (Clear or Almost Clear with at least a two-category improvement from Baseline) at Week 16 for subjects with scalp PSO at Baseline
- PASI90 response at Week 12 and 52
- IGA response (Clear or Almost Clear with at least a two-category improvement from Baseline) at Week 12 and 52

#### 2.2.1.3 Other efficacy variables

Change from Baseline variables evaluated during the Initial Treatment Period are relative to the nor simplicity, "change from Baseline" is used below for all such variables. Greater detail will be provided below in the Section 3.2. Note that PASI responder rates will always be calculated relative to the Baseline (first dose) Visit.

The other efficacy variables are listed below and will be and in the protocol schedule of account. Baseline (first dose) Visit. For subjects who switch treatment at the Week 16 Visit, change from

and secondary efficacy variables (which will be summarized separately):

- PASI50, PASI75, PASI90, and PASI100 response
- Time to PASI75, PASI90, and PASI100 response during the Initial Period
- Absolute and percent change from Baseline in PASI score
- Percent of subjects with absolute PASI score  $\leq 1, \leq 2, \leq 3$ , and
- IGA response (Clear with at least 2 category improvement relative to Baseline)
- IGA response (Clear or Almost Clear with at least 2 category improvement relative to Baseline)
- Shift from Baseline in IGA score
- Absolute and percent change from Baseline in the body surface area (BSA) affected by PSO
- Percent of subjects with absolute BSA=0%,  $\leq 1\%$ ,  $\leq 3\%$ , and  $\leq 5\%$
- Absolute and percent change from Baseline in the product of IGA and BSA (IGAxBSA)
- Change from Baseline in Dermatology Life Quality Index (DLQI)
- Percent of subjects achieving a DLQI total score of 0 and 1
- Percent of subjects achieving a minimal clinically important difference (improvement from Baseline of 4 or more) in the DLQI
- American College of Rheumatology (ACR) 20, 50, 70% response (ACR20, 50, 70) in the subpopulation of subjects with PsA at Baseline
- Change from Baseline in the Patient's Global Assessment of Disease Activity (PGADA) for the arthritis visual analog scale (VAS) in subjects with PsA at Baseline
- Change from Baseline in Patient Global Assessment of PSO score
- Change from Baseline in the Patient Symptom Diary responses
- Scalp-specific Investigator's Global Assessment (scalp IGA) response (Clear or Almost Clear with at least a two-category improvement from Baseline) for subjects with scalp PSO at Baseline

- Change from Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) score for subjects with nail PSO at Baseline
- mNAPSI75 response (defined as a subject that achieves at least a 75% reduction from Baseline in the mNAPSI score)
- mNAPSI90 response (defined as a subject that achieves at least a 90% reduction from Baseline in the mNAPSI score)
- mNAPSI100 response (defined as a subject that achieves a 100% reduction from Baseline in the mNAPSI score)
- Palmoplantar Investigator's Global Assessment (pp-IGA) response (Clear or Almost Clear with at least a two-category improvement from Baseline) for subjects with palmoplantar PSO at Baseline
- Change from Baseline in the HAQ-DI for subjects with PsA at Baseline
- Change from Baseline in the PASE questionnaire scores (function score, symptom score, and total score)
- Shift from Baseline in PASE score suggestive of PsA (<47 versus ≥47)
- Change from Baseline in Short Form 36-item Health Survey (SF-36) Physical Component Summary (PCS) score, and Mental Component Summary (MCS) score, and individual domains
- Responses to Euro-Quality of Life 5-Dimensions, 3 levels (EQ-5D-3L), absolute and changes from Baseline in EQ-5D-3L VAS scores
- Change from Baseline in Work Productivity and Activity Impairment Questionnaire-specific health problem (WPAI-SHP) V2.0 adapted to PSO scores

#### 2.2.2 Pharmacokinetic variable

The pharmacokinetic (PK) variable is the plasma concentration of bimekizumab.

#### 2.2.3 Safety variables

#### 2.2.3.1 Secondary safety variables

The secondary safety variables include the following treatment emergent adverse events (TEAEs) and serious adverse events (SAEs).

- TEAEs adjusted by duration of subject exposure to study treatment
- SAEs adjusted by duration of subject exposure to study treatment
- TEAEs leading to withdrawal adjusted by duration of subject exposure to study treatment

# 2.2.3.2 Other safety variables

Safety variables to be assessed are:

- Severity and frequency of AEs (including serious AEs)
- Change from Baseline in vital signs

- Electrocardiogram (ECG) results
- Change from Baseline in clinical laboratory values (chemistry and hematology)

Pharmacogenomic variables

Additional blood samples will be collected from subjects who consent to participate in the substudy at specific time points and stored at -80°C for up to 20 years.

Genomic, genetic, epigenetic, proteins, and metabolite biomarkers the relationship with response to treatment with 1 inflammatory and immune analyses. analyses will be determined when the results of the main study made available.

The candidate exploratory variables are the blood or blood derivative (eg, serum) concentrations of cytokines and chemokines of relevance to interleukin-17 A/F (ILAI7A/F) signaling pathway and PSO biology.

Additional variables may include but will not be limited to serum complement concentrations.

#### 2.2.5 Immunological variable

The immunological variable is the anti bimekizumab antibody level prior to and following investigational medicinal product (IMP).

### Study design and conduct 2.3

### Study description 2.3.1

PS0009 is a phase 3, multicenter, randomized, double-blind, placebo- and active comparatorcontrolled study to evaluate efficacy and safety, pharmacokinetics (PK) of bimekizumab administered sc to subjects with PSO. To be eligible to participate in this study, subjects must be adults with a diagnosis of moderate to severe plaque PSO (PASI\ge 12 and BSA\ge 10\% and IGA score  $\geq 3$  [on a 5-point scale]) who are a candidate for ustekinumab, or for systemic PSO therapy and/or phototherapy. Subjects may have been previously exposed to a biologic therapy.

#### 2.3.2 Study periods

This study will include 4 periods, a Screening Period (2 to 5 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (36 weeks), and a safety follow-up (SFU) Period (20 weeks after the final dose of IMP). The Maintenance Treatment Period starts with the first study drug administration on or after the Week 16 visit. After completion of the Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study. Subjects cenrolling into the open-label study will not have the PS0009 SFU Visit.

The assessments for each period are specified in protocol Table 5-1.

#### 2.3.2.1 **Screening Period**

The Screening Period will last 2 weeks, but can be extended up to a total of 5 weeks in cases where a laboratory assessment needs to be repeated or to allow washout of prohibited

 medications. During this time, eligible subjects will be informed about the study and sign the Informed Consent Form (ICF), laboratory data (hematology, urine, and biochemistry tests) will be obtained, and the doses of medications used to treat PsA, will be verified as stable. The Screening Period will also enable washout of any medications not permitted for use during the study. Subjects who require prophylaxis for latent tuberculosis infection must be on treatment for at least 8 weeks prior to their first dose of IMP. These subjects may be rescreened once they have completed the first 8 weeks of prophylaxis treatment.

One rescreening may be allowed after consultation with the Medical Monitor.

### 2.3.2.2 Initial Treatment Period

During the 16-week Initial Treatment Period, approximately 560 subjects will be randomized 4:2:1 to receive the following blinded IMP regimens:

- Bimekizumab 320mg administered sc every four weeks (Q4W) (320 subjects)
- Ustekinumab (160 subjects)
  - For subjects weighing ≤100kg (220lbs) at Baseline, 45mg sc initially and 4 weeks later
  - For subjects weighing >100kg (220lbs) at Baseline, 90mg sc initially and 4 weeks later
- Placebo administered sc Q4W (80 subjects)

Investigational medicinal product will be administered in the clinic by sc injection at the time points specified in the protocol Table 5-1. Subjects withdrawing early from the study will undergo the premature end of treatment (PEOT) Visit assessments and will enter the SFU Period. Subjects withdrawing early from the study will not be eligible for inclusion in the open-label study.

Subjects will be followed in the double-blinded fashion. Subjects may receive placebo injections at certain visits in order to blind the IMP.

Subjects will be classified as completing the initial treatment period if they complete the Week 16 Visit without early withdrawal from the study or if they start treatment in the maintenance treatment period. The start of the maintenance treatment period marks the end of the initial treatment period.

### 2.3.2.3 Maintenance Treatment Period

After the 16-week Initial Treatment Period, subjects will enter the 36-week Maintenance Treatment Period. The Maintenance Treatment Period will start with the first study drug administration on or after Week 16 and subjects will return to the clinic Q4W through Week 52.

Treatment during the Maintenance Treatment Period will be based on initial treatment, per following rules:

- Subjects in the bimekizumab 320mg treatment arm will continue to receive bimekizumab 320mg Q4W.
- Subjects in the ustekinumab treatment arm will continue on ustekinumab (subjects weighing ≤100kg [220lbs] at Baseline will receive 45mg sc every 12 weeks; subjects weighing >100kg [220lbs] at Baseline will receive 90mg sc every 12 weeks).

• Subjects in the placebo arm will receive bimekizumab 320mg Q4W.

Subjects may receive placebo injections at certain visits in order to blind the IMP.

At the end of the Maintenance Treatment Period, all subjects enrolling in the open-label study will, after signing a new ICF, undergo the Week 52 study assessments and then receive their first dose of bimekizumab in the open-label study. All subjects not enrolling in the open-label study will have the Week 52 study assessments and will enter the SFU Period.

### 2.3.2.4 Safety Follow-Up Period

All subjects not continuing in the open-label study, including those withdrawn from IMP<sub>0</sub>will have SFU Visit 20 weeks after their final dose of IMP.

### 2.3.2.5 Premature End of Treatment

Subjects withdrawing early from the study will undergo PEOT Visit assessments and will enter the SFU Period.

### 2.3.3 Study duration per subject

For each subject, the study will last a maximum of up to 73 weeks, as follows:

- Screening Period: 2 to 5 weeks
- Double-blind, placebo- and active comparator-controlled Initial Treatment Period: 16 weeks
- Double-blind, active comparator-controlled Maintenance Treatment Period: 36 weeks
- Safety Follow-Up Period: a SFU Visit is planned 20 weeks after the final dose of IMP (for subjects not enrolling in the open-label study)

After the 36-week Maintenance Treatment Period, subjects will be allowed to enroll in an open-label study, in which case subjects will undergo the Week 52 study assessments before receiving their first open-label IMP dose. The SFU Visit will not be required for subjects who enroll in the open-label study.

The end of study is defined as the date of the last visit of the last subject in the study.

### 2.3.4 Planned number of subjects and sites

Approximately 750 subjects will be screened in order to have 560 subjects randomized in the study. There will be approximately 320 subjects in the bimekizumab 320mg treatment arm, 160 subjects in the ustekinumab treatment arm, and 80 subjects in the placebo treatment arm. The planned number of study sites is approximately 100. Every eligible subject who signs an ICF will be randomized.

## 2.3.5 Anticipated regions and countries

The regions planned for study conduct are North America, Western Europe, Central/Eastern Europe, and Asia/Australia.

A subset of tables, listings, and figures will be repeated for the subgroup of subjects randomized in Japan. A list of these outputs will be added to the TLF shells.


#### 2.4 **Determination of sample size**

Variations thereof. A total of 560 subjects will be randomly assigned in a 4:2:1 ratio to the following treatment groups:

- Bimekizumab 320mg (320 subjects)
- Ustekinumab (160 subjects)
- Placebo (80 subjects)

The primary efficacy analysis is based on the comparison of bimekizumab to placebo for the coprimary efficacy variables of PASI90 response and IGA response at Week 16. However, Week 16 comparisons of bimekizumab against ustekinumab for PASI90 response and IGA response will also be part of a fixed sequence testing procedure to control for multiplicity. Therefore, this study has been powered to show statistical superiority to ustekinumab based on the co-primary endpoints.

The assumed responder rates for PASI90 at Week 16 are 75%, 58%, and 2% for bimekizumab, ustekinumab, and placebo, respectively. Additionally, the assumed responder rates for IGA are 85%, 68%, and 5% for bimekizumab, ustekinumab, and placebo, respectively. The assumed responder rates for bimekizumab are based on the Phase 2b PS0010 data. The assumptions related to the responder rates for ustekinumab are based on those observed in the CLEAR study (Thaci et al, 2015). The power to show statistical superiority of bimekizumab relative to placebo under these assumptions is >99% for the co-primary endpoints.

The power to detect a statistically significant difference between bimekizumab and ustekinumab at a 2-sided significance level of 0.05 is 95% for PASI90 response and 98% for IGA response. Because both co-primary endpoints are highly powered independently, and because PASI and IGA response tend to be highly correlated, the overall power for achieving superiority on both co-primary endpoints is not calculated here. Note that the power for the non-inferiority testing between bimekizumab and ustekinumab for both PASI90 and IGA responses is >99% based on a 1-sided significance level of 0.025 and a non-inferiority margin of 10%.

### DATA ANALYSIS CONSIDERATIONS 3

### General presentation of summaries and analyses 3.1

Statistical analysis and generation of tables, figures, subject data listings, and statistical output will be performed using SAS Version 9.3 or higher. All tables and listings will use Courier New font size 9.

Descriptive statistics will be displayed to provide an overview of the study results. For continuous variables, descriptive statistics will include number of subjects with available measurements (n), mean, standard deviation (SD), median, minimum, and maximum.

For categorical variables, the number and percentage of subjects in each category will be presented. Unless otherwise noted, the denominator for percentages should be based on the number of subjects included in the respective analysis set. Subjects with missing data will be accounted for using the following approaches:


- For summaries of demographics and Baseline characteristics: summarize percentages based on all subjects in the analysis set and include a "Missing" category (corresponding to subjects with missing data for the variable being summarized) as the last row in the list of categories being summarized.
- For summaries of efficacy and safety endpoints, unless otherwise specified: summarize percentages based only on those subjects with observed data for the variable being summarized. As the denominator may be different from the number of subjects in the analysis set being considered, the denominator should be displayed in the table. The general format for displaying this will be "n/Nsub (%)."

Percentages will be presented to 1 decimal place. If the percentage is 100%, do not present a decimal. If the percentage is 0, do not present the percentage. Typically, the % sign should be presented in the column header, but not with each individual value.

For bimekizumab PK concentrations, summary statistics will include geometric mean, geometric coefficient of variation (CV), 95% confidence intervals for geometric mean, arithmetic mean, SD, median, minimum, and maximum. All summaries of PK variables will be based on the observed values. No imputation will be used.

Decimal places for descriptive statistics will always apply the following rules:

- "n" will be an integer
- Mean, SD, and median will use one additional decimal place compared to the original data
- CV[%] will be presented with one decimal place
- Minimum and maximum will have the same number of decimal places as the original value.

Derived variables in general will display the mean, SD and median to 1 more decimal place than the variables used in the derivation. If the number of decimal places reported in the raw data is varied then use either the maximum raw number of reported decimal places or 3, whichever is the lowest, as a guide for the descriptive statistics.

Statistical tests of efficacy variables will be presented as two-sided p-values rounded to three decimal places. P-values less than 0.001 will be presented as "<0.001" and p-values greater than 0.999 will be presented as ">0.999." Statistical comparisons will be two-sided and will be performed at the 0.05 level of significance.

A complete set of data listings containing all documented data as well as calculated data (eg, change from Baseline) will be generated.

Per protocol, visit windows of  $\pm 3$  days from the first dose to Week 24 and  $\pm 7$  days from Week 28 to Week 52 are permissible. For the SFU Visit, visit window is  $\pm 7$  days from final dose. All by-visit summaries will contain nominal (i.e. scheduled) visits only. Unscheduled visits will not be mapped to scheduled visits except for assessments that occur within a 3-day time window of a scheduled visit. In that case, the assessment will be mapped to the corresponding scheduled visit and will be used for the analysis. This will only occur for some vendor data.

#### 3.2 **Definition of Baseline values**

A Baseline value for a subject is defined as the latest measurement for that subject up to and including the day of administration of first study medication, unless otherwise stated. If a Baseline assessment is taken on the same day as first administration of study medication, it is eligible to be used as the Baseline value, even in the case that the time of the assessment is recorded as taking place after the time of first study medication administration. This is considered acceptable as this measurement is still the best representation of the Baseline value of the given assessment since it is highly unlikely that the study medication could have an impact on any measurement in such a short period of time. However, such cases should be rare as study center personnel are instructed to do all assessments at the Baseline visit prior to administering study medication. One exception to this rule is plasma concentration. If Baseline plasma concentration is measured at a time after the first administration of study medication, then it should not be eligible to be considered as a Baseline plasma concentration. Such cases should be discussed with the quantitative clinical pharmacologist. If a Baseline measurement is missing or not collected, and a Screening value is available, the Screening value will be utilized as Baseline instead.

For subjects who switch treatment from placebo to bimekizumab at the Week 16 Visit, the variables listed below, will have an additional Baseline defined as the Baseline for Maintenance Treatment Period. Baseline for Maintenance Treatment Period is the latest measurement on/prior to the day of first dose in the maintenance period.

Laboratory data (only in shift tables)

te that for any laboratory value the that for any laboratory value the that for any laboratory value the the tables to the tables. Note that for any laboratory value that occurs on the day of treatment switch, that lab value will be attributed and summarized for the treatment they were on previously. For subjects that switch treatment, the Baseline value is the laboratory value of the day of treatment switch.

Baseline values for component scores should be computed using components from the same visit where the relevant measurements were recorded prior to dosing. For example, if the Screening visit has all of the components, but the Baseline visit is missing one or more components, the Baseline value for the component score should be calculated using the Screening visit values.

### Mapping of data from early withdrawal visits 3.3

If the early withdrawal visit occurs at a scheduled visit as outlined in the schedule of assessments, then no mapping is necessary, and any early withdrawal assessments should correspond to that scheduled visit. Premature study withdrawal visit assessments that occur on a date after a scheduled visit will be assigned to the next scheduled site visit per the protocol following the last visit where assessments were available. This approach means that there is a chance that data will be mapped to a visit where a given assessment was not actually collected per the protocol schedule of assessments. Such data will not be summarized in by-visit tables (though it will be available in the listings).


The only exception to the above rule is for anti-bimekizumab antibody assessments, in which all onscneduled visits will not be mapped to scheduled visits. Note that based on the early withdrawal mapping conventions described above, a mapped early withdrawal visit is considered as observed at that visit and should be summarized as such in the tables.

3.4 Protocol deviations

Important protocol deviations are deviations from the protocol which not meaningful impact on study and the protocol which not meaningful impact on study and the protocol which not the protocol which early withdrawal visit assessments will be assigned to the next scheduled visit at which anti-

meaningful impact on study conduct or on the primary efficacy, key safety, or PK outcomes for an individual subject. The criteria for identifying important protocol deviations will be defined within the appropriate protocol-specific document at study start. Important protocol deviations will be reviewed as part of the ongoing data cleaning process. Important protocol deviations including those that lead to exclusion from the analysis sets will be identified and documented prior to unblinding.

#### 3.5 **Analysis sets**

For all analysis sets, each unique subject will only be included once, even if the same subject has more than one unique subject identification.

#### 3.5.1 **Enrolled Set**

The Enrolled Set (ES) will consist of all subjects who have given informed consent.

#### 3.5.2 **Randomized Set**

The Randomized Set (RS) will consist of all randomized subjects.

#### 3.5.3 **Safety Set**

The Safety Set (SS) will consist of all subjects that received at least 1 dose of IMP.

#### Full Analysis Set 3.5.4

The Full Analysis Set (FAS) will consist of all randomized subjects that received at least 1 dose of the IMP and have a valid measurement for each of the co-primary efficacy variables at Baseline.

#### **Active Medication Set** 3.5.5

The Active Medication Set (AMS) will consist of all subjects who have received at least 1 dose of active MP (bimekizumab or ustekinumab). The AMS will be used for summaries of safety that include all data from the initial Treatment Period and/or Maintenance Treatment Period.

#### 3.5.6 **Maintenance Set**

The Maintenance Set (MS) will consist of all subjects who have received at least 1 dose of active IMP (bimekizumab or ustekinumab) in the Maintenance Treatment Period.

#### 3.5.7 **Per Protocol Set**

The Per-Protocol Set (PPS) will consist of all subjects in the RS who had no important protocol deviations affecting the co-primary efficacy variables. Important protocol deviations will be

 predefined and subjects with important protocol deviations will be evaluated during ongoing data cleaning meetings prior to unblinding of the data.

#### 3.5.8 **Pharmacokinetics Per-Protocol Set**

The Pharmacokinetics Per-Protocol Set (PK-PPS) will consist of randomized subjects who received at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration post-dose without important protocol deviations that would affect the concentration.

#### 3.6 Treatment assignment and treatment groups

It is expected that subjects receive treatment as randomized and hence safety analyses will be based on the SS, as randomized. However, if after unblinding it is determined that subjects randomized to placebo or ustekinumab received bimekizumab at any time, then for safety analyses these subjects will be reallocated to the appropriate bimekizumab treatment group, unless otherwise specified. Subjects randomized to bimekizumab will only be reallocated to the placebo or ustekinumab treatment group if they never received bimekizumab. Subjects randomized to ustekinumab will only be reallocated to the placebo if they never received ustekinumab or bimekizumab.

Efficacy analyses should be performed according to randomized treatment and not actual treatment received.

#### Center pooling strategy 3.7

The subject treatment assignment is stratified by prior biologic exposure and region. Geographic regions have been categorized as North America, Western Europe, Central/Eastern Europe, and Asia/Australia. Below is a table of geographic regions with corresponding countries.

Table 3–1: Geographic regions and corresponding countries

| Region | Countries |
|------------------------|-----------------------------------------|
| North America | Canada, United States |
| Western Europe | Belgium, Germany, Italy, United Kingdom |
| Central/Eastern Europe | Hungary, Poland, Russian Federation |
| Asia/Australia | Australia, Japan |

The following center pooling algorithm will be used for each geographic region:

- If a center has 21 or more subjects, then no pooling will be done for that center.
- Centers with fewer than 21 subjects will be ordered from largest to smallest with pooling
  - Two or more centers will be combined until the cumulative subject total is at least 21.
- Two or more centers will 1

   Once ^ Once a pooled center has at least 21 subjects, the process will continue in an iterative fashion for the subsequent centers in the ordered list, where a new pooled center begins each time at least 21 subjects has been reached in the previous pool.


 If this iterative process reaches the end of the ordered list of centers where the final pooled center has fewer than 21 subjects, then the subjects from the centers in that pool

In the event that the percentage of randomized subjects is less than 10% in either of the Asia/Australia or Western Europe regions, the two regions will be combined as a geographic region stratum for efficacy modeling, so that there are no modeling convergence issues across efficacy variables.

3.8 Coding dictionaries

All medications of

**UCB** 

All medications other than study drug will be classified by WHO Anatomical Therapeutic Chemical (ATC) Classification, presenting Anatomical Main Group (ATC Level 1), Pharmacological Subgroup (ATC level 3), and preferred term, using version SEP/2015 of the World Health Organization Drug Dictionary (WHO-DD), according to UCB standard operating procedures.

All AEs will be classified by primary system organ class (SOC), high level term (HLT) and preferred term (PT) using version 19.0 of MedDRA® according to UCB Standard Operating Procedures.

Previous and ongoing medical history will be classified by version 19.0 of MedDRA® SOC and PT.

### 3.9 Relative day

The relative day will be included in different listings and will be calculated as follows:

- If the start (stop) date occurred on or after the first dose, but prior to the double-blind drug stop date, relative day is calculated as start (stop) date minus first dose date + 1
- If the start (stop) date occurred after the last dose of double-blind drug, the relative day to the most recent dose is calculated as start (stop) date minus most recent dose date. The relative day in this situation should be preceded by a '+'
- If the start (stop) date occurred before the first dose, the relative day is calculated as start (stop) date minus first dose date. The relative day in this situation should be preceded by a ٠-٠.

For AEs, relative days for start and stop dates will be calculated as the number of days since the in non-treatment emergent AEs, relative to the first dose. Relative da computed for fully completed dates and will be missing for partial dates.

3.10 Changes to protocol-defined. first injection of the medication. For non-treatment emergent AEs, relative day of onset will be negative if the event started and stopped before the first dose. Relative day will only be

The following variable was added as a secondary efficacy variable and added to the sequential testing procedure:

• IGA response (defined as Clear with at least a 2-category improvement relative to Baseline) at Week 16.

For the following endpoints, the definition of response has been clarified:

- Scalp IGA response (clear or almost clear with at least a two-category improvement from Baseline) for subjects with scalp PSO at Baseline
- Palmoplantar Investigator's Global Assessment (pp-IGA) response (clear or almost clear) with at least a two-category improvement from Baseline) for subjects with palmoplantar PSO at Baseline

The following endpoints are not listed in the protocol, but have been added to the SAP in order to achieve consistency with other studies from the program:

- mNAPSI75/90/100 response (defined as a subject that achieves at least a 75%, 90% and 100% reduction from Baseline in the mNAPSI score)
- Percent of subjects with absolute PASI score  $\leq 1, \leq 2, \leq 3$ , and  $\leq 5$
- Percent of subjects with absolute BSA=0%, ≤1%, ≤3%, and ≤5%

The following additional changes were made:

- The calculation of nominal p-values has been added for selected other efficacy variables
- Modifications have been made to the text regarding the multiple imputation algorithm for clarity
- Change from Baseline in PHQ-9 score is listed an efficacy variable in the protocol. However, it is considered as a safety variable in this SAP.
- Selected TEAE tables were added to include calculation of risk differences.

### 4 STATISTICAL/ANALYTICAL ISSUES

## 4.1 Adjustments for covariates

The primary efficacy analyses and selected secondary analyses will be adjusted for the following covariates:

- Prior biologic exposure
- Region

## 4.2 Handling of dropouts or missing data

## 4.2.1 Handling missing data for efficacy variables

Based on previous studies of biologics in subjects with moderate to severe chronic plaque psoriasis, it is expected that the number of subjects who discontinue prior to Week 16 will be low. For the small percentage of subjects for whom primary endpoint data are unavailable at Week 16, this lack of data is suggestive of an ineffective study treatment, thereby supporting the imputation of nonresponse. Achieving the clinical response and making it through 16 weeks of study treatment are both critical components of the primary outcome. Therefore, nonresponder


PS0009

imputation (NRI) will be used as the method for handling missing data in the primary analysis for binary efficacy variables.

If a subject discontinues study treatment without terminating from the study and still continues with scheduled assessments, all efficacy data after discontinuation of study treatment will be treated as missing and subject to imputation as applicable.

#### 4.2.1.1 Handling missing data for the primary efficacy variable

Missing data for co-primary efficacy variables will be imputed using NRI as primary method. That is, subjects with missing data at Week 16 or who discontinue treatment prior to Week 16 will be counted as non-responders for the analysis.

In addition, sensitivity analyses using MI-MCMC/monotone regression, MI-MCMC/reference based methods, last observation carried forward (LOCF), and observed case (OC) method will be performed which will assess the impact of different methods of handling missing data. These methods are described in Section 8.1.3.1 - Section 8.1.3.3.

#### 4.2.1.2 Handling missing data for the secondary efficacy variables

For secondary binary efficacy variables, missing data will be imputed using NRI as primary method. MI-MCMC/monotone regression and OC methods will be performed as sensitivity analysis.

For secondary continuous efficacy variables, MPMCMC/monotone regression is the primary method for imputing missing data. If the imputation model cannot converge, last observation carried forward (LOCF) will be used. OC method will be performed as sensitivity analysis.

#### Handling missing data for the other efficacy variables 4.2.1.3

For other binary efficacy variables, missing data will be imputed using NRI as primary method.

For other continuous efficacy variables, MI-MCMC/monotone regression method will be used to impute missing data as primary method. If the imputation model cannot converge, last observation carried forward (LOCF) will be used.

For other ordinal variables (EQ-5D-3L, shift in IGA score, and Patient Global Assessment of PSO), OC method will be applied as the primary analysis method. No imputation is applied.

For those other efficacy variables that were included in the sequence testing procedure, OC method will also be applied as sensitivity analysis.

## Handling missing data for subgroup analyses

For subgroup analyses specified in Section 4.8, NRI will be used for responder variables. Only descriptive statistics will be provided.

## Missing data overview and summary

In In In summary, the approaches listed below will be used in this study for handling missing data for efficacy variables as appropriate:

Non-responder imputation (NRI): Subjects who have missing data at the time point of interest are treated as though they did not respond to the treatment.


- Multiple Imputation (MI) Markov Chain Monte Carlo (MCMC) / Monotone Regression: Using multiple imputation methodology, intermittent missing data are imputed based on the
- MCMC / Reference-based imputation: Using multiple imputation methodology, intermittent missing data are imputed based on the MCMC method, and monotone missing data are imputed using an imputation model based on placebo (reference) data.

  Last observation carried forward (LOCF): Post-Baseline missing data are imputed by carrying forward the last available observation (including Baseline).

  Observed case (OC): Missing data are not imputed by the last available observation (including Baseline).
- have not discontinued study treatment at the given time point are considered.

The following table depicts which missing data handling approaches should be used based on variable priority (primary, secondary, other) and variable type (responder, continuous, ordinal).

Table 4-1: Missing data handling approach by variable priority and type

| Variable<br>Priority | Variable Type | NRI | MI<br>(MCMC/<br>Monotone<br>Regression) | MI<br>(MCMC/<br>Reference-<br>based) | LOCF | ОС |
|---|---|---|---|---|---|---|
| Primary | Responder | P | Sagar. | Sa | S | S |
| Secondary | Responder | P | $S^a$ | | | S |
| | Continuous | 2E':C | P | | В | S |
| Other | Responder | P | | | | S <sup>b, c</sup> |
| | Continuous <sup>e</sup> | , Mai | P | | В | $S^b$ |
| | Ordinal | any | | | | $\mathbf{P}^{\mathrm{d}}$ |

P=Primary method, S=Sensitivity method, B=Backup method, NRI=Nonresponder imputation, MI=Multiple imputation, MCMC=Markov Chain Monte Carlo, LOCF=Last observation carried forward, OC=Observed Case Note: Backup method is only applicable when the primary method is unable to converge due to challenges with the imputation model.

#### 4.2.1.6 Missing data algorithms

### MI – MCMC / Monotone Regression

Investigators will be given discretion to discontinue study treatment for subjects not responding in order to provide them with alternative therapy to treat the condition. Therefore, in many cases, missing efficacy data due to study treatment discontinuation should be dependent on the observed efficacy scores, but independent of unobserved data. This would be consistent with a

<sup>&</sup>lt;sup>a</sup> Imputation method is applied on continuous data, and responder variable is derived from the continuous variable based on complete data set.

<sup>&</sup>lt;sup>b</sup> Only applies to by-visit summaries of variables that are in the multiplicity-controlled testing procedure.

<sup>&</sup>lt;sup>c</sup> Includes PASI75, PASI90, PASI100, Scalp IGA, IGA responses, and PSD responder variables

<sup>&</sup>lt;sup>d</sup> Includes Patient Global Assessment of PSO, IGA score, and EQ-5D-3L responses

<sup>&</sup>lt;sup>e</sup> For PASE, OC is the primary analysis method.

missing at random (MAR) pattern of missingness. To investigate the efficacy results under the assumption of data being MAR, a multiple imputation method will be applied as follows:

beyond the first when using a by statement), of subjects with observed values and those needing estimation by multiple imputation. The intermittent missing PASI/IGA values in each data set (ie, missing values for a given subject that has available data before and after the missing time point) will be filled in using the MCMC method with other multiple imputations being performed. The seed was 1.2 other multiple imputations as the seed cannot be set for by groups or each treatment group as the seed cannot be seed cannot be set for by groups or each treatment group as the seed cannot be set for by groups or each treatment group as the seed cannot be set for by groups or each treatment group as the seed cannot be set for by groups or each treatment group as t 1. Create a data set, one for each treatment group (note that a separate imputation procedure other multiple imputation procedures described in this SAP related to MCMC/Monotone Regression analyses will use this same seed as well). For monotone missing data (ie, where all subject data is missing after a given time point), monotone regression will be used to impute missing data. Again, this will be based on the 100 sets of imputations already created using the MCMC method such that there will be 100 imputation in total. In both cases, biologic exposure, geographic region and PASI/IGA values at Baseline and at each post-Baseline visit (in chronological order, see additional notes below about visits to include for different analysis sets) will be included in the imputation model. Note that PASI scores at earlier visits will also be used as predictors for the model of PASI at later visits. The resulting data sets for each treatment arm will be combined into one complete data set based on each of the 100 imputations.

Note: The imputation model will only allow continuous variables. Therefore, prior biologic exposure and region will be re-coded as indicator variables. For prior biologic exposure, this will simply be 0 for biologic-naïve subjects and 1 for biologic-exposed subjects. For region, which has 4 levels, one indicator variable will be defined as 0 for regions other than North America and 1 for North America. Two more indicator variables will be defined similarly replacing North America with Central/Eastern Europe, and Western Europe respectively. An indicator variable for Asia/Australia is not needed as the fourth region will be adequately represented by the other region indicator variables all being 0. In the event that the percentage of randomized subjects is less than 10% in either of the Asia/Australia or Western Europe regions, the two regions will be combined as a geographic region stratum for efficacy modeling, so that there are no modeling convergence issues across efficacy variables. In order to achieve model convergence, prior biologic exposure may be dropped from the model. If convergence is still not obtained, then region may also be dropped from the model.

2. For each complete imputed data set, the dichotomous responder variable (PASI90/IGA 0 or 1) based on the PASI/IGA scores will be computed. Each complete imputed data set will then be analyzed based on the stratified CMH test.

Note: For derivation of PASI90 response, the PASI value at Week 16 in the imputed data sets will be compared directly to the observed Baseline PASI value to determine whether or not a reduction of at least 90% was achieved. If values outside of the pre-defined range of values for PASI (0-72) are imputed, they will be cut off as appropriate after the multiple imputation procedure but before deriving the responder variable. For example, an imputed PASI value of -0.5 would be changed to 0 before deriving the PASI90 responder variable.


Note: Standard rounding rules will be applied to the imputed IGA values in order to derive appropriate after the multiple and IGA score imputed as 1.4 (and assuming a Baseline IGA score of 3), this imputed value would be rounded down to 1, and the minimum change from Baseline of 2 would have been met. Therefore, this subject would be considered an IGA 0/1 responder.

Additional ranges of values for other variables are defined. the binary IGA 0/1 responder variable. In addition, if values outside of the pre-defined range sions or varife

Table 4–2: Allowable ranges for imputation by variable

| Variable | Minimum value | Maximum value | Integer values only |
|---|---|---|---|
| PASI | 0 | 72 | No & |
| IGA | 0 | 4 | Yes |
| PSD item | 0 | 10 | No |
| Scalp IGA | 0 | 4 | Yes dill |
| mNAPSI | 0 | 130 | Nogo |
| BSA | 0 | 100 | Yes |
| IGAxBSA | 0 | 400 | Yes |
| DLQI | 0 | 30 PC 14170 | Yes |
| PGADA | 0 | 100 | Yes |
| HAQ-DI | 0 | 3 2000 | No |
| SF-36 | 0 | 100 | No |
| EQ-5D-3L VAS | o and | 100 | Yes |
| WPAI<br>dimension<br>scores | 0 SUPPORT | 100 | No for variables: "Percent work time missed due to problem" and "Percent overall work impairment due to problem". Yes for variables: "Percent impairment |
| anot be u | o support | | while working due to problem" and "Percent activity impairment due to problem". These two variables can only take values that are multiples of 10. |
| PHQ-9 | 0 | 27 | Yes |

3. The Week 16 results from the specified statistical analysis (e.g. stratified CMH, logistic regression) of each of the 100 imputed data sets will be combined for overall inference using Rubin's rules, which account for the uncertainty associated with the imputed values (Rubin, 1987). This will be done using SAS PROC MIANALYZE.

 Some key points to consider relative to the calculation of the odds ratios and corresponding confidence intervals are noted below:

If stratified CMH or logistic regression are used, the estimates of the odds ratios from the logistic regression model in step 3 follow a log-normal distribution, and a log transformation is needed to normalize these estimates since the procedures for combining results from multiple imputed datasets are based on the assumption that the statistics estimated from each imputed dataset are normally distributed. Therefore, the log of the odds ratio estimates from the logistic regression model are used when combining into a single inference (the use of PROC MIANALYZE in step 3). Appropriate transformations to the standard errors and p-values should also be made in order to get the correct confidence intervals, for the CMH test using the p-value for the general association the Wilson-Hilferty transformation should be used (Ratitch, 2013).

Missing data for continuous primary or secondary efficacy variables will be imputed using MI as appropriate (see Table 4–1). The MI procedure for continuous variables will be similar to that described above with the following differences: 1). No dichotomization will be necessary; and 2) the analysis model will be based on an analysis of covariance (ANCOVA) model.

For other continuous efficacy variables, MI will be used to impute missing data when possible. If the imputation model cannot converge, LOCF will be used. The MI procedure will also be similar to that described above with the following differences: 1) No dichotomization will be necessary; 2) instead of using the stratified CMH test or logistic regression, the imputed data sets will be combined and simple means and standard errors will be calculated using Rubin's rules (via SAS PROC MIANALYZE). For calculation of other descriptive statistics such as the median, min and max, Rubin's rules do not apply. Multiple imputation estimates will be computed by simply averaging the estimates from the multiple repetitions of the imputation algorithm. This is the same approach that will be used when summarizing continuous secondary efficacy variables by subgroup.

Further details about imputation for different analysis sets are provided below:

- Randomized Set When programming multiple imputation based on the RS, PROC MI will be used with a separate data set for each of the 3 randomized treatment groups (Placebo, Bimekizumab 320mg Q4W, Ustekinumab). For Bimekizumab 320mg Q4W and Ustekinumab, include all scheduled assessment visits from Baseline to Week 52. For Placebo, include all scheduled assessment visits from Baseline to Week 16.
- Maintenance Set When programming multiple imputation based on the MS, PROC MI will be used with a separate data set for each of the 3 randomized treatment groups (Placebo, Bimekizumab 320mg Q4W, Ustekinumab) including all scheduled assessment visits from Baseline to Week 52.

### MI – MCMC / Reference-based imputation

In this case, placebo will be described as the reference arm.

This procedure will use an imputation model developed based on data from the placebo group only (Mallinckrodt, 2013). Reference-based multiple imputation assumes that the statistical


behavior of the bimekizumab and placebo-treated subjects after discontinuing study medication Multiple imputations are used to replace missing outcomes for bimekizumab- and placebotreated subjects who discontinued using multiple draws from the posterior predictive distribution estimated from the placebo arm. For binary efficacy variables (eg, PASI90 at Week 16), imputation will be done on the raw PASI before assessing the imputed results for PASI90 response.

The steps for the procedure are as follows:

1. For non-monotone (intermittent) missing data, MCMC will be used to impute PASI with biologic exposure, geographic region. and PASI-11 becomes that of the placebo-treated subjects. All time points after discontinuation of the double-

- Baseline visit (in chronological order, as described in the MCMC step in the previous missing data algorithm) being included in the imputation model. This will be done only once for each subject in order to provide a dataset with monotone missing data.
- 2. Data will be processed sequentially by repeatedly calling SAS® PROC MI to impute missing outcome data at visits t=1,.... T, where T is Week 16 for PASI90 or IGA (as the reference arm (placebo) dataset created in Step 1 only includes assessments from Baseline to Week 16, data cannot be imputed beyond Week 16 in Step 2)...
  - a. *Initialization*. Set t=1 (Baseline visit)
  - b. Iteration. Set t=t+1. Create a data set combining records from bimekizumab- and placebo-treated subjects with columns for covariates (prior biologic exposure and geographic region) and outcomes at visits 1 to t. Outcomes for all bimekizumabtreated subjects are set to missing at visit t and set to observed or previously imputed values at visits 1 to t-1. Outcomes for placebo-treated subjects are set to observed at visit t or observed or previously imputed values at visits 1 to t-1.
  - c. *Imputation*. Run MCMC to impute missing values for visit t using previous outcomes for visits 1 to t-1, prior biologic exposure, and geographic region. Note that only placebo data will be used to estimate the imputation model since no outcome is available for bimekizumab-treated subjects at visit t.
  - d. Repeat steps 2a-2c, 100 times with different seed values (seeds ranging from 853 to 952) to create 100 imputed complete data sets.
    - Analysis. For each completed data set, the outcome (response or change from Baseline) will be calculated using the complete datasets (with no missing data).

Each complete imputed data set will then be analyzed based on the statistical model specified in this study (stratified CMH test). The Week 16 results from stratified CMH test of each of the 100 imputed data sets will be combined for overall inference using Rubin's rules, which account for the uncertainty associated with the imputed values (Rubin, 1987). This will be done using SAS PROC MIANALYZE

#### 4.2.2 Handling missing data for safety variables

For analyses of AEs and concomitant medication usage, a complete date must be established in order to correctly identify the AE or medication as occurring during treatment or not. For purposes of imputing missing components of partially-reported start and stop dates for AEs and concomitant medication will be displayed as reported in the subject data listings (i.e., no imputed values will be displayed in data listings).

Partial AE and concomitant medication start dates will be imputed as follows:

Imputation of Partial Start Dates

- If only the month and year are specified and the month and year of first dose is not the same as the month and year of the start date, then use the 1st of the month
- If only the month and year are specified and the month and year of first dose is the same as the month and year of the start, then use the date of first dose
- If only the year is specified, and the year of first dose is not the same as the year of the start date, then use the 1st of January of the year of the start date
- If only the year is specified, and the year of first dose is the same as the year of the start date, then use the date of first dose
- If the start date is completely unknown and the stop date is unknown or not prior to the date of first dose, then use the date of first dose.

Imputation of Partial Stop Dates

- If only the month and year are specified, then use the last day of the month
- If only the year is specified, then use December 31st of that year
- If the stop date is completely unknown, do not impute the stop date.

In the event of ambiguity or incomplete data which makes it impossible to determine whether a medication was concomitant or an adverse event was treatment emergent, the medication will be considered as concomitant or the adverse event will be considered treatment emergent.

#### Interim analyses and data monitoring 4.3

After the final Week 52 visit, an interim analysis will be performed and a corresponding interim clinical study report (CSR) may be written. A final analysis and updated final CSR will be prepared once all data (through the safety follow-up (SFU) visit) have been collected.

In addition, an independent Data Monitoring Committee (DMC) will periodically review and

Cardiovascular and Neuropsychiatric A 3. ....
monitor relevant Cardiovascular and Neuropsychiatric Adjudication Committees will also periodically review and monitor relevant safety data from this study and advise UCB. Details will be provided in the DMC Charter and in the Adjudication Committee Charters.

Further details related to the DMC will be outlined in a separate analysis plan.


### 4.4 Multicenter studies

The center-by-treatment interaction will be tested by replacing region with center in the logistic regression model used for the sensitivity analysis (Section 8.1.3.6) and adding a center-by-treatment interaction term (Section 8.1.3.7). In the model, center will be based on the original centers prior to pooling (Section 3.7). However, if the model is unable to converge due to a low number of subjects at a given center, a pooling by center will be applied in order to allow the model to converge. If convergence is still not achieved a pooling by region will be applied. If convergence still cannot be achieved, this analysis will not be performed. Detailed strategy in the Section 3.7 will be applied in order to allow the model to converge.

### 4.5 Multiple comparisons/multiplicity

The statistical analysis of the co-primary efficacy variables and selected secondary efficacy variables will account for multiplicity and control the familywise Type I error rate at a 2-sided alpha level of 0.05 by using a fixed sequence testing procedure.

The hypotheses (H<sub>1</sub>, H<sub>2</sub>, H<sub>3</sub>, H<sub>4</sub>, H<sub>5</sub>, H<sub>6</sub>, H<sub>7</sub>, H<sub>8</sub>, H<sub>9</sub>, H<sub>10</sub>, H<sub>11</sub>, H<sub>12</sub>, H<sub>13</sub>, H<sub>14</sub>, H<sub>15</sub>, H<sub>16</sub>, H<sub>17</sub> and H<sub>18</sub>) comparing bimekizumab vs. placebo or bimekizumab vs. ustekinumab will be tested at a 2-sided alpha level of 0.05. The pairwise comparisons will follow the sequential testing sequence in Figure 4–1 and the formal evaluation of statistical significance of each comparison is dependent upon the previous comparison achieving statistical significance at the 5% 2-sided level.

The first 2 hypotheses (H<sub>1</sub> and H<sub>2</sub>) test whether bimekizumab is superior to placebo for PASI90 response and IGA response at Week 16. These are the hypothesis tests corresponding to the coprimary endpoints. If both are rejected at a 2-sided alpha level of 0.05, that alpha will be passed to the next test in the sequence, allowing the testing procedure to proceed.

The hypotheses associated with the subsequent tests are for secondary efficacy endpoints and are based on testing for non-inferiority/superiority relative to ustekinumab or for superiority relative to placebo. Note that while subjects randomized to ustekinumab may receive either the 45mg or 90mg dose (according to weight at Baseline), all subjects randomized to ustekinumab will be analyzed as a single group (and not broken out by dose) since the proposed strategy is consistent with the recommended weight-based dosing for ustekinumab. See Figure 4–1 for details on this procedure.


Figure 4-1: Sequence of testing



BL=Baseline; IGA=Investigator's Global Assessment; PASI=Psoriasis Area Severity Index, PSD=patient symptom diary; PSO=psoriasis; Q4W=every 4 weeks; Q8W=every 8 weeks.


#### 4.6 Use of an efficacy subset of subjects

Active-control studies intended to show equivalence

A non-inferiority margin of 10% has been selected as this is considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO.

4.8 Examination of subgroups

Subgroup analyzers ....

Subgroup analyses will be performed on the PASI75/90/100 and IGA. The following subgroups ion and any exter for analysis will be determined using Baseline data:

- Age (<40 years, 40 to <65 years,  $\ge65$  years)
- Gender (male, female)
- Disease duration (<median, ≥median)
- Region (North America [Canada, USA], Western Europe [Belgium, Germany, Italy, United Kingdom], Central/Eastern Europe [Hungary, Poland, Russian Federation], Asia/Australia [Australia, Japan])
- Weight ( $\leq 100 \text{ kg}, > 100 \text{ kg}$ )
- BMI ( $<25 \text{ kg/m}^2$ , 25 to  $<30 \text{ kg/m}^2$ ,  $\ge 30 \text{ kg/m}^2$ )
- Prior systemic chemotherapy or phototherapy (yes, no)
- Prior biologic exposure (yes, no)
- Prior systemic therapy of any kind (yes, no)
- Baseline disease severity (PASI<20, PASI≥20)
- Antibody positivity (confirmatory assay: negative or positive)

Antibody positivity is the only subgroup that is not determined by Baseline data. It will be presented in a separate table.

The definition of prior systemic therapy of any kind is if a subject received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic chemotherapy or phototherapy. Subjects who never received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic chemotherapy or phototherapy will be classified as not receiving prior systemic treatment for psoriasis.

In addition, in order to assess whether an early response to treatment is predictive of response at later time points, subgroup analyses will be performed for the RS on PASI90/100 and IGA over time using the following early response subgroups:

- PASI75 response (OC) at Week 4 (yes, no) to predict PASI90/100 and IGA (NRI) through Week 52
- PASI90 response (OC) at Week 16 (yes, no) to predict PASI100 (NRI) through Week 52


All summaries will be based on imputed data as appropriate and will include descriptive statistics only.

### 5 STUDY POPULATION CHARACTERISTICS

### 5.1 Subject disposition

Summaries of reasons for screen failures (for all subjects screened), disposition of subjects (for all subjects screened), disposition of analysis sets (for RS), disposition and discontinuation reasons in Initial Treatment Period (for RS) and in Maintenance Treatment Period (for RS), as well as the subjects who discontinued due to AEs in Initial Treatment Period (for RS) and in Maintenance Treatment Period (for MS) will be produced. The disposition of subjects for all subjects screened will include the number of subjects included in each analysis set (RS, SS, FAS, AMS, MS, PPS, and PK-PPS) overall and by site.

The following listings for subject disposition will be provided: subjects who did not meet study eligibility criteria (all subjects screened), subject disposition (all subjects screened), study discontinuation (RS), visit dates (RS), subjects excluded from efficacy analysis (RS).

### 5.2 Protocol deviations

A summary, using the RS, displaying the number and percentage of subjects with an important protocol deviation (including a summary of subjects excluded from the PPS or PK-PPS due to important protocol deviations) by treatment group and in Initial Treatment Period and in Maintenance Treatment Period will be provided.

A by-subject listing of important protocol deviations will be provided.

# 6 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

All summaries detailed in this section will be performed on the RS by treatment group. Summaries for demographics and other Baseline characteristics will also be repeated in SS and MS. If the RS and SS analysis sets are identical the summaries will not be repeated.

### 6.1 Demographics

Demographic variables will be summarized by treatment group and overall.

The following continuous variables will be summarized using descriptive statistics (number of subjects, mean, SD, minimum, median and maximum).

- Age at the time of study entry (years)
  - Height (cm)
- Weight (kg)
- BMI (kg/m²)

BMI (kg/m<sup>2</sup>) will be calculated as:


$$BMI = \frac{\text{Weight (kg)}}{(\text{Height (m)})^2}$$

ition and any extensions or variations thereof.
be . The following categorical variables will be summarized using frequency counts and percentages.

- Age group  $(18 < 65, 65 < 85, \ge 85 \text{ years})$
- Age group ( $\le 18, 19 < 65, \ge 65 \text{ years}$ )
- Age group ( $<40, 40-<65, \ge 65 \text{ years}$ )
- Body weight ( $\leq 100 \text{ kg}$ ,  $\geq 100 \text{ kg}$ )
- Gender
- Race
- Ethnicity
- BMI ( $<25 \text{ kg/m}^2$ , 25 to  $<30 \text{ kg/m}^2$ ,  $\ge 30 \text{ kg/m}^2$ )

By-subject listings of demographics for all subjects screened will be provided.

#### Other Baseline characteristics 6.2

Baseline characteristics (including Baseline clinical measures) will be summarized by treatment group and overall.

Generally, the following continuous variables will be summarized using descriptive statistics (number of subjects, mean, SD, minimum, median and maximum).

- Psoriasis Body Surface Area (BSA; %)
- Psoriasis Area and Severity Index (PASI) score
- Modified Nail Psoriasis Severity Index (mNAPSI) total score
- Modified Nail Psoriasis Severity Index (mNAPSI) total score for subjects with nail involvement (i.e. mNAPSI>0)
- Patient Global Assessment of Disease Activity (PGADA) for arthritis visual analogue scale (VAS) score
- Dermatology Life Quality Index (DLQI) total score
- Duration of disease (years)

Duration of disease (years) will be calculated as:

Disease Duration = 
$$\frac{\text{(Date of randomization - Date of onset of Plaque Psoriasis}^1\text{)}}{365.25}$$

<sup>1</sup>If the date of onset of plaque psoriasis is partial, it should be imputed to the most recent feasible date (ie, last day of the month if only day is missing, or the last day of the year if day and month


are missing). Note that if the date of randomization is missing then the duration of disease will be derived using the date of screening.

The following categorical variables will be summarized using frequency counts and percentages.

ASI≥20)

.no)
.olvement (yes, no)
.ogic therapy (yes, no)
Prior anti-TNF therapy (yes, no)
Any prior systemic therapy (yes, no)
SD item scores: Pain, Iteh, Scaling
ne nail, scalp, and palmoplante
ing mNAPSI>0, Scalp [6]
ubjects received pridule. Prior antiumab.

+1' Baseline nail, scalp, and palmoplantar involvement are based on the number of subjects achieving mNAPSI>0, Scalp IGA>0, and pp-IGA>0, respectively. The categorization of whether or not subjects received prior biologic therapy will be based on the Psoriasis Treatment History CRF module. Prior anti-TNFs include etanercept, adalimumab, infliximab, certolizumab pegol, and golimumab.

By-subject listings of Baseline characteristics will be provided.

### Medical history and concomitant diseases 6.3

Previous and ongoing medical history will be summarized by treatment groups, system organ class (SOC) and preferred term (PT) using MedDRA®. Medical procedures are not coded.

The following listings for medical history and concomitant diseases will be provided: medical history, psoriasis history, concomitant medical procedures, previous and ongoing medical history glossary, previous and ongoing medical history conditions, and procedure history.

### Prior and concomitant medications

Medication start and stop dates will be compared to the date of first dose of treatment to allow medications to be classified as either Prior or Concomitant.
Details of imputation methods for missing or partial dates are described in Section 4.2.2.

Ine number and percentage of subjects taking prior medications (excluding past psoriasis medications) will be summarized by treatment group, overall and by Anatomical Therapeutic Chemical classification (ATC) class, presenting Anatomical Main Group (ATC Level 1).

Pharmacological Subgroup (ATC level 3), and preferred term. The pure 1 taking concomitant medications will be summaria.

Past psoriasis medications will be captured separately and will also be summarized by treatment group. These medications are not subject to dictionary coding. In addition, subjects who failed past psoriasis biologic treatment will be summarized by reason of failure as captured on the Psoriasis Treatment History CRF module.

By-subject listings of all Prior and Concomitant medications, prior and concomitant medications glossary, and psoriasis treatment history will be provided.

#### MEASUREMENTS OF TREATMENT COMPLIANCE 7

Due to the method of administration of the treatments, compliance will be examined in terms of completed injections.

Treatment compliance will be calculated as:

total number of completed injections total number of expected injections

where the total number of expected injections is derived relative to when the subject finishes treatment. In this study, Baseline visit and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 are dosing visits. Two injections are administered at each given visit either with active dosing or placebo injection. It is expected that a subject should complete total 26 injections by the end of study. If a subject discontinues early, then the number of expected injections is based on the time of early discontinuation relative to the dosing visits. For example, if a subject discontinues after Week 8 visit and prior to Week 12 visit, the total number of expected injections will be 6.

A summary of percent treatment compliance categorized as <75% and >≥75% will be provided by treatment group and study periods (Initial Treatment Period for the SS, Maintenance Treatment Period for the MS, and the Initial and Maintenance Treatment Period for the AMS).

A by-subject listing of treatment compliance will be provided.

Table 7-1: Dosing scheme

| Dose Assignment | Baseline<br>(first dose) | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 365 | 40 | 44 | 48 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Bimekizumab 320mg Q4W | •• | •• | •• | •• | •• | •• | •• | •• | · Xe | •• | •• | •• | •• |
| Ustekinumab 45mg<br>(subjects ≤100kg) | ▲ ○ | ▲ ○ | 00 | 00 | ▲ ○ | 00 | 00 | A O OFF | 300 | 00 | ▲ 0 | 00 | 00 |
| Ustekinumab 90mg<br>(subjects >100kg) | <b>A A</b> | <b>A A</b> | 00 | 00 | <b>A A</b> | 00 | 00 | <b>A</b> | 00 | 00 | <b>A A</b> | 00 | 00 |
| Placebo/ bimekizumab 320mg Q4W Q4W=every 4 weeks Notes: A bimekizumab 160m depicted by a black triangle | 00 | 00 | 00 | 00 | •• | •• 7 | • ilcail | •• | •• | •• | •• | •• | •• |
| | | | | Q_V | $\sim$ 0) | | | | | | | | |

### 8 EFFICACY ANALYSES

All efficacy analyses will be performed on the RS unless otherwise specified. All efficacy summary tables will be displayed by treatment group unless otherwise specified.

# 8.1 Statistical analysis of the co-primary efficacy variables

## 8.1.1 Derivations of co-primary efficacy variables

### 8.1.1.1 Psoriasis Area and Severity Index (PASI)

PASI90 is defined to be equal to 1 if the percentage improvement from Baseline in the PASI scores is 90% or greater and 0 if the percentage improvement from Baseline is less than 90%. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = non-responder).

PASI scoring of psoriatic plaques is based on three criteria: redness (R), thickness (T), and scaliness (S). Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for very marked involvement). The body is divided into four areas comprising the head (h), upper extremities (u), trunk (t), and lower extremities (l). In each of these areas, the fraction of total surface area affected is graded on a 0-6 scale (0 for no involvement; up to 6 for 90% - 100% involvement).

The various body regions are weighted to reflect their respective proportion of BSA. The composite PASI score is then calculated by multiplying the sum of the individual-severity scores for each area by the weighted area-of-involvement score for that respective area, and then summing the four resulting quantities as follows (note for R, T, and S scores are as follows: 0 = none, 1 = slight, 2 = moderate, 3 = marked, and 4 = very marked):

$$\begin{aligned} \text{PASI} &= (0.1 \times (R_{\text{h}} + T_{\text{h}} + S_{\text{h}}) \times A_{\text{h}}) + (0.2 \times (R_{\text{u}} + T_{\text{u}} + S_{\text{u}}) \times A_{\text{u}}) \\ &+ (0.3 \times (R_{\text{t}} + T_{\text{t}} + S_{\text{t}}) \times A_{\text{t}}) + (0.4 \times (R_{\text{l}} + T_{\text{l}} + S_{\text{l}}) \times A_{\text{l}}) \end{aligned}$$

where

 $R_h$ ,  $R_u$ ,  $R_t$ ,  $R_l$  = redness score of plaques on the head, upper extremities, trunk, and lower extremities, scored 0-4 respectively;

 $T_h$ ,  $T_u$ ,  $T_t$ ,  $T_l$  = thickness score of plaques on the head, upper extremities, trunk, and lower extremities, scored 0-4 respectively;

 $S_h$ ,  $S_u$ ,  $S_t$ ,  $S_l$  = scaliness score of plaques on the head, upper extremities, trunk, and lower extremities, scored 0-4 respectively;

 $A_h$ ,  $A_v$ ,  $A_t$ ,  $A_l$  = numerical value translation of % area of psoriatic involvement score for the head, upper extremities, trunk, and lower extremities, respectively (where 0 = 0% [clear], 1 = 20% to 10%, 2 = 10% to 30%, 3 = 30% to 50%, 4 = 50% to 70%, 5 = 70% to 90%, and 6 = 90% to 100%).

The highest potential PASI score is 72 for severe disease; the lowest is 0 for no psoriasis lesions. PASI scores are treated as continuous. The percent improvement in PASI scores from Baseline will be computed as:

Baseline PASI — Post Baseline PASI Percent improvement from Baseline =  $100 \times 100$ 

If a subject has experienced an improvement, this measure will be positive. If a subject has experienced a worsening in their condition, this measure will be negative.

lations thereof. If a subject is missing 1 or 2 severity measurements for a certain region, the average of the remaining severity measurement(s) within that region will be utilized to substitute for the missing severity measurement(s) in that region. If the area of affected skin and/or all severity measurements for up to 2 regions are missing, then the missing (R+T+S) x A for a region will be substituted by the average of the available (R+T+S) x A. Otherwise, the PASI will be set to missing.

#### 8.1.1.2 PASI90 response at Week 16

A categorical response variable, PASI90 at Week 16 is defined to be equal to 1 if the percentage improvement from Baseline to Week 16 in the PASI scores is 90% or greater and 0 if the percentage improvement from Baseline to Week 16 is less than 90%. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = non-responder).

#### Investigator's Global Assessment (IGA) Response at Week 16 8.1.1.3

A static IGA for psoriasis will be used to assess disease severity in all subjects during the study. The Investigator will assess the overall severity of psoriasis using the following five-point scale:

Table 8-1: Investigator's Global Assessment

| Score | <b>Short Descriptor</b> | Definition |
|---|---|---|
| 0 | Clear | No signs of psoriasis; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | No thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling |
| 4 | Severe | Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions |

IGA response is defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline at Week 16.

#### 8.1.2 Primary analysis of the co-primary efficacy variables

The co-primary efficacy variables for this study are PASI90 response and IGA response at Week 16, and the corresponding analyses are based on the RS. A subject will be classified as a PASI90 responder if the PASI score at Week 16 has improved at least 90% from Baseline, and IGA

 responder is any subject with a score of 0 or 1 (Clear or Almost Clear) with at least a 2-category improvement from Baseline to Week 16 in IGA score.

The primary analysis will be based on the stratified Cochran-Mantel-Haenszel (CMH) test where region and prior biologic exposure (yes/no) will be used as stratification variables. For the assessment of noninferiority, a noninferiority margin of 10% will be used and evaluated based on some state of the second the confidence interval for the stratified Cochran Mantel-Haenszel risk difference between bimekizumab and ustekinumab. A non-inferiority margin of 10% has been selected as this is? considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO. Therefore, a difference within the 10% non-inferiority margin would suggest a similar impact on efficacy between the treatments. The evaluation of superiority to placebo will use pairwise treatment comparisons based on the CMH test using the p-value for the general association. The odds ratio and associated confidence interval (CI) based on the Wald test will be presented. If one of the treatment groups has 0 or very low response where CMH can no longer be used, the logit method will be applied instead.

To calculate the stratified Mantel-Haenszel risk difference, the method of Greenland and Robins (1985) is used. For each combination of strata, a 2x2 table of treatment group and response is created. A theoretical 2x2 table for a given stratum is shown below, where n = a+b+c+d.

| | Response | |
|-----------------|----------|----|
| Treatment Group | Yes | No |
| Bimekizumab | LOA auth | c |
| Ustekinumab | Piling | d |

Given that structure, the stratified Mantel-Haenszel risk difference, standard error, and two-sided

$$RD_{MH} = \frac{\sum_{i} ((a_i * (b_i + d_i)/n_i) - (b_i * (a_i + c_i)/n_i)}{\sum_{i} ((a_i + c_i) * (b_i + d_i))/n_i}$$

Given that structure, the stratified Mantel-Haenszel risk difference, standard (1-
$$\alpha$$
)\*100% confidence interval may be written as follows: 
$$RD_{MH} = \frac{\sum_{i}((a_{i}*(b_{i}+d_{i})/n_{i}) - (b_{i}*(a_{i}+c_{i})/n_{i})}{\sum_{i}((a_{i}*c_{i}*(b_{i}+d_{i})^{3}] + [b_{i}*d_{i}*(a_{i}+c_{i})^{3}]}}$$

$$SE_{MH} = \sqrt{\frac{\sum_{i}\left\{\frac{[a_{i}*c_{i}*(b_{i}+d_{i})^{3}] + [b_{i}*d_{i}*(a_{i}+c_{i})^{3}]}{(a_{i}+c_{i})*(b_{i}+d_{i})*n_{i}^{2}}\right\}^{2}}}$$

$$CI_{MH} = RD_{MH} \pm \text{probit}(1-(\alpha/2))*SE_{MH}$$

$$CI_{MH} = RD_{MH} \pm \text{probit}(1 - (\alpha/2)) * SE_{MH}$$

For the assessment of non-inferiority of bimekizumab to ustekinumab, the lower 97.5% confidence limit for the stratified Mantel-Haenszel risk difference will be considered. If that value is greater than -10%, then non-inferiority will have been established.

Non-responder imputation will be used to account for missing data in the primary analysis. Specifically, any subject who withdraws from IMP prior to Week 16 or who has missing data for the co-primary efficacy variables at the Week 16 time point will be considered as a non-responder.

The number and percentage of subjects who are PASI90 responders at Week 16 will be summarized. IGA response will be summarized in the same manner as PASI90 responder variable.

A line plot of the percentage improvement from Baseline in PASI score over time by treatment group will be produced.

By-subject listings of PASI and IGA responder variables, PASI and IGA data will be provided.

# 8.1.3 Sensitivity analyses of the co-primary efficacy variables

The following sensitivity analyses for the co-primary efficacy variables will be performed to evaluate the assumptions related to the handling of missing data:

# 8.1.3.1 Sensitivity Analysis #1

Missing data will be addressed by using MI (Markov-Chain Monte Carlo [MCMC] method for intermittent missing data, followed by monotone regression for monotone missing data, see Section 4.2.1.6) to evaluate the effect of the method for handling missing data on the analysis. The actual PASI/IGA scores will be imputed and then dichotomized to obtain the response status. The treatment differences for each imputed data set will subsequently be evaluated using the stratified CMH test as used in the primary analysis. The results from each of the imputed data sets will be combined for overall inference using Rubin's rules, which account for the uncertainty associated with the imputed values (Rubin, 1987). This will be done using SAS PROC MIANALYZE. This procedure assumes a missing at random (MAR) pattern of missingness and corresponds to an estimand of the difference in outcome improvement if all subjects tolerated or adhered to treatment (Mallinckrodt et al, 2012). This is an estimand of efficacy to evaluate the de jure hypothesis.

# 8.1.3.2 Sensitivity Analysis #2

Deviations from the MAR pattern assumed above will be evaluated. A sensitivity analysis will be performed in which, as with the above analysis, intermittent missing data will be imputed using MI based on the MCMC method. However, the remaining monotone missing data will be assumed to follow a missing not at random (MNAR) pattern. These data will be imputed using reference-based imputation in which the imputation model is based on data from placebo group (see Section 4.2.1.6), thereby assuming that monotone missing data follow a trajectory similar to the placebo group (Mallinckrodt et al, 2012). As specified in the previous procedure, actual PASI/IGA scores will be imputed and then dichotomized to get the response status. The treatment differences for each imputed data set will subsequently be evaluated using the

stratified CMH test as used in the primary analysis. The estimand in this procedure is the Sensitivity Analysis #3

This sensitivity analysis will be based on observed data at Week 16. Subjects with missing data or who have prematurely discontinued IMP will be treated as missing (see Section 4.2.1.6 Notes as in the primary efficacy analysis will be sensitivity Analysis.

8.1.3.4 Sensitivity Analysis difference in outcome improvement in all randomized subjects at the planned endpoint of the

The primary efficacy analyses from Section 8.1.2 will be repeated using LOCF as the imputation method (see Section 4.2.1.5).

#### 8.1.3.5 Sensitivity Analysis #5

The primary efficacy analyses from Section 8.1.2 will be repeated based on the FAS and the PPS.

#### 8.1.3.6 Sensitivity Analysis #6

As a sensitivity analysis to the primary analysis method, logistic regression based on the RS will be used. The odds ratio of the responder rates at Week 16 will be estimated and tested between treatment groups using a logistic regression model with factors of treatment group, region, and prior biologic exposure (yes/no). The odds ratio, associated confidence interval (CI), and p-value based on the Wald test will be presented. If the logistic regression model is unable to converge, then prior biologic exposure may be dropped from the model to facilitate convergence. If the model is still unable to converge, then region may be removed from the model as well. In addition, if the logistic regression model cannot converge, then Fisher's exact test will be used for inferential comparisons. As with the primary analysis, missing data will be handled using NRI.

#### Sensitivity Analysis #7 8.1.3.7

The center-by-treatment interaction will be tested by replacing region with center in the logistic regression model described in Section 8.1.3.6 and adding a center-by-treatment interaction term. In the model, center will be based on the original centers prior to pooling. However, if the model is unable to converge due to a low number of subjects at a given center, a pooling (see Section 3.7) will be described in order to allow the model to converge. In order to obtain reasonable estimates of variability for a treatment arm at a given center, a minimum of 21 subjects will be considered acceptable for a center to be included in the model without pooling. Given the 4:2:1 randomization allocation scheme, this should provide a minimum of about 12 subjects in the bimekizumab arm, 6 subjects in the ustekinumab arm, and 3 subjects in the placebo arm. Centers with fewer than 21 subjects will be eligible for pooling. The pooling algorithm used is described in Section 3.7.

In order to achieve model convergence, other explanatory variables e.g. other prior biologic exposure may be dropped from the model as for the logistic regression with region.


If the center-by-treatment interaction is not found to be significant ( $\alpha$ =0.10), then no further analyses will be performed. On the other hand, if the interaction is significant, further analyses will be conducted to determine which center or centers may be the source of interaction. This will be done by running the logistic regression model (including the interaction term) where each center will be systematically removed from the model. This impact of a given center will be based on the change in the interaction p-value when that center is removed. The center or centers that appear to be driving the significant interaction effect will then be removed from the model to verify that conclusions remain the same with or without the influential center(s). This sensitivity analysis will be based on RS with NRI for missing data.

# Statistical analysis of the secondary efficacy variables 8.2

#### **Derivations of secondary efficacy variables** 8.2.1

#### 8.2.1.1 PASI100 response at Week 16

A categorical response variable, PASI100 at Week 16 is defined to be equal to 1 if the percentage improvement from Baseline to Week 16 in the PASI scores is 100% and 0 if the percentage improvement from Baseline to Week 16 is less than 100%. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = non-responder). The definition of percentage improvement from Baseline is given in Section 8.1.1.1.

#### IGA Response at Week 16 8.2.1.2

A categorical response variable, IGA response (Clear with at least 2-category improvement from Baseline) is defined as an IGA score of zero (Table 8-1) with at least 2-category improvement from Baseline.

#### PASI75 response at Week 4 8.2.1.3

A categorical response variable, RASI75 at Week 4 is defined to be equal to 1 if the percentage improvement from Baseline to Week 4 in the PASI scores is 75% or greater and 0 if the percentage improvement from Baseline to Week 4 is less than 75%. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = nonresponder). The definition of percentage improvement from Baseline is given in Section 8.1.1.1.

#### 8.2.1.4 **Patient Symptom Diary (PSD)**

A patient reported outcome (PRO) measure, the Patient Symptom Diary (PSD), will be used to assess key symptoms relevant to subjects with moderate to severe chronic plaque PSO. The electronic (ePRO) diary will be administered on a daily basis from Screening to the end of the Week 16 Visit.

The PSD consists of 14 different items, each measuring an aspect of the disease and its impact on the subject's quality of life. Each item will be scored separately on a 0-10 scale with 0 for no symptom and 10 for very severe or worst symptom. Weekly averages will be derived for each of the 14 items of the Psoriasis Diary up to Week 16. A weekly average is the sum of the scored item over the course of the study week (up to the actual visit date) divided by the number of days on which the item was completed and will be set to missing if four or more daily assessments (irrespective of whether these are consecutive or not) were missing of the corresponding

 question. The Baseline value is also based on a weekly average (up to and including the Baseline visit) and will be computed in the same manner.

Each of three PSD response scores -itch, pain, and scaling, will be characterized in terms of the cumulative percent of subjects demonstrating a pre-specified point improvement at Week 16. The thresholds for the PSD response score of itch, pain, and scaling, will be characterized in terms of the cumulative percent of subjects demonstrating a pre-specified point improvement at Week 16. The thresholds for the PSD response score of itch, pain, and scaling are secured to the pain are secured to the pain are s response score at or above the applicable threshold score (ie, at least 2.39, 1.98, and 2.86 for itch, pain and scaling respectively).

#### Scalp IGA response at Week 16 8.2.1.5

A static IGA for PSO will be used to assess disease severity on the scalp in all subjects during the study.

All subjects will complete the scalp IGA at Baseline. Only subjects with scalp involvement at Baseline will complete the scalp IGA at the other visits specified in the schedule of assessments. Subjects with scalp involvement at Baseline are defined as those with a scalp IGA score >0 at Baseline.

Scalp lesions will be assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale as outlined in the Table 8–2 below. This is the same scale with corresponding descriptors used for the overall IGA, but this will be specific to the scalp.

Table 8-2: Scalp IGA

| Score | <b>Short Descriptor</b> | Detailed Descriptor |
|---|---|---|
| 0 | Clear | Scalp has no signs of PSO; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | Scalp has no thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Scalp has just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Scalp has clearly distinguishable to moderate thickening; dull to bright red, moderate scaling |
| 4 | Severe | Scalp has severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions |

Scalp IGA response at Week 16 is defined as clear [0] or almost clear [1] with at least a twocategory improvement from Baseline to Week 16. For analysis purposes, the evaluation of scalp IGA will be limited to subjects with a Baseline scalp IGA of at least 2. Therefore, if a subject has a score of 2 at Baseline, they can only be considered a responder if their IGA is 0 (thereby meeting the criterion for a two-category improvement from Baseline). Subjects with a Baseline scalp IGA of 1 will be assessed per the protocol but will not be part of the scalp IGA analysis.

#### 8.2.1.6 PASI90 response at Week 12 and 52

IGA response at Week 12 and Week 52

IGA response and IGA 5-point scale are outlined in the Section 8.1.1.3, define at Weeks 12 and 52 respectively.

8.2.2 Primary analysis of the secondary of

Binary (responder) variables will be summarized using frequency tables by treatment group for each visit. Continuous variables will be summarized using descriptive statistics by treatment group for each visit. Primary analysis for secondary efficacy variables will be summarized based on imputed data (NRI), unless otherwise specified.

#### 8.2.2.1 **PASI** and IGA responses

For PASI100 response at Week 16, IGA response (clear) at Week 16, PASI75 response at Week 4, PASI90 and IGA response (clear or almost clear) at Week 12, the stratified CMH test similar to the primary analysis will be implemented to test for non-inferiority/superiority.

For the assessment of non-inferiority, a non-inferiority margin of 10% will be used and evaluated based on the confidence interval for the stratified Mantel-Haenszel risk difference between bimekizumab and ustekinumab. A non-inferiority margin of 10% has been selected as this is considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO. Therefore, a difference within the 10% non-inferiority margin would suggest a similar impact on efficacy between the treatments.

To calculate the stratified Mantel-Haenszel risk difference, the method of Greenland and Robins (1985) is used. For each combination of strata, a 2x2 table of treatment group and response is created. A theoretical 2x2 table for a given stratum is shown below, where n = a+b+c+d.

| | Response | |
|-----------------|----------|----|
| Treatment Group | Yes | No |
| Bimekizumab | a | c |
| Ustekinumab 🔍 | ь | d |

Given that structure, the stratified Mantel-Haenszel risk difference, standard error, and two-sided (1- $\alpha$ )\*100% confidence interval may be written as follows:

$$RD_{MH=} \frac{\sum_{i} ((a_i * (b_i + d_i)/n_i) - (b_i * (a_i + c_i)/n_i)}{\sum_{i} ((a_i + c_i) * (b_i + d_i))/n_i}$$

$$SE_{MH} = \sqrt{\frac{\sum_{i} \left\{ \frac{[a_{i} * c_{i} * (b_{i} + d_{i})^{3}] + [b_{i} * d_{i} * (a_{i} + c_{i})^{3}]}{(a_{i} + c_{i}) * (b_{i} + d_{i}) * n_{i}^{2}} \right\}} \frac{\sum_{i} \left\{ \sum_{i} \left[ \frac{(a_{i} + c_{i}) * (b_{i} + d_{i})}{n_{i}} \right] \right\}^{2}}{\left\{ \sum_{i} \left[ \frac{(a_{i} + c_{i}) * (b_{i} + d_{i})}{n_{i}} \right] \right\}^{2}} \right\}}$$

$$CI_{MH} = RD_{MH} \pm \operatorname{probit}(1 - (\alpha/2)) * SE_{MH}$$

For the assessment of non-inferiority of bimekizumab to ustekinumab, the lower 97.5% confidence limit for the stratified Mantel-Haenszel risk difference will be considered. If that value is greater than -100/2 then non-inferiority will have been established.

Because all place!

Because all placebo subjects will receive bimekizumab treatment starting at Week 16, statistical comparisons against placebo after Week 16 will not be performed.

#### 8.2.2.2 Scalp IGA response

For scalp IGA (Clear or Almost Clear) at Week 16, the stratified CMH test similar to the primary analysis will be applied.

#### 8.2.2.3 **Patient Symptom Diary (PSD)**

For each of the three PSD response scores of itch, pain, and scaling, the following analyses will be performed for the purpose of supporting each item as individual key secondary variables.

Each of three PSD response scores itch, pain, and scaling, will be characterized in terms of the cumulative percent of subjects demonstrating a pre-specified point improvement at Week 16. The thresholds for the PSD response scores of itch, pain, and scaling are 2.39, 1.98, and 2.86, respectively. For this responder analysis, it will be limited to the subjects with a Baseline PSD response score at or above the applicable threshold score (ie, at least 2.39, 1.98, and 2.86 for itch, pain and scaling respectively). Stratified CMH test, similar to the primary efficacy analysis will be applied within each of these responder analyses.

Lastly, the entire distribution of responses for each of PSD response scores of itch, pain and scaling will be evaluated via continuous plots showing the absolute and percent change from Baseline on the X-axis and the percent of subjects experiencing that change on the Y-axis. This distribution curve will reveal the extent to which overall results are driven by outliers who improve or worsen more than others. The cumulative distribution function (CDF) is the probability that the variable takes a value less than or equal to x. That is:

$$x \mapsto F_X(x) = P(X \le x)$$

where the right-hand side represents the probability that the random variable X takes on a value less than or equal to x. The probability that X lies in the interval [a, b] is therefore:

$$F_X(b) - F_X(a)$$
 if  $a < b$ 

Note that cumulative distribution plots will be provided for absolute and percent change from Baseline PSD at Week 16 for itch, pain, and scaling.

#### 8.2.3 Sensitivity analyses of the secondary efficacy variables

For binary response variables (PASI100 at Week 16, IGA Response (clear) at Week 16, PASI75 at Week 4, Patient Symptom Diary responses for Pain, Itch, Scaling, and Scalp IGA at Week 12 and 52, and IGA at Weeks 12 and 52) (Sections 8.1.3.1, 8.1.3.3.) will 1

Missing data for binary secondary efficacy variables will be imputed using NRI. Specifically, if a subject has missing data at the respective visit or has discontinued from study treatment, they will be treated as a non-responder at the respective visit for this analysis.

Missing data for these PSD responder variables will use the MI procedure similar to the sensitivity analysis #1 (Section 8.1.3.1) for the co-primary efficacy variables with the following differences:

- 1. The data included in the imputation model will be limited only to those subjects with sufficiently high Baseline values to achieve the response for a given item (based on observed cases).
- 2. The PSD item value will be imputed. Once imputation has been performed across the 100 iterations specified, any values below 0 and above 10 will be truncated to 0 and 10, respectively.
- 3. The change from Baseline values will be computed based on the complete data sets.
- 4. The analysis model will be based on the CMH test.

### Statistical analysis of the other efficacy variables 8.3

The other efficacy variables are listed below and will be evaluated according to the planned assessments in the protocol, this excludes the timepoints for the primary and secondary variables specified above in Section 8.1.1 and Section 8.2.1.

Binary (responder) variables will be summarized using frequency tables by treatment group for each visit. Continuous variables will be summarized using descriptive statistics by treatment group for each visit. All variables will be summarized based on imputed data (NRI and MCMC/Monotone Regression for binary and continuous variables, respectively), unless otherwise specified.

Missing data for continuous secondary efficacy variables will be imputed using MI. The MI procedure for continuous variables will be similar to sensitivity analysis #1 described in Section 8.1.3.1 for the co-primary efficacy endpoints with the following difference – no dichotomization will be necessary. Also, no requirement of meeting minimum threshold at baseline is needed to be included in imputation for a continuous variable.

For variables that are part of the sequence testing procedure, summaries based on observed case data will also be provided. There may be cases where the multiple imputation model fails to

converge. In such situations, the last observation carried forward (LOCF) approach will instead be used to impute the missing data.

Note that in addition, for subjects who change to bimekizumab from placebo at Week 16, change from two Baselines (i.e. Baseline at Week 0 visit and Baseline at Week 16) will be summarized in MS.

Lastly, by visit summaries will include the bimekizumab and ustekinumab treatment groups. There will be 2 key approaches for understanding the data in the Maintenance Treatment Period:

- 1. Summary of data for the RS through Week 52 based on randomized treatment group.
- 2. Summary of Maintenance Treatment Period data among Week 16 responders only for PASI90, PASI100, IGA (0/1), and DLQI respectively.

Selected summaries for subjects switching from Placebo to Bimekizumab will be provided separately for the MS.

### 8.3.1 PASI

# 8.3.1.1 PASI50, PASI75, PASI90, and PASI100 response

Categorical response variables, PASI50, PASI75, PASI90 and PASI100 over time are defined to be equal to 1 if the percentage improvement from Baseline to visit timepoint in the PASI scores is 50%, 75%, 90% and 100% respectively or greater and 0 if the percentage improvement from Baseline to visit timepoint is less than 50%, 75%, 90% and 100% respectively. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = non-responder). The definition of PASI score percentage improvement from Baseline is given in Section 8.1.1.1.

A line plot of the PASI responder (PASI50, PASI75, PASI90, and PASI100) rate over time, by treatment group will be produced.

# 8.3.1.2 Time to PASI50, PASI75, PASI90, and PASI100 response during the Initial Treatment Period

Time to PASI50, PASI75, PASI90, and PASI100 response (in days) during the Initial Treatment Period will each be calculated as:

Min (Date of first PASIxx response, Date of Week 16 visit) – Date of Baseline visit + 1, with xx representing 50, 75, 90, 100 respectively. All visits including unscheduled visits are considered.

Subjects who discontinue study treatment without achieving a given PASI response prior to Week 16 visit will be censored at the date of the last observed PASI assessment on or prior to the date of treatment discontinuation. Subjects who reach the Week 16 Visit without achieving the given response will be censored at the date of the last observed PASI assessment on or prior to the Week 16 Visit. Subjects will be censored at Baseline if there is no Baseline PASI assessment or no Post Baseline PASI assessment.

Time to PASI50, PASI75, PASI90, and PASI100 response during Initial Treatment Period will each be estimated and presented using the Kaplan-Meier product-limit method for each treatment group.

Kaplan-Meier plots of time to PASI responses will also be presented by treatment group. In these Kaplan-Meier plots, the line will start at 0 (since there are no responders at Week 0) and will increase over time, representing time to achieving the response.

The median time to response, including the two-sided 95% confidence interval, will be calculated for each treatment. Comparisons of bimekizumab vs placebo or ustekinumab will be analyzed using a log-rank test stratified by region and prior biologic exposure.

### 8.3.1.3 **PASI** score

Absolute and percent change from Baseline in PASI score is defined in Section 8.1.1.1.

The percent of subjects with absolute PASI score  $\le 1, \le 2, \le 3$  and  $\le 5$  will be presented over time using NRI.

# 8.3.2 Modified Nail Psoriasis Severity Index (mNAPSI) score

Psoriatic nail disease will be evaluated at the Baseline visit using the mNAPSI. All affected nails will be scored (0 to 3) for onycholysis/oil drop dyschromia, nail plate crumbling, and pitting and will be scored (0 for "no" or 1 for "yes") for leukonychia, nail bed hyperkeratosis, splinter haemorrhages and red spots in the lunula. The score for an individual nail ranges from 0 to 13 with higher scores indicative of more severe nail disease. The total mNAPSI score is the sum of the scores for each individual nail. If a nail is unaffected, it will be recorded as such and will not contribute to the total mNAPSI score.

If any of the 7 response items that contribute to mNAPSI is present, while other items are missing (ie, partial mNAPSI data), then the missing items are assumed to be 0 for the mNAPSI calculation. In some cases, the data may be captured in such a way that only non-zero component scores are present in the database. Again, those components that are not present are simply assumed to be 0 for the mNAPSI calculation.

Change from Baseline in Modified Nail Psoriasis Index (mNAPSI) score for subjects with nail PSO at Baseline is defined as Post-Baseline mNAPSI score minus Baseline mNAPSI.

An mNAPSI75 responder is defined as a subject who achieved at least a 75% improvement from Baseline in the mNAPSI score. mNAPSI90 and mNAPSI100 are defined accordingly. The proportion of mNAPSI75/90/100 responders over time will be summarized for each treatment group.

# 8.3.3 IGA response

IGA response (Clear) is defined as IGA score of zero (Table 8–1) with at least a two-category improvement from Baseline at visit timepoint.

• IGA response (Clear or Almost Clear with at least 2 category improvement relative to Baseline) is defined as IGA score of clear [0] or almost clear [1] with at least a two-category improvement from Baseline at visit timepoint.

- Shift from Baseline in IGA score is defined at each Post-Baseline visit timepoint relative to Baseline.
- Scalp-specific IGA response definition and derivation are outlined in Section 8.2.1.5.
- Palmoplantar Investigator's Global Assessment (pp-IGA) response

A static IGA for palmoplantar PSO will be used to assess palmoplantar disease severity.

Only subjects with palmoplantar involvement at Baseline will complete the pp-IGA at the other visits specified in the protocol. Subjects with palmoplantar involvement at Baseline are defined as those with a pp-IGA score >0 at Baseline.

Palmoplantar disease will be assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale as outlined in the table below.

Table 8–3: Palmoplantar IGA

| Score | Short Descriptor | Detailed Descriptor |
|---|---|---|
| 0 | Clear | Palmoplantar has no signs of PSO; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | Palmoplantar has no thickening, normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Palmoplantar has just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Palmoplantar has clearly distinguishable to moderate thickening; dull to bright red and clearly distinguishable coloration; moderate scaling |
| 4 | Severe | Palmoplantar has severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions; numerous fissures |

PSO=psoriasis; pp-IGA=palmoplantar-specific Investigator's Global Assessment

Palmoplantar IGA response is defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline. For analysis purposes, the evaluation of pp-IGA will be limited to subjects with a Baseline pp-IGA of at least 2. Therefore, if a subject has a score of 2 at Baseline, they can only be considered a responder if their IGA is 0 (thereby meeting the criterion for a two-category improvement from Baseline). Subjects with a Baseline pp-IGA of 1 will be assessed per the protocol but will not be part of the palmoplantar IGA analysis.

A line plot of the IGA responder rates (both clear or almost clear and clear) over time, by treatment group will be produced.

# **Body Surface Area (BSA)**

- His docure. Absolute change from Baseline in the BSA affected by PSO is defined as Post Baseline BSA minus Baseline BSA affected by PSO.
  - Percent change from Baseline in BSA affected by PSO is defined as

Percent change from Baseline  $= 100 \times \frac{\text{Post Baseline BSA} - \text{Baseline BSA}}{\text{Baseline BSA}}$ 

The percent of subjects with absolute BSA=0%,  $\leq$ 1%,  $\leq$ 3% and  $\leq$ 5% will be presented over time.

### 8.3.5 Product of IGA and BSA (IGAxBSA)

- Absolute change from Baseline in the product IGAxBSA is defined as Post Baseline IGAxBSA minus product of Baseline IGAxBSA.
- Percent change from Baseline in the product of IGAxBSA is defined as

Percent change from Baseline  $= 100 \times \frac{\text{Post Baseline IGAxBSA} - \text{Baseline IGAxBSA}}{\text{Baseline IGAxBSA}}$ 

# 8.3.6 Dermatology Life Quality Index (DLQI)

The DLQI questionnaire is used for patients with psoriasis and consists of 10-questions. This is validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment, as assessed over the past week.

The scoring of each answer for the DLQI is as follows:

Table 8-4: Dermatology Life Quality Index

| DLQI Scoring | dilati |
|----------------------------------------|--------|
| Response | Score |
| Very much | 3 |
| A lot | 2 |
| A little | 1 |
| Not at all | 0 |
| Not relevant | 0 |
| Question unanswered | 0 |
| Q7: 'prevented work or studying' = yes | 3 |

The DLQI total score is calculated by adding the score of each question. The maximum score is 30, and the minimum score is 0. The higher the score, the more quality of life is impaired.

Meaning of DLQI Scores

0-1 = no effect at all on patient's life

2-5 = small effect on patient's life

6-10 = moderate effect on patient's life

11-20 = very large effect on patient's life

21-30 = extremely large effect on patient's life

13 Sep 2019 PS0009

This categorization will not be utilized in the analysis.

Because Q7 has a sub-question (referred to as Q7a here) after the leading yes/no question, some clarifying rules for scoring are provided:

- If Q7 is marked as "no", "not relevant", or is missing and Q7a is "A lot", a score of 2 is given.

  If Q7 is marked as "no", "not relevant" or is missing and Q7a is "A lot", a score of 2 is likely given.
- If Q7 is marked as "no", "not relevant", or is missing and Q7a is "Not at all", a score of 0 is given.
- If Q7 is marked as "no" or "not relevant" and Q7a is missing, a score of 0 is given.
- If Q7 is missing and Q7a is missing, Q7 is considered unanswered (see below for details on how this impacts the overall DLQI score).

If 1 question is left unanswered, this is scored 0 and the scores are summed and expressed as usual out of a maximum of 30. If 2 or more questions are left unanswered, the questionnaire is not scored.

A subject is considered to have achieved the minimally clinical important difference (MCID) if their individual improvement from Baseline score is > 4. A 4-point improvement in the DLQI score (DLQI response) has been reported to be meaningful for the subject (within-subject MCID).

A DLQI absolute score of 0 or 1 indicates no or small impact of the disease on health-related quality of life.

The DLQI related efficacy variables are defined as follows:

- Change from Baseline in DLQI is defined as Post-Baseline DLQI minus Baseline DLQI.
- Percent of subjects achieving a DLQI total score of 0 or 1 is defined as the number of subjects with DLQI absolute score of 0 or 1 divided by the number of subjects in RS.
- Percent of subjects achieving a MCID in DLQI is defined as the number of subjects with improvement from Baseline score of 4 or more divided by the number of subjects in RS. Only subjects with a Baseline DLQI of 4 or greater will be considered for this analysis.

# Patient's Global Assessment of Disease Activity (PGADA) for arthritis visual analog scale (VAS)

The PGADA for the arthritis VAS will be used to provide an overall evaluation of arthritis disease symptoms. Subjects will respond to the question, "Considering all the ways your arthritis affects you, please mark a vertical line on the scale below to show how you are feeling today," using a VAS where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms."

All subjects will complete the PGADA at Baseline. Subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47) will complete the PGADA at the visits specified in

Patient Global Assessment of PSO score

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question, "How severe are your psoriasis-related symptoms right now"."

Possible response to the question are "no symptoms", "mild symptoms" "severe symptoms", or "very severe symptoms"."

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question, "How severe are your psoriasis-related symptoms right now"."

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question, "How severe are your psoriasis-related symptoms."

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question are "no symptoms."

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question are "no symptoms."

The Patient Global Assessment of psoriasis will be summarized based on OC as the primary analysis. No imputation is applied.

Shift from Baseline in PGA (Patient Global Assessment) of PSO score is defined to each Post-Baseline visit timepoint relative to Baseline.

#### 8.3.9 **Patient Symptom Diary (PSD)**

Absolute and percent changes from Baseline PSD for each item will be summarized by visit for each treatment group.

For PSD responder analysis, the threshold criteria in term of changes from Baseline are set to 3.05, 1.99, 2.01, 3.04, 2.82, 2.60, 2.69, 2.68, 1.51, 2.43, and 2.14 respectively for the redness, burning, cracking, dryness, irritation, sensitivity, lesions, thickening, fatigue, embarrassment, choice of clothing. Number and percentage of subjects who are responders will be summarized based on each of these items.

In addition, cumulative distribution plots (see details in Section 8.2.2.3) will be provided for absolute and percent change from Baseline PSD at Week 16 for each item.

#### Health Assessment Questionnaire-Disability Index (HAQ-DI) score 8.3.10

The HAQ-DI assesses the degree of difficulty a subject has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category or domain consists of 2 or 3 items. For each question in the questionnaire, the level of difficulty is scored from 0 to 3 with 0 representing "without any difficulty," 1 as "with some difficulty," 2 as "with much difficulty," and 3 as "unable to do". The domain score for each domain is the maximum (ie, worst) of the scores from the items/questions within the domain. If this domain score is > 2, no further adjustment is needed. If it is < 2 (ie, 0 or 1) but no aids, devices or help from another person is indicated, then also no adjustment is needed. However, if it is < 2 and any aid, device or help from another person is indicated, then it is further adjusted upward to 2.

For each domain, the domain score will be determined by non missing scores from the questions. A domain score will only be missing if all scores within the domain are missing. The HAQ-DI total score is the average of all the 8 domain scores. If > 2 domain scores are not complete or missing, HAQ-DI score is considered missing, else the HAQ DI score is computed as the average of the non missing domain scores.

 **UCB** 

Change from Baseline in HAQ-DI is defined as Post-Baseline HAQ-DI minus Baseline HAQ-DI.

(Husni et al, 2014). The questionnaire consists of 15 items that are divided into a 7-item symptoms subscale and an 8-item functions subscale. Standardized responses are based on 5 categories relating to agreement (strongly agree [5], agree [4], no idea [3], disagree [2], and strongly disagree [1]). The total maximum score is 75 points (symptom score: 35 points and function score: 40 points). Psoriatic Arthritis Screening and Evaluation points are indicative of active PsA.

PASE will 1

PASE will be collected at Baseline and Week 52/PEOT visit. PASE will be summarized based on OC only. No imputation is applied.

Change from Baseline in the PASE questionnaire scores (function score, symptom score, and total score) is defined as Post-Baseline PASE questionnaire score (function, symptom, and total) minus Baseline PASE questionnaire score (function, symptom, and total).

Shift from Baseline in PASE score suggestive of PsA (<47 versus ≥47) is defined to Week 52/PEOT visit timepoint relative to Baseline.

#### Short Form - 36 Items Health Survey (SF-36) 8.3.12

The SF-36v2, standard recall, measures the following 8 health domains as rated by the subjects over the past four weeks: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health (Maruish, 2011).

The SF-36 Physical and Mental Component Summary scores (PCS and MCS, respectively) are used to measure the two broad components, or aspects, of health-physical and mental. PCS and MCS are based on the aggregate of 8 health concepts described above and all of the 8 health domain scales are used to score both components summary measures.

One additional item asks respondents about health change over the past year.

The SF-36 will be used using QualityMetric's Health Outcomes<sup>TM</sup> Scoring Software version 5.1 or later. The software uses updates 2009 U.S. population norms and applies a Full Missing Score Estimation (Full MSE) method as follows:

- A health domain score (except the physical functioning (PF) domain) will be estimated provided that at least one non-missing response is available within that domain.
- For the PF domain item response theory will be used to develop a model for estimates of the missing score (Thomas and Cyr, 2002).
- Regression methods are then applied to estimate the PCS and the MCS on the basis of the available domains.
- Change from Baseline in Short Form 36-item Health Survey PCS score, and MCS score, and individual domains is defined as respective score at Post-Baseline timepoint minus the Baseline score.


#### 8.3.13 **Euro-Quality of Life 5-Dimensions, 3 levels (EQ-5D-3L)**

Responses to EQ-5D-3L are scored as 1 for "no problem", 2 for "some or moderate problems", and 3 for "extreme problems"

Absolute EQ-5D-3L VAS score records the respondent". The EQ-5D-3L health questionnaire provides a descriptive profile and a single index value for

20cm scale, 0 to 100 graduated (0=worst imaginable health status, 100=best imaginable health status)

Change from Baseline in EQ-5D-3L VAS scores is defined as Post-Baseline EQ-5D-3L VAS score minus Baseline EQ-5D-3L VAS score.

Responses to EQ-5D-3L will be summarized based on OC only as primary analysis. No imputation is applied to responses to EQ-5D-3L but is applied to EQ-5D-3L VAS scores.

### Work Productivity and Activity Impairment Questionnaire - Specific 8.3.14 **Health Problem (WPAI-SHP)**

The WPAI-SHP is a subject-reported questionnaire that assesses subject's employment status, work absenteeism, work impairment while working, overall work, and daily activity impairment attributable to a specific health problem. Five out of 6 items of the WPAI-SHP are regrouped into the 4 dimensions, with scores expressed as percentage, where higher numbers indicate greater impairment and less productivity, ie, worse outcomes, as described in the WPAI-SHP scoring rules.

The scoring rules for the WPAI-SHP are as follows:

Questions:



Percent work time missed due to problem: [Q2 hours/(Q2 hours +Q4 hours)] \*100

- Percent impairment while working due to problem: [Q5 score/10] \*100
- Percent overall work impairment due to problem: [Q2 hours/(Q2 hours +Q4 hours)+[(1-(Q2 hours/(Q2 hours +Q4 hours))x(Q5 score/10)]] \*100
- Percent activity impairment due to problem: [Q6 score/10] \*100

Change from Baseline score is derived as post Baseline score minus Baseline score. A The Point for the subject.

Statistical analysis of PsA related efficacy variables

The following PsA related efficacy variables will only be assessed for subjects enrolled in Japan:

Swollen and tender joint count

Physician's Global Assessment of Disease Activity (PhGADA)

Patient's Assessment of Arthritis Pain VAS

C-Reactive Protein (CRP)

Subsequently, also ACR20/50/70 are only calculated for subjects. negative change score indicates a reduction in the score/improvement for the subject.

The Patient's Assessment of Arthritis Pain VAS, PGADA, and HAQ-DI will be assessed for all subjects at Baseline. At all subsequent visits, the Patient's Assessment of Arthritis Pain VAS, PGADA, and HAQ-DI will be assessed only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47). Only subjects with PsA at Baseline will be assessed with swollen and tender joint count, and PhGADA at Baseline and subsequent visits.

The number and percentage of subjects with ACR20, ACR50, ACR70 will be summarized by treatment group and visit in subjects with PsA at Baseline.

By-subject listings of ACR responder variables and percent change in ACR components (swelling joints count, tender joints count, PGADA and PhGADA VAS, Patient's Assessment of Arthritis Pain VAS, HAQ-DI, and CRP) from Baseline data will be provided.

#### ACR20, ACR50, and ACR70 responses 8.4.1

American College of Rheumatology (ACR) ACR20/50/70 represents at least 20%, 50%, or 70% respective improvement from Baseline for each of the following:

- Tender joint counts (TJC)
- Swelling joint counts (SJC)
- At least 3 of the 5 remaining core set measures:
  - Disease activity as assessed by PGADA
  - Disease activity as assessed by PhGADA
  - Pain as assessed by Patient's Assessment of Arthritis Pain VAS
    - Physical function as assessed by the HAQ-DI
  - Acute phase response as assessed by the C-reactive protein (CRP)

For all non-missed visits, if any of the component scores are missing, then those scores will be considered as not having met the criteria for improvement for the respective component. For component scores with a Baseline value of 0, the percentage improvement is not calculable and is treated as missing. For component scores with a Baseline value >0 and a post-Baseline value of 0, percentage improvement will be calculated as for any other non-missing data.

#### 8.4.2 Swollen and tender joint counts (66/68 joints evaluations)

Upper body (6): bilateral temporomandibular, sternoclavicular, and acromioclavicular joints

Upper extremity (34): bilateral shoulders, elbows, wrists (includes radiocarred and carpometacarpal bones considered as a single unit). The following 68 joints are to be examined for tenderness by an Investigator who has documented training performing the assessment. The Investigator can also delegate the assessment to a rheumatologist. Preferably the same assessor should evaluate the subject at each arthritis assessment (see Table 8–5).

- Lower extremity (28): bilateral hips, knees, ankles, tarsi (includes subtalar, transverse tarsal, and tarsometatarsal considered as a single unit), metatarsophalangeals (MTP I, II, III, IV, and V), great toe interphalangeals, and proximal interphalangeals (PIP II, III, IV, and V)
- The assessment for swelling is made on 66 joints from the above list. The hip joints are excluded.

Artificial and ankylosed joints are excluded from both tenderness and swelling assessments.



#### **PGADA** 8.4.3

The definition and analysis of PGADA VAS score is given in Section 8.3.7.

#### Physician's Global Assessment of Disease Activity (PhGADA) 8.4.4

The Investigator will assess the overall status of the subject with respect to their PsA signs and symptoms and functional capacity (considering both joint and skin components) using a VAS where 0 is "very good, asymptomatic and no limitation of normal activities" and 100 is "very poor, very severe symptoms which are intolerable and inability to carry out all normal activities."

### Patient's Assessment of Arthritis Pain VAS 8.4.5

The Patient's Assessment of Arthritis Pain VAS or "Pain VAS" is part of the ACR core set of measures in arthritis (Felson et al, 1993).

The Pain VAS consists of a horizontal line 100mm in length on which subjects are asked to Indicate the level of their arthritis pain at the day of the visit between 0 ("no pain") and 100 ("most severe pain") in response to the question: "Please mark a vertical line on the scale below to show how much pain you have from your arthritis today" (Dworkin et al, 2008).

#### 8.4.6 HAQ-DI

The definition, derivation, and analysis of HAQ-DI score is given in Section 8.3.10.

# 8.5 Additional statistical analysis of other efficacy variables

For selected other efficacy variables, it is of interest to perform statistical tests and to calculate inferential statistics. As these tests are not part of the multiplicity-controlled procedure, the associated p-values are considered nominal and are not controlled for multiplicity.

For responder variables, the analysis will follow what was specified for the primary analysis. Specifically, a stratified Cochran-Mantel-Haenszel (CMH) test will be used, where region and prior biologic exposure (yes/no) will be stratification variables. The p-value will be based on the CMH test for a general association. Missing values will be imputed using NRI.

For continuous variables, the MI – MCMC / Monotone Regression approach used for other continuous variables will be applied for the imputation model. The analysis model will be based on analysis of covariance (ANCOVA) with fixed effects of treatment, region, and prior biologic exposure and Baseline value as a covariate.

Below is a list of variables for which these nominal p-values will be calculated (with the time points in parentheses). The results of these inferential tests will all be presented in a single table summarizing the testing performed outside of the multiplicity-controlled testing procedure.

- PASI90
  - Bimekizumab vs Placebo (Weeks 1, 2, 4, 8, and 12)
  - Bimekizumab vs Ustekinumab (Weeks 1, 2, 4, and 8)
- IGA Clear or Almost Clear
  - Bimekizumab vs Placebo (Weeks 1, 2, 4, 8, and 12)
  - Bimekizumab vs Ustekinumab (Weeks 1, 2, 4, and 8)
- PASI100
  - Bimekizumab vs Placebo (Weeks 4, 8, and 12)
  - Bimekizumab vs Ustekinumab (Weeks 4, 8, 12, 16, and 52)
- IGA Clear
  - Bimekizumab vs Placebo (Weeks 4, 8, and 12)
  - Bimekizumab vs Ustekinumab (Weeks 4, 8, 12, 16, and 52)
- PASI95

Bimekizumab vs Placebo (Weeks 1, 2, and 16)

- Bimekizumab vs Ustekinumab (Weeks 1, 2, 4, and 16)
- PSD Response Pain
  - Bimekizumab vs Placebo (Weeks 1, 2, and 4)
  - Bimekizumab vs Ustekinumab (Week 16)
- PSD Response Itch

- Bimekizumab vs Placebo (Weeks 1, 2, and 4)
- Bimekizumab vs Ustekinumab (Week 16)
- PSD Response Scaling
  - Bimekizumab vs Placebo (Weeks 1, 2, and 4)
  - Bimekizumab vs Ustekinumab (Week 16)
- Scalp IGA Clear or Almost Clear (subjects with Baseline Scalp IGA ≥2)
  - Bimekizumab vs Placebo (Weeks 1, 2, and 4)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- pp-IGA Clear or Almost Clear (subjects with Baseline pp-IGA ≥2)
  - Bimekizumab vs Placebo (Week 16)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- mNAPSI change from Baseline (subjects with Baseline mNAPSI>0)
  - Bimekizumab vs Placebo (Week 16)
- mNAPSI75 response (subjects with Baseline mNAPSI>0)
  - Bimekizumab vs Placebo (Week 16)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- mNAPSI90 response (subjects with Baseline mNAPSI>0)
  - Bimekizumab vs Placebo (Week 16)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- mNAPSI100 response (subjects with Baseline mNAPSI>0)
  - Bimekizumab vs Placebo (Week 16)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- DLQI change from Baseline
  - Bimekizumab vs Placebo (Week 16)
- DLQI 0/1 response
  - Bimekizumab vs Placebo (Week 16)
  - Bimekizumab vs Ustekinumab (Weeks 16 and 52)
- SF-36 PCS change from Baseline
  - Bimekizumab vs Placebo (Week 16)
- SF-36 MCS change from Baseline

- Bimekizumab vs Placebo (Week 16)
- any extensions or variations thereof. WPAI-SHP change from Baseline (percent impairment while working, percent overall work impairment, percent activity impairment)
  - Bimekizumab vs Placebo (Week 16)
- PASI percentage change from Baseline
  - Bimekizumab vs Placebo (Weeks 1, 2, 4, 8, 12, and 16)
- PASI ≤2 response
  - Bimekizumab vs Placebo (Weeks 1, 2, 4, 8, 12, and 16)
- PASI ≤5 response
  - Bimekizumab vs Placebo (Weeks 1, 2, 4, 8, 12, and 16)

#### PHARMACOKINETICS AND PHARMACODYNAMICS 9

#### 9.1 **Pharmacokinetics**

Pharmacokinetic variables will be analyzed for all subjects in the PK-PPS. Bimekizumab plasma concentrations will be summarized for each treatment at each scheduled visit.

PK summaries will be based on observed values. No imputation will be used. However, if plasma concentration measurements are below the level of quantification (BLQ), then for calculation of the derived statistics the result will be set to 0.125 µg/ml, which is ½ of the lower level of quantification (LLOQ). Descriptive statistics including geometric mean, geometric coefficient of variation, and geometric mean 95% CI if applicable will be calculated if at least 2/3 of the values of interest are above the LLOQ. If this is not the case, only median, minimum, and maximum will be presented.

In addition, geometric mean plasma concentration will be plotted by treatment group, and by cumulative antibody status for subjects randomized to bimekizumab on linear and log linear scale.

If the dosing for a visit is +/- 21 days out of window, then the plasma concentration from that visit and all subsequent visits will be excluded from the PK summary.

If the PK sampling date is >1 day after the dosing date data points will be excluded from the PK summary tables and figures, but not from the listing.

However, all PK concentrations will be listed.

The PK will be subject to a population PK and PK/PD analysis and will be described in a separate analysis plan and reported independently.

#### 9.2 **Pharmacodynamics**

Not applicable

#### 9.3 **Immunogenicity**

Anti-bimekizumab antibodies

Anti-bimekizumab antibodies will be measured using a three tiered assay approach: screening assay, confirmatory assay and titration assay. Samples confirmed as positive within the confirmatory assay, will be further evaluated in a neutralizing assay to evaluate the ADAb to neutralize the activity of Bimekizumab (II 174) were taken at Baseline, Week 4, Week 8 Week 52 and in subject. weeks after the last dose.

Anti-bimekizumab antibody samples are not analyzed when subjects are on a treatment other than bimekizumab. For subjects who switch from placebo to bimekizumab, samples are analyzed starting at the visit when the switch to bimekizumab occurs. The sample at the visit when the switch occurs will act as the Baseline for that treatment group. For subjects randomized to Ustekinumab, no ADAb samples will be analysed.

In subjects randomized to placebo for the first 16 weeks, no samples will be analysed until Week 16 which will act as the Baseline for this treatment group.

Screening, confirmatory and titer cut points of the respective assays will be determined by the bioanalytical laboratory based either on using commercially available drug-naïve samples or on the pre-dose samples of the study itself. In case cut point is being set on commercially available samples, the representative for the study population is being checked. The screening cut point will be used to determine the status of ADA in test sample as above the cut point or below the cut point. Samples presenting ADA levels above the cut point, will be further evaluated in the confirmatory assay, the result of which will be reported as either "confirmed positive" or "not confirmed positive".

- Values ≤ screening cut point (BCP) or above the screening cut point and confirmed negative (NCP) are defined as anti-bimekizumab antibody negative
- Values > predefined screening cut point (ACP) and confirmed positive (CP) are defined as anti-bimekizumab antibody positive

Confirmed positive samples will be titrated, and the titer (reciprocal dilution factor including MRD) reported. The samples (or a subset) will also be subject to a neutralizing assay to evaluate whether the anti-bimekizumab antibody neutralizes the activity of bimekizumab (IL17 A or IL17F or both) in-vitro. This will be reported subsequent to the main DBL and CSR.

### Subject Classification:

Pre anti-bimekizumab antibody negative – treatment emergent anti-bimekizumab antibody negative: Includes subjects who are negative at Baseline and antibody negative at all sampling points post treatment (excluding SFU)


- Pre anti-bimekizumab antibody negative treatment emergent anti-bimekizumab rre anti-bimekizumab antibody positive – treatment emergent reduced antibimekizumab antibody: Includes subjects who are positive at Baseline, and antibody negative at all sampling points post treatment (excluding SFU).

  Pre anti-bimekizumab antibody positive – treatment emergent reduced antibimekizumab antibody positive – treatment emergent em antibody positive: Includes subjects who are negative at Baseline and antibody positive at
- positive at any sampling point post treatment (excluding SFU) with titer values of the same magnitude as Baseline (ie, less than a 2.07 fold difference from the Baseline value).
- Pre anti-bimekizumab antibody positive treatment emergent anti-bimekizumab antibody boosted positive: Includes subjects who are positive at Baseline and are positive at any sampling point post treatment (excluding SFU) with increased titer values compared to baseline (greater than a 2.07 fold difference increase from Baseline value which will be defined within the validation of the assay).
- **Inconclusive**: Includes subjects who have a positive pre-treatment sample and some posttreatment samples are missing, while other post-treatment samples are anti-bimekizumab antibody negative.

Derivation for above classification will be different for the interim analysis and the final analysis. For the interim analysis no SFU data will be considered. Only for the final analysis, when all SFU data will be available, data from the SFU visits will be considered. That is, each instance of "excluding SFU" in the categories above, should be changed to "including SFU."

In the case that a sample is collected one or more days following the scheduled visit date in which the drug was administered, the anti-bimekizumab antibody results for that sample will be associated with the scheduled visit and summarized accordingly. Such samples will also be considered when anti-bimekizumab antibody results are summarized over a given study period.

### Analysis:

Immunogenicity will be assessed through summary tables and figures, and listing of individual results by subject. All analyses will be run on the safety population, unless specified otherwise.

- Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at the time of each visit, separated by treatment group
- Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at any visit during the treatment period, separated by treatment group.
- The time-point of the first occurrence of anti-bimekizumab anti-body positivity during the treatment period) will be summarized for each treatment group. A plot of the Titre versus elapsed time will be plotted
- All individual subject-level anti-bimekizumab antibody results will be listed.

- The number and percentage of subject in each of the 6 categories will be tabulated and separated by treatment group with an additional category combining subjects in categories 2 and 5, summarized as total treatment emergent. In addition, the counts and percentage of subjects who are pre-anti-bimekizumab positive will be calculated (this is the sum of categories 3,4, and 5).
- The prevalence of immunogenicity, separated by treatment group, and defined subcategory, will be reported per time point, defined as (cumulative) proportion of subjects having confirmed positive ADAb samples at any point up to and including that time point. Missing samples will not be included in the denominator.
- The time to achieving treatment-emergent ADAb positivity, separated by treatment group and defined sub-category, will be analyzed based on Kaplan-Meier approach, subjects will be considered to have an event at time where treatment emergent ADAb positive is first achieved. Subjects classified as treatment-emergent ADAb negative will be censored at time of last available ADAb result.
- A summary of PASI 90 responder, separated by treatment group and defined subcategory, at Weeks 16 and 52 as a function of ADAb titer will be presented graphically.
   This will be repeated for PASI 100 and 75 responders.
- Individual plots of Bimekizumab Concentrations/ADAb titer and % Change from Baseline (all Y-axes) versus time (x-axis) for the full treatment period, including SFU where a patient has not progressed into the OLE. Plots should be labeled and grouped into the 6 sub-categories.
- Spaghetti plots of ADAb titer (Y-axis) against time (X-axis), separated by treatment group for all ADAb positive subjects, including Baseline positive subjects.
- Box plots of all Bimekizumab concentrations where ADAb titers exists versus ADAb titer classification (group 1 >; group 2 >; group 3 >) presented on a linear scale. Cut points will be determined on availability of the titre data.

For purposes of efficacy subgroup analyses based on anti-bimekizumab antibody status, two categories will be used:

- Anti-bimekizumab antibody positive This is defined as subjects who have antibimekizumab antibody levels above the specified cut point on at least 2 time points while on treatment (ie, excluding Baseline, excluding SFU).
- Anti-bimekizumab antibody negative Subjects who are not defined as anti-bimekizumab positive (as described above) will be defined as anti-bimekizumab antibody negative.

# 10 SAFETY ANALYSES

If not specified otherwise, all safety summaries and listings will be created using all subjects in the SS.

Statistical Analysis Plan Bimekizumab

The AMS will be used for summaries of safety that include data from the Initial Treatment Period and/or Maintenance Treatment Period.

medication duration in days. In addition, total study medication duration and time at risk will be summarized in years by treatment group and treatment period (i.e., the Initial Treatment Period, and the Initial and Maintenance Treatment Period (i.e., the Initial Treatment Period). duration will be summarized for subjects exposed for given durations of time, with four weekly categories through Week 16 and 24. For the cumulative duration through Week 52 the following categories for duration will be used:

- >0 weeks
- >=16 weeks
- >=24 weeks
- >=52 weeks

Definitions for study medication duration and time at risk in days are provided in this section. Time at risk will be summarized in years. Time at risk in years is calculated by dividing the time at risk in days by 365.25.

Throughout this section, date of last clinical contact for each subject is defined as the maximum of [last visit date including SFU visit, last imputed AE start date, date of study termination or completion, last date of study drug administration].

### **Exposure during the Initial Treatment Period** 10.1.1

Definitions for study medication duration (days) and time at risk (days) during the Initial Period are provided as follows:

# Study medication duration (days)

- Date of last dose in the Initial Period date of first dose in the Initial Period + 28 days.
  - Note: If date of last dose in the Initial Period + 28 days extends to a date beyond the date of first dose in the Maintenance Treatment Period, then this calculation reverts to:
    - Date of first dose in the Maintenance Treatment Period date of first dose in the Initial Period + 1.

Note: For subjects who die during the Initial Period, if date of last dose in the Initial Period + 28 days extends to a date beyond the date of death, then this calculation reverts to:

 $\circ$  Date of death – date of first dose in the Initial Period + 1.

### Time at risk (days)

For subjects who complete the final visit of the Initial Period and continue to the Maintenance Treatment Period: Date of first dose in the Maintenance Treatment Period – date of first dose in the Initial Period +1.


- For subjects who die prior to the final visit of the Initial Period: Date of death date of first dose in the Initial Period +1.
- Date of last clinical contact date of first. • For subjects who discontinue on or prior to the final visit of the Initial Period, use the minimum of the following:

#### 10.1.2 **Exposure during the Maintenance Treatment Period**

Definitions for study medication duration (days) and time at risk (days) during the Maintenance Period are provided as follows:

## Study medication duration (days)

Date of last dose in the Maintenance Treatment Period – date of first dose in the Maintenance Treatment Period + 28 days.

Note: If date of last dose in the Maintenance Treatment Period + 28 days extends to a date beyond the final visit date of the Maintenance Treatment Period (including PEOT, but not including SFU), then this calculation reverts to:

o Final visit date of the Maintenance Treatment Period (including PEOT, but not including SFU) – date of first dose in the Maintenance Treatment Period + 1.

Note: For subjects who die during the Maintenance Treatment Period, if date of last dose in the Maintenance Treatment Period + 28 days extends to a date beyond the date of death, then this calculation reverts to:

O Date of death – date of first dose in the Maintenance Treatment Period + 1.

### Time at risk (days)

- For subjects who complete the Maintenance Treatment Period as planned and continue into an openlabel study (and, therefore, do not have the SFU visit in the feeder study): Final visit date of the Maintenance Treatment Period – date of first dose in the Maintenance Treatment Period + 1.
- For subjects who die prior to the final visit of the Maintenance Treatment Period: Date of death date of first dose in the Maintenance Treatment Period + 1.
- For all other subjects, use the minimum of the following:
  - Date of last dose in the Maintenance Treatment Period date of first dose in the Maintenance Treatment Period + 140 days.
  - Date of last clinical contact date of first dose in the Maintenance Treatment Period + 1.
    - Note: This group could include subjects who discontinue the Maintenance Treatment Period early, subjects who complete the Maintenance Treatment Period as scheduled but choose not to continue into an open-label study, or subjects who are ongoing in the SFU period at the time of the data snapshot.

### 10.1.3 Exposure during the Initial and Maintenance Treatment Period

Definitions for study medication duration (days) and time at risk (days) during the entire study treatment period (the Initial and Maintenance Treatment Period combined) are provided as follows:

### Study medication duration (days)

For subjects who do not switch study treatments:

• Date of last dose – date of first dose + 28 days.

Note: If date of last dose + 28 days extends to a date beyond the final visit date (including PEOT, but not including SFU), then this calculation reverts to:

o Final visit date (including PEOT, but not including SFU) – date of first dose + 1.

Note: For subjects who die, if date of last dose + 28 days extends to a date beyond the date of death, then this calculation reverts to:

 $\circ$  Date of death – date of first dose + 1.

For subjects who switch study treatments (between Initial and Maintenance Treatment Periods):

- Initial Period (attributed to initially randomized treatment):
  - Date of last dose in the Initial Period date of first dose in the Initial Period + 28 days.
     Note: If date of last dose in the Initial Period + 28 days extends to a date beyond the date of first dose in the Maintenance Treatment Period, then this calculation reverts to:
  - Date of first dose in the Maintenance Treatment Period date of first dose in the Initial Period + 1.
- Maintenance Treatment Period (attributed to the treatment initiated in the Maintenance Treatment Period):
  - Use the study medication duration algorithm specified for the Maintenance Treatment Period.

### Time at risk (days):

For subjects who do not switch study treatments:

- For subjects who complete the Maintenance Treatment Period as planned and continue into an openlabel study (and, therefore, do not have the SFU visit in the feeder study): Final visit date – date of first dose + 1.
- For subjects who die prior to the final visit: Date of death date of first dose in the + 1.
- For all other subjects, use the minimum of the following:
  - Date of last dose date of first dose + 140 days.
  - Date of last clinical contact date of first dose + 1.

Note: This group could include subjects who discontinue early, subjects who complete the Maintenance Treatment Period as scheduled but choose not to continue into an open-label study, or subjects who are ongoing in the SFU period at the time of the data snapshot.

For subjects who switch study treatments (between Initial and Maintenance Treatment Periods):

- Initial Period (attributed to initially randomized treatment):
  - Date of first dose in the Maintenance Treatment Period date of first dose in the Initial Period + 1. (Note: This assumes that anyone in this category has completed the Initial Period and doses [with a new study treatment] in the Maintenance Treatment Period.)
- Maintenance Treatment Period (attributed to the treatment initiated in the Maintenance Treatment Period):
  - o Use the time at risk algorithm specified for the Maintenance Treatment Period.

A by-subject listing of exposure to study medications will be provided by treatment group.

### 10.2 Adverse events

An AE is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA version 19.0). For subjects who switch from placebo to bimekizumab at Week 16, any adverse events that occur after initiation of the new treatment are attributable to the new treatment. If an adverse event occurs on the date of a treatment switch, the event is attributed to the original treatment. The only exception to this is if the AE fulfills any of the criteria specified below:

- Events that fulfill the anaphylaxis criteria for acute events (refer to Appendix A in Section 12.1)
- Hypersensitivity events identified by the SMQ "Hypersensitivity (SMQ)" (see Section 12.1 Appendix A)
- Events with an HLT of "Administration site reactions NEC"
- Events with an HLT of "Injection site reactions"

### **10.2.1** Data considerations

Treatment-emergent AEs (TEAEs) are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period). If it is not possible (due to partial dates) to determine whether or not an AE is treatment-emergent then it will be assumed to be a TEAE.

The rules for imputing partial start or stop dates are outlined in Section 4.2.2.

AEs will be presented as "number of subjects (percentage of subjects) [number of events]". In this style of output, "[number of events]" will include all cases of an AE including repeat occurrences in individual subjects, while "number of subjects" will count each subject only once.

Subject time at risk represents the time a subject is at risk for having an AE. The definitions for subject time at risk (in days) are outlined in Section 10.1. These definitions will be used for exposure-adjusted AE summaries.

Selected AE summaries will include the exposure adjusted incidence rate (EAIR) with associated 95% confidence interval and the exposure adjusted event rate (EAER).

The EAIR is defined as the number of subjects (n) with a specific AE adjusted for the exposure and will be scaled to 100 patient-years:

EAIR = 
$$100 \times n / \sum_{i=1}^{N} (T_{Exp(i)})$$

If a subject has multiple events, the time of exposure is calculated to the first occurrence of the AE being considered. If a subject has no events, the total time at risk is used.

Exact Poisson 95% confidence intervals for incidence rates are calculated using the relationship between the Poisson and the Chi-square distribution (Ulm, 1990; Fay and Feuer, 1997):

$$UCL = \chi_{2n,\alpha/2}^{2}/2$$

$$UCL = \chi_{2(n+1),1-\alpha/2}^{2}/2$$

where n is the number of subjects with a specific AE for the incidence rate of interest and is the basis for the number of the degrees of freedom for the chi-square quantile for the upper tail probability  $\chi^2$ .

The EAER will be the number of AEs including repeat occurrences in individual subjects divided by the total time at risk scaled to 100 patient-years and calculated using:

$$EAER = 100 \times N_{AE} / \sum_{i=1}^{N} (T_{Risk(i)})$$

where N<sub>AE</sub> is the total number of AEs.

No confidence interval will be computed for EAER.

Selected summaries, as specified in Section 10.2.2, will include the risk difference between bimekizumab and ustekinumab. The risk difference is calculated as:

$$RD = IP_{BKZ} - IP_{ADA}$$

where  $IP_{BKZ}$  is the incidence proportion for the bimekizumab-treated group and  $IP_{PBO}$  is the incidence proportion for the placebo group. Note that incidence proportion simply refers to the percentage of subjects within the specified treatment group that experienced a given adverse event.

The standard error for the risk difference is calculated as follows:

$$SE_{RD} = \sqrt{\left(IP_{BKZ} \times \left(\frac{1 - IP_{BKZ}}{n_{BKZ}}\right)\right) + \left(IP_{PBO} \times \left(\frac{1 - IP_{PBO}}{n_{PBO}}\right)\right)}$$

where  $n_{BKZ}$  is the number of subjects in the bimekizumab-treated group and  $n_{PBO}$  is the number of subjects in the placebo group.

The corresponding confidence interval for the risk difference is as follows:  $CI_{RD} = RD \pm Z_{1-\alpha/2} \times (SE_{RD})$ 

$$CI_{RD} = RD \pm Z_{1-\alpha/2} \times (SE_{RD})$$

where  $Z_{1-\alpha/2}$  is the Z statistic for the corresponding level of alpha. For the risk difference confidence intervals calculated in this SAP, 1.96 will be used (corresponding to a two-sided alpha of 0.05 and 95% confidence interval).

#### 10.2.2 **AE Summaries**

The following summaries will be provided in three different ways: by treatment in the Initial Treatment Period for the SS, by treatment during the Maintenance Treatment Period for the MS, and by treatment during the Initial and Maintenance Treatment Period (combined) for the AMS:

- Incidence of TEAEs Overview
- Incidence of TEAEs per 100 subject years by SOC, HLT, and PT
- Incidence of Serious TEAEs per 100 subject years by SOC, HLT, and PT
- Incidence of TEAEs Leading to Discontinuation per 100 subject years by SOC, HLT, and PT

The following summaries will be provided in two different ways: by treatment in the Initial Treatment Period for the SS, and by treatment in the Initial and Maintenance Treatment Period (combined) for the AMS:

- Incidence of TEAEs Leading to Death by SOC, HLT, and PT
- Incidence of TEAEs by Maximum Relationship by SOC, HLT, and PT
- Incidence of Serious TEAEs by Relationship SOC, HLT, and PT Note: For EudraCT reporting purposes
- Incidence of Related Serious TEAEs by SOC, HLT, and PT
- Incidence of TEAEs Leading to Death by Relationship by SOC, HLT, and PT Note: For EudraCT reporting purposes
- Incidence of TEAEs by Maximum Severity, SOC, HLT, and PT

- Incidence of TEAEs by decreasing frequency of PT
- Incidence of Non-Serious TEAEs Above Reporting Threshold of 5% by SOC and PT
- Incidence of Non-Serious TEAEs by SOC, HLT, and PT
- Incidence of Non-Serious TEAEs by Maximum Relationship SOC, HLT, and PT
- Incidence of Non-Serious TEAEs Above Reporting Threshold of 5% by SOC and PT
- Incidence of Non-Serious TEAEs Above Reporting Threshold of 5% by Relationship SOC and PT
- Incidence of Related TEAEs by SOC, HLT, and PT
- Incidence of Related TEAEs Above Reporting Threshold of 5% by SOC and PT

The following summary will be provided by treatment for the Initial Treatment Period for the SS:

- Incidence of TEAEs Above Reporting Threshold of 5% with Risk Differences by SOC and
- Incidence of Serious TEAEs and Risk Differences by SOC and PT

The following summary will be provided by treatment for the Initial and Maintenance Treatment Period (combined) for the SS (only subjects treated with BKZ):

Incidence of TEAEs per 100 subject years by SOC, HLT, and PT and by Time of Onset Relative to Anti-bimekizumab Antibody Status

In addition, all summaries of TEAEs based on "100 subject years" will include EAIR (with 95% confidence interval) and EAER.

The tables with risk differences will also be accompanied by figures (dot plots) which show the incidence of the adverse events and corresponding 95% risk difference confidence intervals. These will be ordered by descending order of risk difference (bimekizumab vs ustekinumab).

For AEs that emerged after 112 days but still within the 140 days window, those AEs would be classified as TEAE. These AEs will be excluded from the outputs based on the Initial Period but included in the AE summaries for Initial and Maintenance Treatment Period.

# Other Safety topics of interest

Along with the tables described, there will be a table which distributed and statistical analyses confidence interval.

Along with the tables described, there will be a table which displays the risk difference and 95% confidence intervals for each of the topics of interest. A corresponding figure (with dot plots) will be prepared.

#### 10.2.3.1 Infections (serious, opportunistic, fungal and TB)

Incidence of Fungal Infection TEAEs per 100 subject years by SOC, HLT and PT

Fungal infections will be summarized in a stand-alone table. The table will include the serious and non-serious) which code into the High T infectious disorders."

Incidence of Fungal Infection TEAEs per 100 subject years by SOC, HLT and PT

Incidence

Incidence of Opportunistic Infection TEAEs per 100 subject years by SOC, HLT and

Opportunistic infections (including tuberculosis) will be summarized in a stand-alone table. The table will include all TEAEs identified using UCB-defined search criteria (refer to Excel spreadsheet on "OI - MedDRA v19.0.xlsx" in "Bimekizumab-Safety-Topics-of-Interest.docx").

The following steps are followed for identifying and reviewing opportunistic infections:

### **Identification Process**

The two steps below outline two ways in which opportunistic infections (or potential opportunistic infections) can be identified:

Step 1: Refer to column B of the spreadsheet which identifies the Preferred Terms (PTs) to be classified as opportunistic infections using either a single 'x' or a double 'xx'.

- TEAEs which code to a PT flagged with a single 'x' need to also be serious to be considered an opportunistic infection.
- All TEAEs which code to a PT flagged with a double 'xx' are considered to be an opportunistic infection, regardless of seriousness.

Step 2: Refer to column C of the spreadsheet which identifies the PTs that need to be evaluated on a case-by-case basis by the study physician to determine whether or not it is an opportunistic infection. If Column C has a single 'x', then the corresponding preferred term should be flagged for case-bycase review by the study physician.

## **Review Process**

Opportunistic infections for a given study will be reviewed on the following occasions:

At quarterly Infectious Disease Committee (IDC) Meetings, listings will be produced for each study (see details below) and reviewed by the corresponding study physician ahead of the IDC Meeting. These listings will be posted as part of the broader SSD deliverable to a folder named for the given quarter (eg, 2018Q4) on the SharePoint. They should be based on the same data cut as the one used for SSD and should be delivered at the same time as the SSD
outputs. The IDC will then agree on the final adjudication for each potential opportunistic infection.

In each of the circumstances described above, the study programming team will produce an Excel listing that will be provided to the project lead statistician, project lead programmer, and to the study physician (who will subsequently provide it to the IDC). The Excel following columns (using the descriptions had Adverse Event

Outcome

EAE Flag

Serious Adverse Event?

Relationship to Study Medication
Intensity
Action Taken with IMP

pportunistic Infection

portunistic Infection

portunistic Infection

- Data Cut Date
- Opportunistic Infection Final Adjudication

Note the following about the final 5 variables in this listing:

- Opportunistic Infection Automatic: This is flagged as "Y" if the criteria for automatic selection as described in "Step 1" of the identification process are met.
- Opportunistic Infection Manual Review: This is flagged as "Y" if the criteria for caseby-case selection as described in "Step 2" of the identification process are met.
- Flag This has a value of either "NEW" or "OLD". It is marked as "NEW" if the event is appearing for the first time in that run of the listing. Otherwise, if it has appeared previously, it is marked as "OLD". Unique records are determined by USUBJID AESPID for purposes of identifying whether an event has been modified from a previous run.
- Date Only for cases where Flag is "NEW", this field will be populated with the data cut date for that particular run of the listing.

Opportunistic Infection - Final Adjudication - For new events, this is always left blank by the programmers. It should be completed by the study physician/IDC for every event

Tollowing each review by the study physician and IDC, the Opportunistic Infection – Final Adjudication column will be completed (as described above), and the spreadsheets for each study will be returned to the study programming team via e-mail (coordinated by the IDC secretary adjudications from previous runs.

### 10.2.3.2

adjudications from previous runs.

2.3.2 Malignancies

Incidence of Malignant or Unspecified Tumours TEAEs per 100 subject years by SOC, **HLT** and **PT** 

These events will be presented in the following tables:

- One table will be based on the criteria Standardized MedDRA Query (SMO) = "Malignant or unspecified tumours (SMQ)"
- One table will be based on the criteria SMQ ="Malignant tumours (SMQ)".

SMQ search should include all TEAEs which code to a PT included in the Scope=Narrow group within each SMQ.

Note that the events included in the "Malignancies" table will be a subset of the events included in the "Malignancies (including unspecified)" table. While the "Malignant tumours (SMQ)" is most relevant, "Malignant or unspecified tumours (SMQ)" must be reviewed for potential malignancies.

The output tables will include 2 different overall incidence rows:

- The first overall incidence row will summarize "Any malignancy" and this row will summarize the incidence of all AEs flagged for inclusion in the table, (using the appropriate SMQ depending on the table) regardless of the High Level Term (HLT) it codes to.
- The second overall incidence row will summarize "Any malignancy" and this row will summarize the incidence of AEs flagged for inclusion in the table (using the appropriate SMQ depending on the table), excluding those which code to an HLT of "skin neoplasms malignant and unspecified (excl melanoma)".

#### 10,2.3.3 Major adverse cardiac event

Incidence of Adjudicated Major Cardiac Event (MACE) TEAEs per 100 subject years by SOC, HLT and PT

Major adverse cardiac events (MACE) will be presented in a table. The classification of an event as MACE is determined by an external cardiovascular event adjudication committee.

A separate table and listing will present the adjudicated cardiovascular events by type. For each cardiovascular event type (24 total), the individual PTs which fall within each event type will be summarized.

Jean or potential review by the cardiovascular event the reach event was the committee for formal review/adjudication.

1.2.3.4 Neutropenia

Incidence of Neutropenia TEAEs per 100 subject years by SOC, HLT and PT is table will be based on the following PTs (regardless of seriousness):

Autoimmune neutropenia

Band neutropenia

Cyclic neutropenia

Febrile neutropenia

Neutropenia

Neutropenia

Neutropenia infection

Neutropenia sepsis

Neutropenia sepsis

Neutrophil count decreased

Suicidal Ideation and Behavior (SIB)

dence of SIB-Adjudicated for and PT Additionally, a listing of all events identified for potential review by the cardiovascular event adjudication committee will be produced. This listing will indicate whether each event was escalated to the committee for formal review/adjudication.

### 10.2.3.4

This table will be based on the following PTs (regardless of seriousness):

### 10.2.3.5

**HLT and PT** 

An external neuropsychiatric adjudication committee will evaluate potential neuropsychiatric events and determine whether any of those events were associated with suicidal ideation and behavior (SIB). If an event is adjudicated as SIB, further information will be provided. A table and a separate listing for SIB events as determined by the adjudication committee will be included.

Additionally, a listing of all events identified for potential review by the neuropsychiatric adjudication committee will be produced. This listing will indicate whether each event was escalated to the committee for formal review/adjudication.

#### 10.2.3.6 Inflammatory bowel disease

Incidence of Inflammatory Bowel Disease TEAEs per 100 subject years by SOC, HLT and PT

These events will be presented in a stand-alone table which will include all TEAEs which code into the HLT of "Colitis excl infective".

Inflammatory bowel disease events will be summarized stratified by subjects with or without a previous medical history of inflammatory bowel disease. Previous medical history of inflammatory bowel disease will be determined using the information recorded on the Extra-Articular Assessment at Screening CRF page ("Does subject have a history of IBD?").

### 10.2.3.7 Anaphylactic reaction

- Incidence of Anaphylactic Reaction TEAEs per 100 subject years by SOC, HLT and PT
- A separate table will be prepared based on the MedDRA anaphylaxis Algorithm (see Appendix A) for acute anaphylactic events (reported on the same day as when an injection was administered or one day after).
- A separate table will be prepared to summarize hypersensitivity events, identified using the SMQ "Hypersensitivity (SMQ)". All TEAEs which code to a PT included in the Scope=Narrow search will be included in this table.

Furthermore, injection site reactions will be evaluated based on the any TEAE table (no separate table needed) by looking under the following HLTs: "Administration site reactions NEC" and "Injection site reactions".

### 10.2.3.8 Hepatic events and drug-induced liver injuries

• Incidence of hepatic events TEAEs per 100 subject years by SOC, HLT and PT

A table for hepatic events will be created based on the SMQ of "Drug related hepatic disorders - comprehensive search (SMQ)". However, these 2 sub-SMQs are to be excluded: "Liver neoplasms, benign (incl cysts and polyps) (SMQ)" and "Liver neoplasms, malignant and unspecified (SMQ)". For each of the above SMQs, include all TEAEs which code to a PT included in the Scope=Broad and/or Scope=Narrow.

Note that all AEs meeting the above criteria are to be included. It should not be limited to events that the investigator determined to be related to study drug.

Cases of Hy's Law will be reported separately in a liver function test table.

A by-subject listing of all AEs of safety topics of interest will be presented by type of safety topics of interest.

### 10.3 Clinical laboratory evaluations

Laboratory values, including markedly abnormal laboratory values will be presented descriptively by treatment group for SS.

Tables presenting markedly abnormal values and those based on CTCAE grade only include selected laboratory variables.

For tables where data are summarized by visit, unscheduled and repeat visits will not be summarized, but these data will be included in listings. For tables where multiple measurements over a period of time are considered (as in shift tables), unscheduled and repeat visits will be considered as long as they were collected in the period being summarized. All summaries will be presented in SI units and will be based on observed case values. In the case where laboratory values are below the lower limit of quantification, then these will be set to the midpoint between

0 and the lower limit of quantification for the purpose of summarizing the data. The following summaries are required:

- A summary of the number and percentage of subjects experiencing markedly abnormal values at any time while on treatment (assessment on or following the first dose of study treatment through the final dose of study treatment = 140 days) by laboratory variable and treatment group. Two separate tables will show results for the initial and maintenance treatment.

  A summary of the number and percentage of subjects experiencing markedly abnormal values at any time while on treatment (assessment on or following the first dose of study treatment proup. Two separate tables will show results for the initial and maintenance treatment.

  A summary of the number and percentage of subjects experiencing markedly abnormal values at any time while on treatment (assessment on or following the first dose of study treatment proup. Two separate tables will show results for the initial and maintenance treatment.
- A summary of the number and percentage of subjects with a given CTCAE grade (0, 1, 2, 3, or 4) based on minimum/maximum post-baseline value by laboratory variable and treatment group. Two separate tables will show results for the initial treatment period (for the SS) and the initial and maintenance treatment period (for the AMS).
- A shift table of the number and percentage of subjects experiencing CTCAE grade 0, 1, 2, 3, or 4 values (as applicable) at Baseline to minimum/maximum post-Baseline CTCAE grade, by laboratory variable and treatment group. Two separate tables will show results for the initial treatment period (for the SS) and the initial and maintenance treatment period (for the AMS).

Shift laboratory summaries will use the Baseline for Maintenance Treatment Period where applicable as described in Section 3.2.

A by-subject listing of all laboratory data will be provided. This listing will be presented by treatment group and will include: center, subject identifier, age, sex, race, weight, visit, laboratory variable, result (with abnormal values flagged as "L" or "H" accordingly) and unit.

Markedly abnormal values are defined as those with a severity of Grade 3 and above based on the common terminology criteria for adverse events (CTCAE) criteria (U.S. Department of Health and Human Services 2010). Definitions of markedly abnormal values using the Grade 3 cut points are given in the tables below for age ranges of  $\geq 17$  years (Table 10-1 for markedly abnormal liver function test values, Table 10-2 for markedly abnormal biochemistry values, and Table 10-3 for markedly abnormal hematology values). Tables summarizing markedly abnormal values should include a summary (counts and percentages) of markedly abnormal labs observed at any time while on treatment (ie, treatment-emergent markedly abnormal [TEMA]). For this summary, Baseline values and values observed more than 140 days after the last administration of study medication are not considered. The laboratory results classified as Grade 3 or Grade 4 will be summarized and listed separately.

Table 10–1: Definitions of Markedly Abnormal Liver Function Values

| | Conv | ventional | Sta | Abnormal | |
|----------------------|------|------------|------|------------|-------------|
| Parameter name | Unit | Criteria | Unit | Criteria | Designation |
| Alkaline Phosphatase | | >5.0 x ULN | | >5.0 x ULN | AH |
| ALT | U/L | >5.0 x ULN | U/L | >5.0 x ULN | AH |

| | Conv | ventional | Sta | Abnormal | |
|-----------------|-------|------------|--------|------------|----|
| AST | U/L | >5.0 x ULN | U/L | >5.0 x ULN | AH |
| Total Bilirubin | mg/dL | >3.0 x ULN | umol/L | >3.0 x ULN | AH |
| GGT | U/L | >5.0 x ULN | U/L | >5.0 x ULN | AH |

Table 10-2: Definitions of Markedly Abnormal Biochemistry Values

| | Con | ventional | Sta | Abnormal | |
|---|---|---|---|---|---|
| Parameter name | Unit Criteria | | Unit | Criteria | Designation |
| Creatinine | mg/dL | >3.0 x ULN | mmol/L | >3.0 x ULN | АН |
| Glucose | mg/dL | <40<br>>250 | mmol/L | <1.7<br>>13.9 | AL<br>AH |
| Calcium | mg/dL | >12.5<br><7.0 | mmol/Li | >3.1<br><1.75 | AH<br>AL |
| Magnesium | mg/dL | >3.00 | mmol/L | >1.23<br><0.4 | AH<br>AL |
| Potassium | mmol/L | 53.0 | mmol/L | >6.0<br><3.0 | AH<br>AL |
| Sodium | mmol/Q | 110 >155<br><130 | mmol/L | >155<br><130 | AH<br>AL |

Table 10-3: Definitions of Markedly Abnormal Hematology Values

| Q | Co | Conventional | | Standard | |
|---|---|---|---|---|---|
| Parameter name | Unit | Criteria | Unit | Criteria | Designation |
| Hemoglobin | g/dL | <8.0 | g/L | <80 | AL |
| USE | | >4.0 above ULN | | >40 above ULN | AH |
| Lymphocytes Absolute | $10^{9}/L$ | < 0.5 | $10^{9}/L$ | < 0.5 | AL |
| anno. | | >20.0 | | >20.0 | AH |
| Neutrophils Absolute | $10^{9}/L$ | <1.0 | $10^{9}/L$ | <1.0 | AL |
| Platelets | 10 <sup>9</sup> /L | <50 | 10 <sup>9</sup> /L | <50 | AL |
| WBC/Leukocytes | 10 <sup>9</sup> /L | <2.0 | 10 <sup>9</sup> /L | <2.0 | AL |
| | | >100 | | >100 | АН |

Abbreviations: AH=abnormal high; AL=abnormal low; ALT= alanine aminotransferase; AST = aspartate aminotransferase; dL = deciliter; GGT: gamma-glutamyltransferase; L = liter; mg = milligram; mmol = millimoles; µg = microgram; ULN = upper limit of normal.

The table for markedly abnormal liver function tests (LFTs) will contain data beyond the CTCAE Grade 3 thresholds outlined in Table 10–1: Definitions of Markedly Abnormal Liver Function Values above in order to allow for a more thorough review of elevated LFTs. There will be one table which will list the count and percentage of subjects meeting the below criteria at any time during the study:

- AST: >3xULN, >5xULN, >8xULN, >10xULN, >20xULN
- ALT: >3xULN, >5xULN, >8xULN, >10xULN, >20xULN
- AST or ALT: >3xULN, >5xULN, >8xULN, >10xULN, >20xULN
- Bilirubin: >1.5xULN, >2xULN

In addition, a table will be produced to summarize potential Hy's Law cases. The following two definitions will be used in that table:

• [AST ≥3xULN or ALT ≥3xULN] and Total Bilirubin ≥2xULN in the absence of ALP >2xULN

In order to meet the above criteria, a subject must experience the elevation in bilirubin and ALT or AST (and the absence of ALP elevation, if applicable) at the same visit. For example, a subject who experiences a  $\ge 2$  x ULN elevation of bilirubin at one visit and a  $\ge 3$ xULN elevation in ALT (or AST) at a subsequent visit has not fulfilled the Hy's law criteria.

# 10.4 Vital signs, physical findings, and other observations related to safety

### 10.4.1 Vital signs

The following vital signs variables should be summarized: systolic blood pressure (mmHg), diastolic blood pressure (mmHg), body temperature (°C) and heart rate (beats/min). The following summaries will be provided for SS:

- A summary of the absolute and change from Baseline value for each vital sign variable by treatment group and visit
- A summary of the number and percentage of subjects experiencing at least one markedly abnormal value for a vital sign variable as defined in Table 10–4, by treatment group.

Table 10-4: Definitions of Markedly Abnormal Blood Pressure Values

| Parameter (unit) | Markedly Abnormal Low | Markedly Abnormal High |
|---|---|---|
| Systolic blood pressure (mmHg) | <90 and a decrease from Baseline of ≥20 | >180 and an increase from Baseline of ≥20 |
| Diastolic blood pressure (mmHg) | <50 and a decrease from Baseline of ≥15 | >105 and an increase from Baseline of ≥15 |

Bimekizumab

A by-subject listing of all vital signs data will be provided. This listing should be presented by treatment group and will include: center, subject identifier, age, sex, race, weight, visit, vital sign

Abnormal results of the physical examination together with details of abnormalities: abnormality clinically significant or not, will be listed by subject and visit for SS.

10.4.3 Electrocardiograms

Electrocardiograms

A summary of the number and percentage of subjects with normal, abnormal ECG results, as determined by the central reader will be presented for all applicable visits.

The following ECG variables will be summarized (absolute visit: QTcF, RR, PR, QRS and QT

The following ECG variables will be summarized (absolute values and change from Baseline) by

QTc outliers are defined as QTcF values following dosing that are greater than 450 ms or are increases from Baseline greater than 30 ms. QTcF outliers will be highlighted in the data listing and summarized using the following categories:

- Values >450 ms, >480 ms, >500 ms
- Increase from Baseline of >30 ms, increase from Baseline of >60 ms, increase from Baseline of >90 ms
- Values >450 ms and increases of >30 ms. Values >500 ms and increases of >60 ms

The number and percentage of subjects who meet the ECG outlier criteria at any assessment post first dose will be summarized.

Two separate by-subject listings of all 12-lead ECG data will be provided based on interpretation from central reader and from site.

#### 10.4.4 Other safety variables

#### 10.4.4.1 Assessment and management of TB and TB risk factors

A summary of the number and percentage of subjects with negative, positive, and indeterminate IGRA (Interferon-Gamma Release Assay) results at all applicable visits will be presented for the Initial and Maintenance Treatment Period (combined).

A by-subject listing of the "Evaluation of signs and symptoms of tuberculosis" questionnaire data and IGRA results will be provided by treatment group.

A by-subject listing of the result of chest x-ray for tuberculosis will be provided by treatment

#### 10.4.4.2 Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)

eC-SSRS questionnaire will be self-administered by the subject and assessed by trained study personnel. This scale will be used to assess suicidal ideation and behavior that may occur during the study. Results of the eC-SSRS will be summarized using the number of subject and

 percentage with (i) suicidal ideation, (iii) suicidal behavior, (iii) suicidal ideation or behavior, ons or variations thereof. and (iv) self-injurious behavior without suicidal intent.

Suicidal ideation is defined as an event in any of the following 5 categories:



Suicidal behavior is defined as an event in any of the following 4 categories:

Suicidal behavior or ideation is defined as an event in any of the above 9 categories.

Self-injurious behavior without suicidal intent is defined as an event in the category non-suicidal self-injurious injuries.

The incidence of subjects with suicidal ideation, suicidal behavior, suicidal ideation or behavior, and self-injurious behavior will be summarized by treatment group.

A by-subject listing of the eC-SSRS questionnaire data will be provided by treatment group.

#### 10.4.4.3 Pregnancy testing

Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.

A by-subject listing of the pregnancy test data will be provided by treatment group.

#### 10.4.4.4 Childbearing potential and Lifestyle

Childbearing potential and lifestyle will be collected at Screening. A by-subject listing will be provided for all the subjects screened.

#### 10.4.45 Patient Health Questionnaire 9 (PHQ-9) scores

The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. The PHQ-9 scores for depression range from 0 to 27 with higher scores indicating worse state. A score of 5-9 is considered to be minimal symptoms of depression. A score of 10 to 14 is considered minor depression, dysthymia, or mild major depression. A score of 15 to 19 is considered to indicate moderately severe major depression, and a score ≥20 is considered to be severe major depression. Change from Baseline in PHQ-9 is derived as post-Baseline score minus Baseline score and will be summarized by treatment group.


#### 11 REFERENCES

Fay MP, Feuer EJ. Confidence intervals for directly standardized rates: A method based on the gamma distribution. Statistics in Medicine 1997; 16(7):791-801

Felson DT, Anderson JJ, Boers M, Bombardier C. Chora Co.

College of Rheumatology.

arthritis clinical trials. The Committee on Outcome Measures in Rheumatoid Arthritis Clinical Trials. Arthritis Rheum. 1993;36(6):729-40.

Food and Drug Administration. Guidance for Industry. Drug-induced liver injury: premarketing clinical evaluation. US Dept of Health and Human Services, Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research, 07/2009.

Greenland S, Robins JM. Estimation of common effect parameter from sparse follow up data. Biometrics 1985;41:55-68.

Husni ME, Qureshi AA, Keonig AS, Pedersen R, Robertson D. Utility of the PASE questionnaire, psoriatic arthritis (PsA) prevalenece and PsA improvement with anti-TNF therapy: results from the PRISTINE trial. J Dermatolog Treat. 2014;25(1):90-5.

Mallinckrodt CH, Watkin JG, Molenberghs G, Carroll RJ. Choice of the primary analysis in longitudinal clinical trials. Pharmaceutical Statistics 2004; 3:161-69

Mallinckrodt CH, Lin Q, Lipkovich I, and Molenberghs G. A structured approach to choosing estimands and estimators in longitudinal clinical trials. Pharmaceutical Statistics 2012; 11:456-

Mallinckrodt CH. Preventing and Treating Missing Data in Longitudinal Clinical Trials: A Practical Guide. New York, NY: Cambridge University Press; 2013.

Maruish, M. E., User's manual for the SF-36v2 Health Survey (3rd ed.). Lincoln, RI: Quality Metric Incorporated, 2011.

Ratitch, B., Lipkovich, I., O'Kelly, M. Combining Analysis Results from Mutiply Imputed Categorical Data, PharmaSUG, 2013, SP03

Rubin D.B. 1987. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley and Sons.

Thomas, D. Roland and Cyr, Andre. Applying Item Response Theory Methods to Complex Survey Data. SSC Annual Meeting, May 2002.

Ulm, K., A simple method to calculate the confidence interval of a standardized mortality ratio. American Journal of Epidemiology, 1990; 131(12), 373-375

U.S. Department of Health and Human Services, Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, June 2010.

### 12

**UCB** 

### 12.1

The SMQ Anaphylactic reaction consists of three parts:

Appendix A: MedDRA algorithmic approach to anaphyalaxis

see SMQ Anaphylactic reaction consists of three parts:

A narrow search containing PTs that represent core anaphylactic reaction terms.

A naphylactic reaction (SMQ)

P1 Anaphylactic transfusion reaction

P1 Anaphylactic transfusion reaction

P1 Anaphylactoid shock

P1 Anaphylactoid shock

P1 Dialysis membrane reaction

P1 Shock

P1 Shock symptom

P1 Type I hypersensitivity

A broad search that contains additional terms that are added to those included in the narrow search. These additional terms are signs and symptoms possibly indicative of anaphylactic □--SMQ Anaphylactic reaction (SMQ)

search. These additional terms are signs and symptoms possibly indicative of anaphylactic reaction and categorized in B, C or D

Cat B Acute respiratory failure ± R Asthma 🗓 🖁 Oedema mouth ⊕ Bronchial oedema ⊕ B Oropharyngeal spasm ± Bronchospasm E Chest discomfort ⊕ Respiratory arrest ± B Choking Respiratory dyskinesia . ☐ Choking sensation ⊕ B Respiratory failure ± Gircumorat oedema E Gough ⊞ Reversible airways obstruction E Cyanosis ⊕ B Sneezing ⊕ 🖁 Dyspnoea ⊕ 🖁 Stridor Hyperventilation 🖁 Irregular breathing ± Tachypnoea Taryngeal dyspnoea ± ☐ I Laryngeal oedema ± Tongue oedema ± B Laryngospasm Tracheal obstruction ± B Laryngotracheal oedema ± Tracheal oedema ± B Upper airway obstruction ± Wheezing

### Cat C



.e apapular extensions of variations thereof.

.aaed contration application and any extensions of variations thereof.

Cat D

⊞ Blood pressure diastolic decreased ⊞ Blood pressure systolic decreased ± Gardiac arrest E Cardio-respiratory arrest E Cardiovascular insufficiency ± ₩ Hypotension

- An algorithmic approach which combines a number of anaphylactic reaction symptoms in order to increase specificity. A case must include either (on either the same day as when an injection was administered or one day after):
  - A narrow term or a term from Category A;
  - A term from Category B (Upper Airway/Respiratory) AND a term from Category C -(Angioedema/Urticaria/Pruritus/Flush);
- [a term from Category C (Angioedema/Urticaria/
  Hypersensitivity events will be identified using the "Hypersensitivity (SMQ)". All TEAEs which code to a PT included in the Scope=Narrow search will be included. A term from Category D - (Cardiovascular/Hypotension) AND [a term from Category B -

### 12.2 Appendix B: Definition of CTCAE grades

Table 12–1: Definitions of CTCAE grades by biochemistry parameter

| Parameter (unit) | Definition | Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|
| Creatinine | High | mmol/L | >ULN-1.5 x<br>ULN | (>1.5 – 3.0)<br>x ULN | (>3.0 – 6.0)<br>x ULN | 6.0 x ULN |
| Sodium | Low | mmol/L | 130- <lln< td=""><td>N/A</td><td>120-&lt;130</td><td>120</td></lln<> | N/A | 120-<130 | 120 |
| Sodium | High | mmol/L | >ULN-150 | >150-155 | >155-160 | >160 |
| Potassium | Low | mmol/L | 3.0- <lln< td=""><td>3.0-<lln< td=""><td>2.5-&lt;3,0</td><td>&lt;2.5</td></lln<></td></lln<> | 3.0- <lln< td=""><td>2.5-&lt;3,0</td><td>&lt;2.5</td></lln<> | 2.5-<3,0 | <2.5 |
| Potassium | High | mmol/L | >ULN-5.5 | >5.5-6.0 | >6.0-7.0 | >7.0 |
| Calcium | Low | mmol/L | 2.0- <lln< td=""><td>1.75-&lt;2.0</td><td>1.5-&lt;1.75</td><td>&lt;1.5</td></lln<> | 1.75-<2.0 | 1.5-<1.75 | <1.5 |
| Calcium | High | mmol/L | >ULN-2.9 | >2.9-3.1 | >3.1-3.4 | >3.4 |
| Magnesium | Low | mmol/L | 0.5- <lln< td=""><td>0.4-≪0.5</td><td>0.3-&lt;0.4</td><td>&lt; 0.3</td></lln<> | 0.4-≪0.5 | 0.3-<0.4 | < 0.3 |
| Magnesium | High | mmol/L | >ULN-1.23 | N/A | >1.23-3.30 | >3.30 |

Table 12–2: Definitions of CTCAE grades by hematology parameter

| Parameter (unit) | Definition | Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|
| Hemoglobin | Low | g/L | 100< <lln< td=""><td>80-&lt;100</td><td>&lt;80</td><td>N/A</td></lln<> | 80-<100 | <80 | N/A |
| Hemoglobin | High | g/L | >0-20 above<br>BL | >20-40<br>above BL | >40 above<br>BL | N/A |
| Platelets | Low | 10%E | 75- <lln< td=""><td>50-&lt;75</td><td>25-&lt;50</td><td>&lt;25</td></lln<> | 50-<75 | 25-<50 | <25 |
| WBC | Low | 10°/L | 3- <lln< td=""><td>2-&lt;3</td><td>1-&lt;2</td><td>&lt;1</td></lln<> | 2-<3 | 1-<2 | <1 |
| WBC | High | 3 10 <sup>9</sup> /L | N/A | N/A | >100 | N/A |
| Lymphocytes | Low | 10 <sup>9</sup> /L | 0.8- <lln< td=""><td>0.5-&lt;0.8</td><td>0.2-&lt;0.5</td><td>&lt; 0.2</td></lln<> | 0.5-<0.8 | 0.2-<0.5 | < 0.2 |
| Lymphocytes | Hìgh | 10 <sup>9</sup> /L | N/A | >4-20 | >20 | N/A |
| Neutrophils | Low | 10 <sup>9</sup> /L | 1.5- <lln< td=""><td>1.0-&lt;1.5</td><td>0.5-&lt;1.0</td><td>&lt; 0.5</td></lln<> | 1.0-<1.5 | 0.5-<1.0 | < 0.5 |

Note that subjects who meet the decreased potassium criterion of 3.0< LLN, which is specified as the decreased potassium lab criterion for both CTCAE Grade 1 and Grade 2, will be counted as Grade 2.

#### 13 AMENDMENT(S) TO THE STATISTICAL ANALYSIS PLAN

#### 13.1 **Amendment 1**

### Rationale of the Amendment

isions or variations thereof. The main purpose of this amendment is to align the SAP with protocol amendment 3 and to achieve consistency with other SAPs of the program.

### **Modification and changes**

### **Global Changes**

The following changes were made throughout the SAP

- As no PD analysis will be performed (see specific change #4) references to PD or the PD-PPS have been removed from the SAP
- For the following endpoints, the definition of response has been clarified by adding the requirement of an improvement of at least two categories:
  - o Scalp IGA response (clear or almost clear with at least a two-category improvement from Baseline) for subjects with scalp PSO at Baseline
  - o Palmoplantar Investigator's Global Assessment (pp-IGA) response (clear or almost clear with at least a two-category improvement from Baseline) for subjects with palmoplantar PSO at Baseline
- The following changes have been done for the list of participating countries throughout the SAP:
  - o Region (North America [Canada, USA], Western Europe [Belgium, France, Germany, Italy, Norway, Spain, Sweden, Switzerland, United Kingdom], Central/Eastern Europe [Czech Republic, Hungary, Poland, Russian Federation], Asia/Australia [Australia, Japan, Korea, Taiwan])
- Throughout section 8.1 the term 'responder' has been replaced by 'response' (e.g. PASI100 response at Week 16 instead of PASI100 responder at Week 16)

## Specific Changes

### Change #1

### List of abbreviation

The following abbreviations have been added:

**ADAb** anti-bimekizumab antibodies

**LFT** liver function test

MedDRA Medical Dictionary for Regulatory Activities nADAb neutralizing anti-bimekizumab antibodies

Bimekizumab Statistical Analysis Plan

**ADAb** 

The following abbreviations have been removed:

DAP

DILI

**HLGT** 

LTB

ocol Set extensions of variations thereof.

cedure cedure and any extensions of variations thereof. PD-PPS

SOP

### Change #2

### 1 Introduction

Protocol Amendment 2.1, 15 Nov 2017

Has been changed to to

Protocol Amendment 3, 06 Apr 2018.

### Change #3

### Section 2.2.1.3 Other efficacy variables

The following variables have been added:

- Percent of subjects with absolute PASI score  $\leq 1, \leq 2, \leq 3$ , and  $\leq 5$
- Percent of subjects with absolute BSA=0\%,  $\leq$ 1\%,  $\leq$ 3\%, and  $\leq$ 5\%
- mNAPSI75 response (defined as a subject that achieves at least a 75% reduction from **Baseline in the mNAPSI score)**
- mNAPSI90 response (defined as a subject that achieves at least a 90% reduction from **Baseline in the mNAPSI score)**
- MNAPSI100 response (defined as a subject that achieves a 100% reduction from **Baseline in the mNAPSI score**)

### Change #4

### 2.2.2 Pharmacokinetic/pharmacodynamic variables

The pharmacokinetic (PK) variable is the plasma concentration of bimekizumab.

For subjects enrolled in participating centers, immunophenotyping by flow cytometry on whole blood will be performed.

### Has been changed to

### 2.2.2 Pharmacokinetic variable

The pharmacokinetic (PK) variable is the plasma concentration of bimekizumab.

### Change #5

### 2.3.1 Study Description

This study will include 4 periods, a Screening Period (2 to 4 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (36 weeks), and a safety follow-up (SFU) Period (20 weeks after the last dose of IMP).

### Has been changed to

This study will include 4 periods, a Screening Period (2 to 4 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (36 weeks), and a safety follow-up (SFU) Period (20 weeks after the final dose of IMP). The Maintenance Treatment Period starts with the first study drug administration on or after the Week 16 visit.

### Change #6

### 2.3.2.1 Screening Period

The Screening Period will last 2 weeks, but can be extended up to a total of 4 weeks.

### Has been changed to

The Screening Period with last 2 weeks, but can be extended up to a total of 5 weeks in cases where a laboratory assessment needs to be repeated or to allow washout of prohibited medications.

### Change #7

### 2.3.22 Initial Treatment Period

For subjects weighing ≤100kg (220lbs)...

### Has been changed to

For subjects weighing ≤100kg (220lbs) at Baseline...

### Change #8

### 3.2 Definition of Baseline Value

EQ-5D-3L VAS

• WPAI-SHP V2.0

Only the following variables remained in the first that the following pooling strategy and 4.2 'ollowing pooling strategy and Asia/Australia or Western Europe regions, the two regions will be combined as a geographic region stratum for efficacy modeling, so that there are no modeling convergence issues across efficacy variables.

# 3.10 Changes to protocol-defined analyses The following text has been added For the

The following text has been added to section 3.10:

For the following endpoints, the definition of response has been clarified:

Scalp IGA response (clear or almost clear with at least a two-category improvement from Baseline) for subjects with scalp PSO at Baseline

 Palmoplantar Investigator's Global Assessment (pp-IGA) response (clear or almost clear with at least a two-category improvement from Baseline) for subjects with palmoplantar PSO at Baseline

The following endpoints are not listed in the protocol, but have been added to the SAP in order to achieve consistency with other studies from the program:

- mNAPS175/90/100 response (defined as a subject that achieves at least a 75%, 90% and 100% reduction from Baseline in the mNAPSI score)
- Percent of subjects with absolute PASI score  $\leq 1, \leq 2, \leq 3$ , and  $\leq 5$
- Percent of subjects with absolute BSA=0%,  $\le 1\%$ ,  $\le 3\%$ , and  $\le 5\%$

### Change #11

### 4.2.1.1 Handling missing data for the primary efficacy variable

In addition, sensitivity analyses using MI-MCMC/monotone regression, MI-MCMC/reference based methods, and observed case (OC) method will be performed which will assess the impact of different methods of handling missing data.

### Has been changed to

In addition, sensitivity analyses using MI-MCMC/monotone regression, MI-MCMC/reference based methods, last observation carried forward (LOCF), and observed case (OC) method will be performed which will assess the impact of different methods of handling missing data.

### Change #12

### 4.2.1.4 Handling missing data for other efficacy variables

For other ordinal variables (EO-5D-3L and Patient Global Assessment of PSO), OC method will be applied as the primary analysis method.

### Has been changed to

For other ordinal variables (EQ-5D-3L, shift in IGA score, and Patient Global Assessment of PSO), OC method will be applied as the primary analysis method.

# 4.2.1.5 Missing data overview and summary

13 Sep 2019

Bimekizumab PS0009

Table 13-1: Missing data handling approach by variable priority and type

| Variable<br>Priority | Variable Type | NRI | MI<br>(MCMC/<br>Monotone<br>Regression) | MI<br>(MCMC/<br>Reference-<br>based) | LOCF | OC |
|---|---|---|---|---|---|---|
| Primary | Responder | P | Sa | Sa | | Silat |
| Secondary | Responder | P | Sa | | | of S |
| | Continuous | | P | | B | S |
| Other | Responder | P | | | Kens | S <sup>b, c</sup> |
| | Continuousf | | P | | J ⊗ T B | S <sup>b, d</sup> |
| | Ordinal | | | 80 | | Pe |

P=Primary method, S=Sensitivity method, B=Backup method

Note: Backup method is only applicable when the primary method is unable to converge due to challenges with the imputation model.

### Has been changed to

Table 13-1: Missing data handling approach by variable priority and type

| Variable<br>Priority | Variable Type | NRKO | MI<br>(MCMC/<br>Monotone<br>Regression) | MI<br>(MCMC/<br>Reference-<br>based) | LOCF | ОС |
|---|---|---|---|---|---|---|
| Primary | Responder | P | $S^a$ | S <sup>a</sup> | S | S |
| Secondary | Responder | P | $S^a$ | | | S |
| | Continuous | | P | | В | S |
| Other | Responder | P | | | | S <sup>b, c</sup> |
| Other Calling ! | Continuousf | | P | | В | S <sup>b, d</sup> |
| ant | Ordinal | | | | | Pe |

P=Primary method, S=Sensitivity method, B=Backup method, NRI=Nonresponder imputation, MI=Multiple imputation, MCMC=Markov Chain Monte Carlo, LOCF=Last observation carried forward, OC=Observed Case

Note: Backup method is only applicable when the primary method is unable to converge due to challenges with the imputation model.


<sup>&</sup>lt;sup>a</sup> Imputation method is applied on continuous data, and responder variable is derived from the continuous variable based on complete data set.

<sup>&</sup>lt;sup>b</sup> Only applies to by-visit summaries of variables that are in the multiplicity-controlled testing procedure.

<sup>&</sup>lt;sup>c</sup> Includes PASI75, PASI90, Scalp IGA, IGA

e includes Patient Global Assessment of PSO and EQ-5D-3L

<sup>&</sup>lt;sup>a</sup> Imputation method is applied on continuous data, and responder variable is derived from the continuous variable based on complete data set.

<sup>b</sup> Only applies to by-visit summaries of variables that are in the multiplicity-controlled testing procedure.

### Change #14

### 4.2.1.6 Missing data algorithms

In bullet point 1 the following sentences have been added:

The seed used for these imputations will be 852 (note that all other multiple imputation procedures described in this SAP related to analyses will use this same seed as well).

The following sentence has been added (as already mentioned in Change #9):

In the event that the percentage of randomized subjects is less than 10% in either of the Asia/Australia or Western Europe regions, the two regions will be combined as a geographic region stratum for efficacy modeling, so that there are no modeling convergence issues across efficacy variables.

In bullet point 2d the seed range has been specified:

Repeat steps 2a-2d, 100 times with different seed values (seeds ranging from 853 to 952) to create 100 imputed complete data sets.

### Change #15

### 4.8 Examination of subgroups

Subgroup analyses will be performed on the PASI75/90/100 and IGA. The following subgroup analyses will be used:

- Age (<40 years, 40 to <65 years,  $\ge65$  years)
- Gender (male, female)
- Disease duration (<median, ≥median)
- Region (North America [Canada, USA], Western Europe [Belgium, France, Germany, Italy, Norway, Spain, Sweden, Switzerland, United Kingdom], Central/Eastern Europe [Czech Republic, Hungary, Poland, Russian Federation], Asia/Australia [Australia, Japan, Korea, Taiwan])
- Weight ( $\leq$ 100 kg, >100 kg)
- BMI ( $<25 \text{ kg/m}^2$ , 25 to  $<30 \text{ kg/m}^2$ ,  $\ge 30 \text{ kg/m}^2$ )
- Prior systemic chemotherapy or photochemotherapy (yes, no)
- Prior biologic exposure (yes, no)

<sup>&</sup>lt;sup>c</sup> Includes PASI75, PASI90, **PASI100**, Scalp IGA, IGA response

<sup>&</sup>lt;sup>d</sup> Includes PSD of PSO for pain, itch, and scaling

e includes Patient Global Assessment of PSO, IGA score, and EQ-5D-3L

<sup>&</sup>lt;sup>f</sup> For PASE, OC is the primary analysis method.

- Prior systemic therapy of any kind (yes, no)

ne definition of prior systemic therapy of any kind is if a subject received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic photochemotherapy or phototherapy. Subjects who never received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic photochemotherapy or phototherapy or photother

### Has been changed to

### 4.8 Examination of subgroups

Subgroup analyses will be performed on the PASI75/90/100 and IGA. The following subgroups **for** analysis will be determined using Baseline data:

- Age (<40 years, 40 to <65 years,  $\ge65$  years)
- Gender (male, female)
- Disease duration (<median, ≥median)
- Region (North America [Canada, USA], Western Europe [Belgium, Germany, Italy, United Kingdom, Central/Eastern Europe [Hungary, Poland, Russian Federation], Asia/Australia [Australia, Japan])
- Weight (≤100 kg, >100 kg)
- BMI ( $<25 \text{ kg/m}^2$ , 25 to  $<30 \text{ kg/m}^2$ ,  $\ge 30 \text{ kg/m}^2$ )
- Prior systemic chemotherapy or phototherapy (yes, no)
- Prior biologic exposure (yes, no)
- Prior systemic therapy of any kind (yes, no)
- Baseline disease severity (PASI<20, PASI≥20)
- Antibody positivity (confirmatory assay: negative or positive)

The definition of prior systemic therapy of any kind is if a subject received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic **chemotherapy** or phototherapy. Subjects who never received previous biologic therapy, previous systemic therapy (non-biologic), or previous systemic **chemotherapy** or phototherapy will be classified as not receiving prior systemic treatment for psoriasis.

In addition, in order to assess whether an early response to treatment is predictive of response at later time points, subgroup analyses will be performed on PASI90/100 and IGA over time using the following early response subgroups:

- PASI75 response at Week 4 (yes, no) to predict PASI90/100 and IGA through Week 16
- PASI90 response at Week 16 (yes, no) to predict PASI100 through Week 52

All summaries detailed in this section will be performed on the SS by treatment group.

Summaries for demographics and other Baseline characteristics will also be repeated in FAS and MS. If the SS and FAS analysis sets are identical the summaries will not be repeated.

Has been changed to

All summaries detailed in this section will be performed on the SS by treatment group.

Summaries will also be repeated in FAS and MS. If the SS and FAS analysis sets are identical the summaries will not be repeated.

All summaries detailed in this section will be performed on the RS by treatment group. Summaries for demographics and other Baseline characteristics will also be repeated in SS and MS. If the **RS** and **SS** analysis sets are identical the summaries will not be repeated.

### Change #17

### **6.2 Other Baseline Characteristics**

Prior phototherapy or chemophototherapy (yes, no)

### Has been changed to

Prior phototherapy or chemotherapy (yes, no)

### Change #18

## 7 MEASUREMENTS OF TREATMENT COMPLIANCE

Table 7-1 has been added:

Table 13-1: Dosing scheme

| Week<br>Dose<br>Assignment | Baselin<br>e (first<br>dose) | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Bimekizumab<br>320mg Q4W | 0. | • | • | • | •• | •• | •• | • | •• | •• | • | •• | •• |
| Ustekinumab<br>45mg (subjects<br>≤100kg) | ▲ ○ | ▲ ○ | 0 | 00 | ▲ ○ | 00 | 00 | • | 00 | 00 | ▲ ○ | 0 | 00 |
| Ustekinumab<br>90mg (subjects<br>>100kg) | <b>A A</b> | <b>A A</b> | 00 | 00 | <b>A A</b> | 00 | 00 | <b>A A</b> | 00 | 00 | <b>A A</b> | 00 | 00 |
| Placebo/<br>bimekizumab<br>320mg Q4W | 00 | 00 | 00 | 00 | •• | •• | •• | •• | •• | •• | •• | •• | •• |

Q4W=every 4 weeks

Statistical Analysis Plan

Notes: A bimekizumab 160mg injection is depicted by a black circle (●). A placebo injection is depicted by a white circle (○). A ustekinumab 45mg injection is depicted by a black triangle (▲).

### Change #19

#### 8.1.1.1 **Psoriasis Area and Severity Index (PASI)**

The following clarification has been added:

PASI90 is defined to be equal to 1 if the percentage improvement from Baseline in the PASI scores is 90% or greater and 0 if the percentage improvement from Baseline is less than 90%. This definition is introduced for the purpose of identifying subjects who respond to the treatment (1 = responder, 0 = non-responder).

8.1.3 Sensitivity analyses of the co-primary efficacy variables

Sensitivity Analysis #4

The primary efficacy or in the primary The primary efficacy analyses from Section 8.1.2 will be repeated based on the FAS and the PPS.

### Has been changed to

The primary efficacy analyses from Section 8.1.2 will be repeated using LOCF as the imputation method (see Section 4.2.1.5).

Sensitivity Analysis 5 has been added

### Sensitivity Analysis #5

The primary efficacy analyses from Section 8.1.2 will be repeated based on the FAS and the PPS.

### Sensitivity Analysis #6 (previously Sensitivity Analysis #5)

In addition, if the logistic regression model cannot converge due to lack of any placebo responders, then Fisher's exact test will be used for inferential comparisons to placebo. As with the primary analysis, missing data will be handled using NRI.

### Has been changed to

In addition, if the logistic regression model cannot converge, then Fisher's exact test will be used is docuMRI. for inferential comparisons. As with the primary analysis, missing data will be handled using

Sensitivity Analysis #7 from SAP version 1.0 has been removed from SAP amendment 1.


### Change #21

### 8.2.3 Sensitivity analyses of the secondary efficacy variables

For binary response variables (PASI100 at Week 16, PASI75 at Week 4, Scalp IGA at Week 16, PASI90 at Weeks 12 and 52, and IGA at Weeks 12 and 52), sensitivity analyses #1 and #3 (Sections 8.1.3.1, 8.1.3.3) will be performed.

In addition, for PASI90 and IGA response at Week 52, sensitivity analysis #7 will be performed.

For change from Baseline in PSD response for itch, pain, and scaling, sensitivity analyses #3 (Section 8.1.3.3) will be performed.

Details regarding Missing data algorithm can be found in Section 4.2.1.6.

### Has been changed to

Sensitivity analyses for the handling of missing data will be performed for the binary and continuous secondary efficacy variables that are part of the fixed sequence testing procedures in Figure 4–1.

For binary response variables (PASI100 at Week 16, PASI75 at Week 4, Scalp IGA at Week 16, PASI90 at Weeks 12 and 52, and IGA at Weeks 12 and 52), sensitivity analyses #1 and #3 (Sections 8.1.3.1, 8.1.3.3) will be performed.

For change from Baseline in PSD response for itch, pain, and scaling, sensitivity analyses #3 (observed cases, Section 8.1.3.3) will be performed.

Missing data for binary secondary efficacy variables will be imputed using NRI.

Missing data for continuous secondary efficacy variables will be imputed using MI. The MI procedure for continuous variables will be similar to sensitivity analysis #1 described in Section 8.1.3.1 for the co-primary efficacy endpoints with the following differences: 1) the imputation model will use the change from Baseline (instead of actual) values by visit and no dichotomization will be necessary; and 2) the analysis model will be based on ANCOVA as opposed to the stratified CMH test.

### Change #22

### 8.3.2 Modified Nail Psoriasis Severity Index (mNAPSI) score

The following sentence has been added

An mNAPSI75 responder is defined as a subject who achieved at least a 75% improvement from Baseline in the mNAPSI score. mNAPSI90 and mNAPSI100 are defined accordingly. The proportion of mNAPSI75/90/100 responders over time will be summarized for each treatment group.

### Change #23

8.3.3 IGA response

13 Sep 2019 PS0009

A line plot of the IGA, scalp IGA responder rate over time, by treatment group will be produced.

### Has been changed to

A line plot of the IGA responder rate over time, by treatment group will be produced.

### Change #24

### 8.3.6 Dermatology Life Quality Index (DLQI)

Percent of subjects achieving a minimal clinically important difference (MICD) in DLQI is defined as the number of subjects with improvement from Baseline score of 4 or more divided by the number of subjects in RS.

### Has been changed to

Percent of subjects achieving a MCID in DLQI is defined as the number of subjects with improvement from Baseline score of 4 or more divided by the number of subjects in RS. Only subjects with a Baseline DLQI of 4 or greater will be considered for this analysis.

### Change #25

### 8.3.7 Patient's Global Assessment of Disease Activity (PGADA)

The PGADA for the arthritis VAS will be used to provide an overall evaluation of arthritis disease symptoms. Subjects will respond to the question, "Considering all the ways your arthritis affects you, please mark a vertical line on the scale below to show how you are feeling today," using a VAS where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms."

Change from Baseline in PGADA is defined as Post-Baseline PGADA minus Baseline PGADA.

### Has been changed to

## 8.3.7 Patient's Global Assessment of Disease Activity (PGADA) for arthritis visual analog scale (VAS)

The PGADA for the arthritis VAS will be used to provide an overall evaluation of arthritis disease symptoms. Subjects will respond to the question, "Considering all the ways your arthritis affects you, please mark a vertical line on the scale below to show how you are feeling today," using a VAS where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms."

All subjects will complete the PGADA at Baseline. Subjects with PsA at Baseline (defined as a past medical history of PsA or PASE  $\geq$ 47) will complete the PGADA at the visits specified in the protocol.

Change from Baseline in PGADA is defined as Post-Baseline PGADA minus Baseline PGADA.

### Change #26

### 8.3.8 Patient Global Assessment of PSO score

The following sentences have been removed:

The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from Screening to Week 16 Visit with a +3 day completion window. During the Maintenance Treatment Period this assessment will be completed at each clinic visit specified in the protocol with a ±3 day completion window.

### Change #27

### 8.3.9 Patient Symptom Diary (PSD)

In addition, cumulative distribution plots (see details in Section 8.2.2.3) will be provided for absolute and percent change from Baseline PSD at Week 16 for each item

### Has been changed to

In addition, cumulative distribution plots (see details in Section 8.2.23) will be provided for absolute change from Baseline PSD at Week 16 for each item

### Change #28

### 8.4 Statistical analysis of PsA related efficacy variables

The following clarification has been added

The following PsA related efficacy variables will only be assessed for subjects enrolled in Japan:

- Swollen and tender joint count
- Physician's Global Assessment of Disease Activity (PhGADA)
- Patient's Assessment of Arthritis Pain VAS
- C-Reactive Protein (CRP)

Subsequently, also ACR20/50/70 are only calculated for subjects enrolled in Japan.

### Change #29

### 9.1 Pharmacokinetics

In addition, geometric mean plasma concentration will be plotted by treatment group, and by cumulative antibody status for subjects randomized to bimekizumab.

PK concentrations will also be listed.

### Has been changed to

In addition, geometric mean plasma concentration will be plotted by treatment group, and by isions of variations thereof cumulative antibody status for subjects randomized to bimekizumab on linear and log linear scale.

If the dosing for a visit is +/- 21 days out of window, then the plasma concentration from that visit and all subsequent visits will be excluded from the PK summary.

However, all PK concentrations will be listed.

### Change #30

**UCB** 

Sections 9.2 Pharmacodynamics and 9.3.1 Auto-antibodies have been set to **not applicable**.

### Change #31

### 9.3.2 Anti-bimekizumab antibodies

Anti-bimekizumab antibody status will be determined for each visit where samples were taken for drug concentration measures. At each visit:

- Values ≤ predefined cut point are defined as anti-bimekizumab antibody -
- Values > predefined cut point are defined as anti-bimekizumab antibody +

In addition, overall anti-bimekizumab antibody status should be determined:

- Subject overall anti-bimekizumab antibody + is defined as having a value > predefined cut point at any time in the treatment period. This does not include Baseline/pre-treatment.
- Subject anti-bimekizumab antibody positivity at Baseline is defined as having a value > predefined cut point at Baseline.
- Subject overall anti-bimekizumab antibody is defined as having no values > predefined cut point during the treatment period.

Note that the predefined cut point value is lab-specific and specific for different indications. Cut-off values must be provided by the lab performing the analysis prior to database lock.

The number and percentage of subjects with anti-bimekizumab antibody levels above the specified cut point will be reported as:

- Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at the time of each visit
- Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at any visit during the treatment period.

In addition, the timepoint of the first occurrence of anti-bimekizumab antibody positivity during the treatment period (excluding Baseline and pre-treatment) will be summarized for each treatment group.

All individual subject-level anti-bimekizumab antibody results will be listed.

screening assay, confirmatory assay and titration assay. Samples confirmed as positive within the confirmatory assay, will be further evaluated in a neutralizing assay to evaluate the potential of the ADAb to neutralize the activity of Bimekizumab (IL17A or II.17E and both) in-vitro. Samples were taken at Baseline, Week 4 Week 24, Week 40. and Week 3. (PS0014) a sample at SFU which is 20 weeks after the last dose.

In subjects randomized to Ustekinumab, no ADAb samples will be analysed.

In subjects randomized to placebo for the first 16 weeks, no samples will be analysed until Week 16 which will act as the Baseline for this treatment group

Screening, confirmatory and titer cut points of the respective assays will be determined by the bioanalytical laboratory based either on using commercially available drug-naïve samples or on the pre-dose samples of the study itself. In case cut point is being set on commercially available samples, the representative for the study population is being checked. The screening cut point will be used to determine the status of ADA in test sample as above the cut point or below the cut point. Samples presenting ADA levels above the cut point, will be further evaluated in the confirmatory assay, the result of which will be reported as either "confirmed positive" or "not confirmed positive".

- Values ≤ screening cut point (BCP) or above the screening cut point and confirmed negative (NCP) are defined as anti-bimekizumab antibody negative
- Values > predefined screening cut point (ACP) and confirmed positive (CP) are defined as anti-bimekizumab antibody positive
- Confirmed positive samples will be titrated, and the titer (reciprocal dilution factor including MRD) reported. The samples (or a subset) will also be subject to a neutralizing assay to evaluate whether the anti-bimekizumab antibody neutralizes the activity of bimekizumab (IL17 A or IL17F or both) in-vitro. This will be reported subsequent to the main DBL and CSR.

### **Subject Classification:**

- For subjects who are negative at Baseline, and antibody negative at all sampling points post treatment (including SFU) - pre ADAb negative - treatment emergent **ADAb** negative
- For subjects who are negative at Baseline, and antibody positive at any sampling point post treatment (including SFU) - pre ADAb negative - treatment emergent ADAb positive. If a subject has a missing pre-treatment sample (either missing or insufficient volume) at Baseline with one or more ADAb positive post-treatment samples will be also classified as pre ADAb negative - treatment emergent ADAb positive

- For subjects who are positive at Baseline, and antibody negative at all sampling points post treatment (including SFU) - pre ADAb positive - treatment emergent
- Subjects who are positive at Baseline, and are positive <u>at any</u> sampling point post treatment (including SFU) with titer values of the same magnitude as Baseline (i.e. ≤ then a predefined fold difference from the Baseline value) pre ADAh positive.

  For all:
- For subjects who are positive at Baseline, and are positive at any sampling point post treatment (including SFU) with increased titer values compared to Baseline (above a predefined fold difference increase from Baseline value which will be defined within the validation of the assay and will be included in the TFLs and/or SAP when available) - pre ADAb positive - treatment emergent ADAb boosted positive.
- For Subjects who have a positive pre-treatment sample and some post-treatment samples are missing, while other post-treatment samples are ADAb negative, the subject will be classed as inconclusive.

In addition to the ADAb classifications, subjects will also receive an overall neutralizing (nADAb) classification for each nADAb assay separately, inclusive of Baseline and post-Baseline results, on the nADAb assay results:

- nADAb negative: no nADAb positive samples at Baseline or post-Baseline
- nADAb positive: one or more positive samples at Baseline or post-Baseline
- Missing: relevant nADAb samples are missing, e.g. if subject had samples selected for nADAb testing based on their ADAb levels, but there was insufficient sample left for nADAb testing. >

### **Analysis**

Immunogenicity will be assessed through summary tables and figures, and listing of individual results by subject. All analyses will be run on the safety population, unless specified otherwise.

- Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at the time of each visit, separated by treatment group
  - Number and percentage of subjects with anti-bimekizumab antibody level above the specified cut point at any visit during the treatment period, separated by treatment group.
- The time-point of the first occurrence of anti-bimekizumab anti-body positivity during the treatment period) will be summarized for each treatment group. A plot of the Titre versus elapsed time will be plotted
- All individual subject-level anti-bimekizumab antibody results will be listed.

- The number and percentage of subject in each of the 6 categories will be tabulated and separated by treatment group with an additional category combining subjects
- The prevalence of immunogenicity, separated by treatment group, and defined subcategory, will be reported per time point, defined as (cumulative) proportion of that time point. Missing samples will
- The time to achieving treatment-emergent ADAb positivity, separated by treatment group and defined sub-category, will be analyzed based on Kaplan-Meier approach, subjects will be considered to have an event at time where treatment emergent ADAb positive is first achieved. Subjects classified as treatment-emergent ADAb negative will be censored at time of last available ADAb result.
- A summary of PASI 90 responder, separated by treatment group and defined subcategory, at Weeks 16 and 52 as a function of ADAb fiter will be presented graphically. This will be repeated for PASI 100 and 75 responders.
- Individual plots of Bimekizumab Concentrations/ADAb titer and % Change from Baseline (all Y-axes) versus time (x-axis) for the full treatment period, including SFU where a patient has not progressed into the OLE. Plots should be labeled and grouped into the 6 sub-categories.
- Spaghetti plots of ADAb titer (Y-axis) against time (X-axis), separated by treatment group for all ADAb positive subjects, including Baseline positive subjects.
- Box plots of all Bimekizumab concentrations where ADAb titers exists versus ADAb titer classification (group 1 >; group 2 >; group 3 >) presented on a linear scale. Cut points will be determined on availability of the titre data.
- A summary table to present the incidence (%) of subjects classified as treatment emergent ADAb positive with incidence of IL17-A and IL17F neturalizing ADAb, respectively over the 52 weeks.

### Change #31

### 10.1 Extent of Exposure

durations of time, the following categories for duration will be used:

• >0 weeks The cumulative study medication duration will be summarized for subjects exposed for given

- >=16 weeks
- $\geq$ =24 weeks

- >=48 weeks

ne cumulative study medication duration will be summarized for subjects exposed for given durations of time, with four weekly categories through Week 16 and 24. For the cumulative duration through Week 52 the following categories for duration will be used:

• >0 weeks

• >=16 weeks ative ative and any extensions of vari

- >=16 weeks
- >=24 weeks
- >=52 weeks

### Change #32

### 10.2 Averse events

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). For subjects who switch from placebo to bimekizumab at Week 16, AEs will be allocated to the treatment the subject was on the day the event occurred. If the event occurs on the day of the switch, it will be attributed to placebo, unless the event has a HLT of "Injection" Site Reactions, in which case it will be attributed to bimekizumab.

### Has been changed to

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA version 19.0). For subjects who switch from placebo to bimekizumab at Week 16, any adverse events that occur after initiation of the new treatment are attributable to the new treatment. If an adverse event occurs on the date of a treatment switch, the event is attributed to the original treatment. The only exception to this is if the AE fulfills any of the criteria specified below:

- Events that fulfill the anaphylaxis criteria for acute events (refer to Appendix A in Section 12.1)
- Events with a reported term containing the term "hypersensitivity"
- Events with an HLT of "Administration site reactions NEC"
- Events with an HLT of "Injection site reactions"

### Change #30

### 10.2.3.1 Infections (serious, opportunistic, fungal and TB)

The embedded OI - MedDRA v19.0.xlsx file has been removed from the document.

### And

- 1. Study programming team creates a spreadsheet which lists all of the subjects with a TEAE present in the database which codes to a PT identified as case-by-case. Information from the AE dataset to be included in the spreadsheet: Subject ID, AE verbatim term, SOC, High Level Term (HLT), Lower Level Term (LLT), PT, AE start date, AE end date, seriousness, severity, relationship to study medication, action taken. Additionally, a column will be included where the study physician can document their decision on the case.
- 2. Study physician reviews the cases in the spreadsheet and indicates in the additional column which AEs are confirmed to be opportunistic infections via a single 'x'.
- 3. Study programming team incorporates these decisions into the AE dataset by merging the study physician decisions for individual subjects / PTs and flagging the confirmed opportunistic infections as such in the dataset.

### Has been changed to

- 1. Study programming team creates a spreadsheet which lists all of the subjects with a TEAE present in the database which codes to a PT identified as case-by-case. Information from the AE dataset to be included in the spreadsheet: Subject ID, AE verbatim term, SOC, High Level Term (HLT), Lower Level Term (LLT), PT, AE start date, AE end date, seriousness, severity, relationship to study medication, action taken. Additionally, a column will be included where the study physician can document their decision on the case.
- 2. Study physician reviews the cases in the spreadsheet and indicates in the additional column which AEs are confirmed to be opportunistic infections via a single 'x'.
- 3. At quarterly Infectious Disease Committee (IDC) Meetings, outputs will be produced and reviewed by the study physician ahead of the IDC Meeting. The IDC will then agree on the final adjudication for each potential opportunistic infection. A final output for opportunistic infections will be produced and agreed upon between the study physician and the IDC prior to finalizing the database.
- 4. Study programming team incorporates these decisions into the AE dataset by merging the **final** decisions for individual subjects / PTs and flagging the confirmed opportunistic infections as such in the dataset.

### Change #33

### 10.2.3.1 Clinical laboratory evaluations

Laboratory values (including markedly abnormal laboratory values), urinary values will be presented descriptively by treatment group for SS.

### Has been changed to

Laboratory values and urinary values will be presented descriptively by treatment group for SS.

Markedly abnormal values and shifts from Baseline (Week 0) will be presented for the SS.

### And

A summary table highlighting the potential cases of Hy's Law, within each treatment group will be presented. Hy's Law is defined as:

- AST >3xULN or ALT >3xULN and
- Total Bilirubin >2xULN

In order to meet the above criteria, a subject must experience the elevation in bilirubin and ALT or AST at the same visit. For example, a subject who experiences a >=2 x ULN elevation of bilirubin at one visit and a 3 x ULN elevation in ALT (or AST) at a subsequent visit has not fulfilled the Hy's law criteria.

### Has been changed to

The table for markedly abnormal liver function tests (LFTs) will contain data beyond the CTCAE Grade 3 thresholds outlined in Table 10–1: Definitions of Markedly Abnormal Liver Function Values above in order to allow for a more thorough review of elevated LFTs. There will be one table which will list the count and percentage of subjects meeting the below criteria at any time during the study:

- AST: >2xULN, >3xULN, >5xULN, >10xULN, >20xULN
- ALT: >2xULN, >3xULN, >5xULN, >10xULN, >20xULN
- AST or ALT: >2xULN, >3xULN, >5xULN, >10xULN, >20xULN
- Bilirubin: >1xULN, >1.5xULN
- ALP: >2xULN

In addition, a table will be produced to summarize potential Hy's Law cases. The following two definitions will be used in that table:

- [AST ≥3xULN or ALT ≥3xULN] and Total Bilirubin ≥2xULN
- [AST ≥3xULN or ALT ≥3xULN] and Total Bilirubin ≥2xULN in the absence of ALP  $\geq 2xULN$

In order to meet either of the above criteria, a subject must experience the elevation in bilirubin and ALT or AST (and the absence of ALP elevation, if applicable) at the same visit. For example, a subject who experiences a  $\geq 2$  x ULN elevation of bilirubin at one visit and a ≥3xULN elevation in ALT (or AST) at a subsequent visit has not fulfilled the Hy's law criteria.

# Change #33

Appendix A: MedDRA algorithmic approach to anaphyalaxis has been added

Statistical Analysis Plan

#### 13.2 **Amendment 2**

### **Rationale of the Amendment**

The main purpose of this amendment is to align the SAP with protocol amendment 4 and to achieve consistency with other SAPs of the program.

### **Modification and changes**

### **Global Changes**

The following changes were made throughout the SAP

- "IGA response (defined as Clear with at least a 2-category improvement relative to Baseline) at Week 16" has been added as a secondary endpoint
- The secondary endpoint "Change from baseline in the Patient Symptom Diary responses for itch, pain, and scaling at Week 16" has been altered to "Patient Symptom Diary responses for itch, pain, and scaling at Week 16"
- "Change from Baseline in Patient Health Questionnaire (PHQ) 9 scores" is no longer seen as an efficacy endpoint and got moved from the efficacy section to the safety section

### **Specific Changes**

### Change #1

### List of abbreviation

The following abbreviation have been added:

SIB suicidal ideation and behavior

### Change #2

### 2.3.2.2 Initial Treatment Period

Subjects will be classified as completing the initial treatment period if they complete the Week 16 Visit without early withdrawal from the study or if they start treatment in the maintenance treatment period. The start of the maintenance treatment period marks the end of the initial treatment period.

### Has been changed to:

Subjects will be classified as completing the initial treatment period if they complete the Week 16 Visit without early withdrawal from the study or if they start treatment in the maintenance treatment period. The start of the maintenance treatment period marks the end of the initial treatment period.

### Change #3

#### 2.3.5 Anticipated regions and countries

The following got added:

A subset of tables, listings, and figures will be repeated for the subgroup of subjects randomized in Japan. A list of these outputs will be added to the TLF shells.

### Change #4

#### 3.2 **Definition of Baseline values**

tensions of variations thereof. A Baseline value for a subject is defined as the latest measurement for that subject up to and including the day of administration of first study medication, unless otherwise stated. If a Baseline assessment is taken on the same day as first administration of study medication, it is eligible to be used as the Baseline value, even in the case that the time of the assessment is recorded as taking place after the time of first study medication administration. This is considered acceptable as this measurement is still the best representation of the Baseline value of the given assessment since it is highly unlikely that the study medication could have an impact on any measurement in such a short period of time. However, such cases should be rare as study center personnel are instructed to do all assessments at the Baseline visit prior to administering study medication. One exception to this rule is plasma concentration. If Baseline plasma concentration is measured at a time after the first administration of study medication, then it should not be eligible to be considered as a Baseline plasma concentration. Such cases should be discussed with the quantitative clinical pharmacologist. If a Baseline measurement is missing or not collected, and a Screening value is available, the Screening value will be utilized as Baseline instead.

For subjects who switch treatment from placebo to bimekizumab at the Week 16 Visit, the variables listed below, will have an additional Baseline defined as the Baseline for Maintenance Treatment Period. Baseline for Maintenance Treatment Period is the latest measurement on/prior to the day of first dose in the maintenance period.

PASI score

### Has been changed to

A Baseline value for a subject is defined as the latest measurement for that subject up to and including the day of administration of first study medication, unless otherwise stated. If a Baseline assessment is taken on the same day as first administration of study medication, it is eligible to be used as the Baseline value, even in the case that the time of The assessment is recorded as taking place after the time of first study medication administration. This is considered acceptable as this measurement is still the best representation of the Baseline value of the given assessment since it is highly unlikely that the study medication could have an impact on any measurement in such a short period of time. However, such cases should be rare as study center personnel are instructed to do all assessments at the Baseline visit prior to administering study medication. One exception to
this rule is plasma concentration. If Baseline plasma concentration is measured at a time after the first administration of study medication, then it should not be eligible to be considered as a Baseline plasma concentration. Such cases should be discussed with the quantitative clinical pharmacologist. If a Baseline measurement is missing or not collected, and a Screening value is available, the Screening value will be utilized as Baseline instead.

For subjects who switch treatment from placebo to bimekizumab at the Week 16 Visit, the variables listed below, will have an additional Baseline defined as the Baseline for Maintenance Treatment Period. Baseline for Maintenance Treatment Period is the latest measurement on/prior to the day of first dose in the maintenance period.

- PASI score
- DLQI
- Laboratory data (only in shift tables)

Note that for any laboratory value that occurs on the day of treatment switch, that lab value will be attributed and summarized for the treatment they were on previously. For subjects that switch treatment, the Baseline value is the laboratory value of the day of treatment switch.

Baseline values for component scores should be computed using components from the same visit where the relevant measurements were recorded prior to dosing. For example, if the Screening visit has all of the components, but the Baseline visit is missing one or more components, the Baseline value for the component score should be calculated using the Screening visit values.

## Change #5

## 4.2.1.6 Missing data algorithms

Modifications have been made to the text regarding the multiple imputation algorithm for clarity.

## **Change #6**

#### 4.4 Multicenter studies

The following has been added:

If convergence still cannot be achieved, this analysis will not be performed.

## Change #7

#### 4.8 Examination of subgroups

The following has been added:

Antibody positivity is the only subgroup that is not determined by Baseline data. It will be presented in a separate table.

#### In the following text analysis sets and imputation methods have been added for clarity:

PASI75 response (OC) at Week 4 (yes, no) to predict PASI90/100 and IGA (NRI) through Week 52

PASI90 response (OC) at Week 16 (yes, no) to predict PASI90/100 and IGA (NRI) through Week 52 In addition, in order to assess whether an early response to treatment is predictive of response at later time points, subgroup analyses will be performed for the RS on PASI90/100 and IGA over time using the following early response subgroups:

- PASI90 response (OC) at Week 16 (yes, no) to predict PASI100 (NRI) through Week 52

#### Change #8

#### 6.2 Other Baseline characteristics

The following variables have been added to the list of other baseline characteristics:

- Nail involvement (yes, no)
- Scalp involvement (yes, no)
- Palmoplantar involvement (yes, no)
- Prior primary failure to biologic (yes/no)
- PSD items: Pain, Itch, Scaling

 PSD items: Pain, Itch, Scaling
 Baseline nail, scalp, and palmoplantar involvement are based on the number of subjects achieving mNAPSI>0, Scalp IGA>0, and pp-IGA>0, respectively.

## Change #9

#### 7 MEASUREMENTS OF TREATMENT COMPLIANCE

The following has been removed:

All summaries detailed in this section will be performed on the SS

#### Percentages and analysis sets have been updated in the following:

A summary of percent treatment compliance categorized as <75% and >>75% will be provided by treatment group and study periods (Initial Treatment Period for the SS, Maintenance Treatment Period for the MS, and the Initial and Maintenance Treatment Period for the AMS).

# Change #10 8.1.2

#### Primary analysis of the co-primary efficacy variables

The primary analysis will be based on the stratified Cochran-Mantel-Haenszel (CMH) test where region and prior biologic exposure (yes/no) will be used as stratification variables. For the assessment of noninferiority, a noninferiority margin of 10% will be used and evaluated based on the confidence interval for the stratified Cochran Mantel-Haenszel risk difference between bimekizumab and ustekinumab. A non-inferiority margin of 10% has been selected as this is considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO. Therefore, a difference within the 10% non-inferiority margin would suggest a similar impact on efficacy between the treatments. The evaluation of superiority will use pairwise treatment comparisons based on the CMH test using the p-value for the general association. The odds ratio and associated confidence interval (CI) based on the Wald test will be presented. If one of the treatment groups has 0 or very low response where CMH can no longer be used, the logit method will be applied instead.

#### Has been changed to:

The primary analysis will be based on the stratified Cochran-Mantel-Haenszel (CMH) test where region and prior biologic exposure (yes/no) will be used as stratification variables. For the assessment of noninferiority, a noninferiority margin of 10% will be used and evaluated based on the confidence interval for the stratified Cochran Mantel-Haenszel risk difference between bimekizumab and ustekinumab. A non-inferiority margin of 10% has been selected as this is considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO. Therefore, a difference within the 10% non-inferiority margin would suggest a similar impact on efficacy between the treatments. The evaluation of superiority will use pairwise treatment comparisons based on the CMH test using the p-value for the general association. The odds ratio and associated confidence interval (CI) based on the Wald test will be presented. If one of the treatment groups has 0 or very low response where CMH can no longer be used, the logit method will be applied instead.

#### And

The number and percentage of subjects who are PASI90 responders and those who are non-responder at Week 16 will be summarized. IGA response will be summarized in the same manner as PASI90 responder variable.

#### Has been changed to

The number and percentage of subjects who are PASI90 responders at Week 16 will be summarized. IGA response will be summarized in the same manner as PASI90 responder variable.

#### And

Details about the calculation of the stratified Mantel-Haenszel risk difference, using the method of Greenland and Robins (1985), have been added.

## **C**hange #11

#### 8.1.3.7 Sensitivity Analysis #7

#### The following has been added:

In order to achieve model convergence, other explanatory variables e.g. other prior biologic exposure may be dropped from the model as for the logistic regression with region.

#### Change #12

#### 8.2.1.4 Patient Symptom Diary (PSD)

The PSD consists of 14 different items, each measuring an aspect of the disease and its impact on the subject's quality of life. Each item will be scored separately on a 0-10 scale with 0 for no symptom and 10 for very severe or worst symptom. Weekly averages will be derived for each of the 14 items of the Psoriasis Diary up to Week 16. A weekly average is the sum of the scored item over the course of the study week divided by the number of days on which the item was completed and will be set to missing if four or more daily assessments (irrespective of whether these are consecutive or not) were missing of the corresponding question. only if there are no data available from any of the daily assessments during the previous week for the corresponding question.

#### Has been changed to:

The PSD consists of 14 different items, each measuring an aspect of the disease and its impact on the subject's quality of life. Each item will be scored separately on a 0-10 scale with 0 for no symptom and 10 for very severe or worst symptom. Weekly averages will be derived for each of the 14 items of the Psoriasis Diary up to Week 16. A weekly average is the sum of the scored item over the course of the study week (up to the actual visit date) divided by the number of days on which the item was completed and will be set to missing if four or more daily assessments (irrespective of whether these are consecutive or not) were missing of the corresponding question. The Baseline value is also based on a weekly average (up to and including the Baseline visit) and will be computed in the same manner.

## Change #13

## 8.2.2 Primary analysis of the secondary efficacy variables

#### The following has been updated:

Primary analysis for secondary efficacy variables will be summarized based on imputed data (NRI and MCMC/Monotone Regression for binary and continuous variables, respectively), unless otherwise specified.

## Change #14

8.2.2.3 Patient Symptom Diary (PSD)

#### The following has been removed

The percentage change as well as the absolute change from Baseline to the Week 16 for the weekly average will be analyzed in separate analyses of covariance (ANCOVA) with fixed effects of treatment, region and prior biologic exposure and Baseline value as a covariate. The

analysis based on the absolute change from Baseline will be the primary analysis. Differences between treatment groups will be determined using least square means and t tests using the pooled error term from the linear model. 95% confidence intervals for the treatment difference will be calculated based on differences in least-square means estimates. All continuous variables in the model will be centered with respect to their mean values. Missing data for these PSD variables will use the MI procedure similar to the sensitivity analysis #1 (Section 8.1.3.1) used in the co-primary analysis with the following differences:

- 1) The imputation model will use change from Baseline (instead of actual) valued by visit and no dichotomization will be necessary;
- 2) The analyses model will be based on analysis of covariance (ANCOVA Cochran-Mantel-Haenszel (CMH) test.

There may be cases where the multiple imputation model fails to converge. In such situations, the last observation carried forward (LOCF) approach will instead be used to impute the missing data. If LOCF is used instead of multiple imputation for this reason, this will be clearly specified in the corresponding table summary. Note that for LOCF imputation, any missing data or data collected following discontinuation of IMP will be imputed with the most recent previous value.

#### Change #15

# Sensitivity analyses of the secondary efficacy variables 8.2.3

The following has been added:

Missing data for these PSD responder variables will use the MI procedure similar to the sensitivity analysis #1 (Section 8.1.3.1) for the co-primary efficacy variables with the following differences:

- 5. The data included in the imputation model will be limited only to those subjects with sufficiently high Baseline values to achieve the response for a given item (based on observed cases).
- 6. The PSD item value will be imputed. Once imputation has been performed across the 100 iterations specified, any values below 0 and above 10 will be truncated to 0 and 10, respectively.
- 7. The change from Baseline values will be computed based on the complete data sets.
- The analysis model will be based on the CMH test.

# Change #16 8.3

### Statistical analysis of the other efficacy variables

#### The following has been added:

Summaries for subjects switching from Placebo to Bimekizumab will be provided separately for the MS.

Time to PASI50, PASI90, and PASI100 response (in days) during the Initial Treatment Period will each be calculated as:

Min (Date of first PASIxx response, Date of Week 17)

with xx representation 70 with xx representing 50, 75, 90, 100 respectively.

Subjects who discontinue study treatment without achieving a given PASI response prior to Week 16 visit will be censored at the date of study treatment discontinuation. Subjects who reach the Week 16 Visit without achieving the given response will be censored at the date of the Week 16 Visit.

#### Has been changed to:

Time to PASI50, PASI75, PASI90, and PASI100 response (in days) during the Initial Treatment Period will each be calculated as:

Min (Date of first PASIxx response, Date of Week 16 visit) - Date of Baseline visit + 1, with xx representing 50, 75, 90, 100 respectively. All visits including unscheduled visits are considered.

Subjects who discontinue study treatment without achieving a given PASI response prior to Week 16 visit will be censored at the date of the last observed PASI assessment on or prior to the date of treatment discontinuation. Subjects who reach the Week 16 Visit without achieving the given response will be censored at the date of the last observed PASI assessment on or prior to the Week 16 Visit, Subjects will be censored at Baseline if there is no Baseline PASI assessment or no Post Baseline PASI assessment.

#### Change #18

#### 8.3.2 Modified Nail Psoriasis Severity Index (mNAPSI) score

If 1 or 2 response items scored on the 0 to 1 scale are missing, the missing response(s) will be imputed by the average of the available responses. Otherwise, the total mNAPSI score will be set to missing.

#### Has been replaced by:

If any of the 7 response items that contribute to mNAPSI is present, while other items are missing (ie, partial mNAPSI data), then the missing items are assumed to be 0 for the mNAPSI calculation. In some cases, the data may be captured in such a way that only nonzero component scores are present in the database. Again, those components that are not present are simply assumed to be 0 for the mNAPSI calculation.

#### Change #19

#### 8.5 Additional statistical analysis of other efficacy variables

Added new Section 8.5 for additional statistical testing for other efficacy variables with nominal p-values

#### Change #20

#### 9.1 Pharmacokinetics

#### Value of LLOG has been added:

...then for calculation of the derived statistics the result will be set to 0.125  $\mu$ g/ml, which is ½ of the lower level of quantification (LLOQ).

#### The following has been added:

If the PK sampling date is >1 day after the dosing date data points will be excluded from the PK summary tables and figures, but not from the listing.

#### Change #21

#### 9.3 Immunogenicity

The analysis of immunogenicity will be based on the PK-PPS.

#### Has been changed to:

The analysis of immunogenicity will be based on the SS.

## Change #22

#### 9.3.2 Anti-bimekizumab antibodies

The following two bullet points for subject classification have been updated:

- For subjects who are positive at Baseline, and are positive at any sampling point post treatment (including SFU) with titer values of the same magnitude as Baseline (i.e. ≤ than a 2.07 fold difference from the Baseline value) pre ADAb positive treatment emergent unaffected ADAb positive
- For subjects who are positive at Baseline, and are positive at any sampling point post treatment (including SFU) with increased titer values compared to Baseline (i.e. > than a 2.07 fold difference from the Baseline value) pre ADAb positive treatment emergent ADAb boosted positive.

The following has been added:

Derivation for above classification will be different for the interim analysis and the final analysis. For the interim analysis no SFU data will be considered. Only for the final analysis, when all SFU data will be available, data from the SFU visits will be considered.

$$RD = IP_{BKZ} - IP_{ADA}$$

Selected summaries, as specified in Section 10.2.2, will include the risk difference between bimekizumab and ustekinumab. The risk difference is calculated as:  $RD = IP_{BKZ} - IP_{ADA}$  where  $IP_{BKZ}$  is the incidence proportion for the bimekizumab-treated group and  $IP_{PBO}$  is the incidence proportion for the placebo group. Note that incidence proportion percentage of subjects within the specified treatment of the proportion of the placebo group.

The standard error for the risk difference is calculated as follows:

$$SE_{RD} = \sqrt{\left(IP_{BKZ} \times \left(\frac{1 - IP_{BKZ}}{n_{BKZ}}\right)\right) + \left(IP_{PBO} \times \left(\frac{1 - IP_{PBO}}{n_{PBO}}\right)\right)}$$

where  $n_{BKZ}$  is the number of subjects in the bimekizumab-treated group and  $n_{PBO}$  is the number of subjects in the placebo group.

The corresponding confidence interval for the risk difference is as follows:

$$CI_{RD} = RD \pm Z_{1-\alpha/2} \times (SE_{RD})$$

where  $Z_{1-\alpha/2}$  is the Z statistic for the corresponding level of alpha. For the risk difference confidence intervals calculated in this SAP, 1.96 will be used (corresponding to a two-sided alpha of 0.05 and 95% confidence interval).

## Change #24

#### 10.2.2 AE Summaries

## Section has been updated to:

The following summaries will be provided in three different ways: by treatment in the Initial Treatment Period for the SS, by treatment during the Maintenance Treatment Period for the MS, and by treatment during the Initial and Maintenance Treatment Period (combined) for the AMS:

- Incidence of TEAEs Overview
- Incidence of TEAEs per 100 subject years by SOC, HLT, and PT
- Incidence of Serious TEAEs per 100 subject years by SOC, HLT, and PT
- Incidence of TEAEs Leading to Discontinuation per 100 subject years by SOC, HLT, and PT


The following summaries will be provided in two different ways: by treatment in the Initial Incidence of Related Serious TEAEs by SOC, HLT, and PT — Note: For EudraCT, with the reporting purposes

Incidence of TEAEs Land:

Ender CT

Incidence of TEAEs Land:

Ender CT Treatment Period for the SS, and by treatment in the Initial and Maintenance Treatment Period (combined) for the AMS:

- Incidence of TEAEs Leading to Death by Relationship by SOC, HLT, and PT Note: EudraCT reporting purposes

  Incidence of TEAEs by Management of TEAEs by Managem
- Incidence of TEAEs by decreasing frequency of PT
- Incidence of TEAEs Above Reporting Threshold of 5% by SOC and PT
- Incidence of Non-Serious TEAEs by SOC, HLT, and PT
- Incidence of Non-Serious TEAEs by Relationship SOC, HLT, and PT
- Incidence of Non-Serious TEAEs Above Reporting Threshold of 5% by SOC and PT
- Incidence of Non-Serious TEAEs Above Reporting Threshold of 5% by Relationship SOC and PT
- Incidence of Related TEAEs by SQC, HLT, and PT
- Incidence of Related TEAEs Above Reporting Threshold of 5% by SOC and PT

The following summary will be provided by treatment for the Initial Treatment Period for the SS:

- Incidence of TEAEs Above Reporting Threshold of 5% with Risk Differences by SOC and PT
- Incidence of Serious TEAEs and Risk Differences by SOC and PT

The following summary will be provided by treatment for the Initial and Maintenance Treatment Period (combined) for the SS (only subjects treated with BKZ):

• Incidence of TEAEs per 100 subject years by SOC, HLT, and PT and by Time of Onset Relative to Anti-bimekizumab Antibody Status

In addition, all summaries of TEAEs based on "100 subject years" will include EAIR (with 95% confidence interval) and EAER.

The tables with risk differences will also be accompanied by figures (dot plots) which show the incidence of the adverse events and corresponding 95% risk difference confidence

13 Sep 2019

PS0009

intervals. These will be ordered by descending order of risk difference (bimekizumab vs ustekinumab).

#### Change #25

#### 10.2.3 Other Safety topics of interest

The section has been updated to:

The following are AEs of other safety topics of interest that require special statistical analyses and will be provided in two different ways: by treatment in the Initial Treatment Period for the SS, and by treatment in the Initial and Maintenance Treatment Period (combined) for the AMS.

Along with the tables described, there will be a table which displays the risk difference and 95% confidence intervals for each of the topics of interest. A corresponding figure (with dot plots) will be prepared.

#### Change #26

10.2.3.1 Infections (serious, opportunistic, fungal and TB)

The whole section about identification and review of opportunistic infections has been updated.

## Change #27

## 10.2.3.3 Major adverse cardiac event

The following has been added:

A separate table and listing will present the adjudicated cardiovascular events by type. For each cardiovascular event type (24 total), the individual PTs which fall within each event type will be summarized.

Additionally, a listing of all events identified for potential review by the cardiovascular event adjudication committee will be produced. This listing will indicate whether each event was escalated to the committee for formal review/adjudication.

## Change #28 10.2.3.5 Section

#### 10.2.3.5 Suicidal Ideation and Behavior (SIB)

Section title has been updated and the following has been removed:

This table is based on the SMQ of "Depression and suicide/self-injury" (all TEAEs which code to a PT included in the Scope=Broad and/or Scope=Narrow).

13 Sep 2019

PS0009

Inflammatory bowel disease events will be summarized stratified by subjects with or without a previous medical history of inflammatory bowel disease. Previous medical history of inflammatory bowel disease will be determined using the information recommend on the Extra-Articular Assessment at Screening CRF page ("Does or IBD?").

#### Change #30

#### 10.2.3.7 **Anaphylactic reaction**

This table will be prepared based on the MedDRA anaphylaxis algorithm (refer to Appendix 1 in Section 12.1") for acute events (reported on the same day) and for treatment-emergent PTs including the term "hypersensitivity" reported at any time.

#### Has been replaced by the following:

- A separate table will be prepared based on the MedDRA anaphylaxis Algorithm (see Appendix A) for acute anaphylactic events (reported on the same day as when an injection was administered or one day after).
- A separate table will be prepared to summarize hypersensitivity events, identified using the SMQ "Hypersensitivity (SMQ)". All TEAEs which code to a PT included in the Scope=Narrow search will be included in this table.

## Change #31

#### Clinical laboratory evaluations 10.3

#### Section has been updated to:

Laboratory values, including markedly abnormal laboratory values and urinary values will be presented descriptively by treatment group for SS.

Tables presenting markedly abnormal values and those based on CTCAE grade only include selected laboratory variables.

For tables where data are summarized by visit, unscheduled and repeat visits will not be summarized, but these data will be included in listings. For tables where multiple measurements over a period of time are considered (as in shift tables), unscheduled and repeat visits will be considered as long as they were collected in the period being summarized. All summaries will be presented in SI units and will be based on observed case values. In the case where laboratory values are below the lower limit of quantification, then these will be set to the midpoint between

0 and the lower limit of quantification for the purpose of summarizing the data. The following summaries are required:

- A summary of the number and percentage of subjects experiencing markedly abnormal values at any time while on treatment (assessment on or following the first dose of study treatment through the final dose of study treatment + 140 1 and treatment group. Two sees period (for the SS) and the initial and maintenance treatment period (for the AMS).
- A summary of the number and percentage of subjects with a given CTCAE grade (0, 1, 2, 3, or 4) based on minimum/maximum post-baseline value by laboratory variable and treatment group. Two separate tables will show results for the initial treatment period (for the SS) and the initial and maintenance treatment period (for the AMS).
- A shift table of the number and percentage of subjects experiencing CTCAE grade 0, 1, 2, 3, or 4 values (as applicable) at Baseline to minimum/maximum post-Baseline CTCAE grade, by laboratory variable and treatment group. Two separate tables will show results for the initial treatment period (for the SS) and the initial and maintenance treatment period (for the AMS).

Shift laboratory summaries will use the Baseling for Maintenance Treatment Period where applicable as described in Section 3.2

A by-subject listing of all laboratory data will be provided. This listing will be presented by treatment group and will include: center, subject identifier, age, sex, race, weight, visit, laboratory variable, result (with abnormal values flagged as "L" or "H" accordingly) and unit.

Markedly abnormal values are defined as those with a severity of Grade 3 and above based on the common terminology criteria for adverse events (CTCAE) criteria (U.S. Department of Health and Human Services 2010). Definitions of markedly abnormal values using the Grade 3 cut points are given in the tables below for age ranges of ≥17 years (Table 10-1 for markedly abnormal liver function test values, Table 10-2 for markedly abnormal biochemistry values, and Table 10-3 for markedly abnormal hematology values). Tables summarizing markedly abnormal values should include a summary (counts and percentages) of markedly abnormal labs observed at any time while on treatment (ie, treatment-emergent markedly abnormal [TEMA]). For this summary, Baseline values and values observed more than 140 days after the last administration of study medication are not considered. The laboratory results classified as Grade 3 or Grade 4 will be summarized and listed separately.

13 Sep 2019 PS0009

of the of the state of the stat


## **Approval Signatures**

| Name: | PS0009-sap-amend-2 | |
|---|---|---|
| Version: | 1.0 | |
| Document Number: | CLIN-000141074 | |
| Title: | PS0009 Statistical Analysis Plan | s Variat |
| Approved Date: | 13 Sep 2019 | sions of |
| | | provals |
| | | dication and |
| | Document Ap | |
| Approval<br>Verdict: Approved | Na<br> Ca <br> Da | me: coacity: Clinical<br>te of Signature: 13-Sep-2019 12:55:45 GMT+0000 |
| Approval<br>Verdict: Approved | RECORDANT Na Cap Da | me:<br>pacity: Clinical<br>te of Signature: 13-Sep-2019 13:07:53 GMT+0000 |
| ised to | Na Ca Da | |
| cument cannot be used to | | |